CLINICAL TRIAL: NCT01525550
Title: A SINGLE-ARM OPEN-LABEL INTERNATIONAL MULTI-CENTER STUDY OF THE EFFICACY AND SAFETY OF SUNITINIB MALATE (SU011248, SUTENT (REGISTERED)) IN PATIENTS WITH PROGRESSIVE ADVANCED METASTATIC WELL-DIFFERENTIATED UNRESECTABLE PANCREATIC NEUROENDOCRINE TUMORS
Brief Title: A Study Of The Efficacy And Safety Of Sunitinib In Patients With Advanced Well-Differentiated Pancreatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Other
Other Study IDs: A6181202; 2011-004363-74 (EudraCT Number)
Record Dates: First submitted 2012-01-13; First posted 2012-02-03 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Well-differentiated Pancreatic Neuroendocrine Tumor
Keywords: neuroendocrine tumors; adenoma islet cells; carcinoma islet cells; pancreatic neoplasms; angiogenesis inhibitors; sunitinib; neoplasms; carcinoma; adenoma
MeSH Terms: conditions — Neuroendocrine Tumors; Pancreatic Neoplasms; Neoplasms; Carcinoma; Adenoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sunitinib (Experimental)
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — Sunitinib capsules will be given orally at continuous daily dosing with a starting dose of 37.5 mg. One cycle is equal to 28 days.

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of sunitinib in subjects with unresectable pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This study is being conducted to meet regulatory post-marketing commitments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of well-differentiated pancreatic neuroendocrine tumor (according to World Health Organization [WHO 2000] classification).
* Disease progression within 12 months prior to study enrollment.
* Disease that is not amenable to surgery, radiation, or combined modality therapy with curative intent.

Exclusion Criteria:

* Patients with poorly differentiated pancreatic neuroendocrine tumors (according to WHO 2000 classification).
* Prior treatment with any tyrosine kinase inhibitors, anti vascular endothelial growth factor (VEGF) angiogenesis inhibitors, non VEGF targeted angiogenesis inhibitors, or mammalian target of rapamycin (mTOR) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-06-06 (Actual); Primary Completion 2016-03-19 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (2):
  - Univeristy of California, Orange, California
  - Columbia University Medical Center, New York, New York
- Barwon Health - University Hospital Geelong, Geelong, Victoria, Australia
- Cliniques Universitaires Saint-Luc, Gastroenterologie, Brussels, Brussels Gewest, Belgium
- China (7):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - 307 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni poliklinika, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- Hôpital Beaujon, Clichy, France
- Semmelweis Egyetem/II. Sz. Belgyogyaszati Klinika, Budapest, Hungary
- Tata Memorial Hospital, Mumbai, Maharashtra, India
- IEO Istituto Europeo di Oncologia, IRCCS, Milan, Italy
- Japan (2):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Romania (2):
  - Centrul de Oncologie Sf. Nectarie, Craiova, Dolj
  - Institutul Clinic Fundeni, Centrul de Gastroenterologie si Hepatologie, Bucharest
- Narodny Onkologicky ustav, Bratislava, Slovakia
- Wits Clinical Research, Johannesburg, Gauteng, South Africa
- Hospital Universitario Madrid Sanchinarro - Centro Integral Oncológico Clara Campal (CIOCC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fazio N, Kulke M, Rosbrook B, Fernandez K, Raymond E. Updated Efficacy and Safety Outcomes for Patients with Well-Differentiated Pancreatic Neuroendocrine Tumors Treated with Sunitinib. Target Oncol. 2021 Jan;16(1):27-35. doi: 10.1007/s11523-020-00784-0. Epub 2021 Jan 7. PMID 33411058
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181202&StudyName=A%20Study%20Of%20The%20Efficacy%20And%20Safety%20Of%20Sunitinib%20In%20Patients%20With%20Advanced%20Well-Differentiated%20Pancreatic%20Neuroendocrine%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: "End of treatment" for outcome measures of ECOG-PS, EORTC QLQ-C30 and EORTC QLQ-GI NET 21 was up to "primary completion date" (PCD) only.
Groups:
- Sunitinib: Treatment Naive Cohort: Sunitinib 37.5 milligram (mg) capsule, orally once daily in each 28-day treatment cycle (up to a maximum of 64 cycles) until death, unacceptable toxicity, consent withdrawal or final analysis in treatment-naive participants.
- Sunitinib: Later-Line Cohort: Sunitinib 37.5 mg capsule, orally once daily in each 28-day treatment cycle (up to a maximum of 64 cycles) until death, unacceptable toxicity, consent withdrawal or final analysis in previously treated/later-line participants (participants who developed progressive disease on or after prior systemic therapy).
Period: Overall Study
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Started | 61 | 45
Completed | 0 | 0
Not Completed | 61 | 45
Not completed — Lost to Follow-up | 8 | 2
Not completed — Death | 19 | 28
Not completed — Other | 0 | 4
Not completed — Sponsor's Decision | 30 | 11
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were enrolled into the study regardless of whether participants received study drug or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort | Total
Number analyzed (Participants) | 61 | 45 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (8.9) | 53.5 (9.1) | 54.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 12 | 43
  Male | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Investigator Assessment
Description: Investigator assessed PFS was defined as the time (in months) from the date of enrollment in study to the date of first documented objective tumor progression or death (due to any cause), whichever occurs first. PFS calculated as (first event date minus date of enrollment plus 1)/30.4. If progression or death was not observed, the participant was censored at the date of the participant's last progression-free tumor assessment prior to the study cut-off date. Progression as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 criteria was defined as: greater than or equal to (>=) 20 percent increase in sum of longest diameter (LD) of target lesions taking as a reference the smallest sum of the LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: FAS included all participants who were enrolled into the study regardless of whether participants received study drug or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
months | 13.2 [7.4 to 16.8] | 13.0 [9.2 to 20.4]

2. Secondary Outcome: Progression-Free Survival (PFS): Independent Radiological Review (IRR) Assessment
Description: IRR assessed PFS was defined as the time (in months) from the date of enrollment in study until the date of first documented objective tumor progression or death (due to any cause), whichever occurs first. PFS calculated as (first event date minus date of enrollment plus 1)/30.4. If progression or death was not observed, the participant was censored at the date of the participant's last progression-free tumor assessment prior to the study cut-off date. Progression as per RECIST 1.0 criteria was defined as: >=20 percent increase in sum of LD of target lesions taking as a reference the smallest sum of the LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
months | 11.1 [5.5 to 16.7] | 9.5 [7.4 to 18.4]

3. Secondary Outcome: Time to Tumor Progression (TTP): Investigator Assessment
Description: Investigator assessed TTP was defined as the time (in months) from the date of enrollment in study until the date of first documentation of objective tumor progression. TTP calculated as (first event date minus date of enrollment plus 1)/30.4. Progression as per RECIST 1.0 was defined as >=20 percent increase in sum of LD of target lesions taking as a reference the smallest sum of the LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until first documented tumor progression (up to 1226 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
months | 14.8 [7.5 to 16.8] | 14.5 [9.2 to 20.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from date of enrollment in study to the date of death due to any cause. If death was not observed, the participant was censored at the earliest of the last date the participant was known to be alive or the end of study. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until death or end of study (up to 1939 days)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Months | NA [41.7 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants who died. | 37.9 [22.9 to 56.1]

5. Secondary Outcome: Percentage of Participants With Objective Response (OR): Investigator Assessment
Description: Investigator assessed OR in participants was defined as having a complete response (CR) or partial response (PR) according to RECIST 1.0 and sustained for at least 4 weeks. CR was defined as disappearance of all target and non-target lesions. PR was defined as >=30 percent decrease in the sum of the LD of the target lesions taking as a reference the baseline sum LD. Percentage of participants with investigator assessed OR were reported.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
percentage of participants | 21.3 [11.9 to 33.7] | 28.9 [16.4 to 44.3]

6. Secondary Outcome: Duration of Response (DOR): Investigator Assessment
Description: Investigator assessed DOR was defined as the time (in months) from the date of first documented objective tumor response (CR or PR), that was subsequently confirmed, to the first documented objective tumor progression or death due to any cause, whichever occurred first. According to RECIST 1.0, CR was defined as disappearance of all target and non-target lesions. PR was defined as >=30 percent decrease in the sum of the LD of the target lesions taking as a reference the baseline sum LD. Progression as per RECIST version 1.0 was defined as >=20 percent increase in sum of LD of target lesions taking as a reference the smallest sum of the LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: Analysis was performed on only those participants who had objective response as per investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 13 | 13
months | 19.1 [10.1 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events. | 14.7 [5.5 to 21.9]

7. Secondary Outcome: Time to Tumor Response (TTR): Investigator Assessment
Description: Investigator assessed TTR was defined as the time (in months) from date of enrollment in study until date of first documentation of objective tumor response (CR or PR) that was subsequently confirmed. TTR was calculated as (first response date minus the date of enrollment plus 1) divided by 30.4. As per RECIST 1.0, CR was defined as disappearance of all target and non-target lesions and PR was defined as >=30 percent decrease in the sum of the LD of the target lesions taking as a reference the baseline sum LD.
Time Frame: Baseline until first documented objective tumor response (up to 1226 days)
Population: Analysis was performed on only those participants who had objective response as per investigator assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 13 | 13
months | 3.8 [1.0 to 11.1] | 3.8 [1.0 to 9.3]

8. Secondary Outcome: Percentage of Participants With Objective Response (OR): Independent Radiological Review (IRR) Assessment
Description: IRR assessed OR in participants was defined as having a CR or PR according to Choi criteria and sustained for at least 4 weeks. According to Choi criteria, CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as a decrease of >=10 percent in tumor size or a decrease in tumor density (HU) of 15 percent or more on Computed tomography (CT) with no new lesions and no obvious progression of non-measurable disease. Percentage of participants with objective response were reported in this outcome measure.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
percentage of participants | 52.5 [39.3 to 65.4] | 55.6 [40.0 to 70.4]

9. Secondary Outcome: Duration of Response (DOR): Independent Radiological Review (IRR) Assessment
Description: IRR assessed DOR was defined as the time (in months) from the date of first documented objective tumor response (CR or PR) that was subsequently confirmed to the first documented objective tumor progression or death due to any cause, whichever occurred first. According to Choi criteria, CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as a decrease of >=10 percent in tumor size or a decrease in tumor density (HU) of 15 percent or more on CT with no new lesions and no obvious progression of non-measurable disease.
Time Frame: Baseline until disease progression or death due to any cause (up to 1226 days)
Population: Analysis was performed on only those participants who had objective response as per IRR assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 32 | 25
months | NA [17.8 to NA] — Median and 95% CI was not estimable due to the small number of participants who encountered tumor progression or death. | 19.2 [15.7 to 35.9]

10. Secondary Outcome: Time to Tumor Response (TTR): Independent Radiological Review (IRR) Assessment
Description: IRR assessed TTR was defined as the time (in months) from date of enrollment in study until first documentation of objective tumor response (CR or PR) that was subsequently confirmed. TTR was calculated as (first response date minus the date of enrollment plus 1) divided by 30.4. According to Choi criteria, CR was defined as disappearance of all target and non-target lesions and no new lesions. PR was defined as a decrease of >=10 percent in tumor size or a decrease in tumor density (HU) of 15 percent or more on CT with no new lesions and no obvious progression of non-measurable disease.
Time Frame: Baseline until first documented objective tumor response (up to 1226 days)
Population: Analysis was performed on only those participants who had objective response as per IRR assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 32 | 25
months | 1.0 [0.8 to 7.3] | 1.0 [0.9 to 3.7]

11. Secondary Outcome: Percentage of Participants With Chromogranin A (CgA) Response
Description: CgA response in participants was defined as having confirmed CgA CR or CgA PR, relative to the population with an elevated baseline CgA value in the blood. CgA CR was defined as decrease from a high baseline value of CgA in the blood to one that fell within the normal range. CgA PR was defined as a decrease of greater than or equal to 50 percent from a high baseline value of CgA. Normal baseline value of CgA in blood was 39.0 ng/mL. Confirmed responses were those that persisted for at least 4 weeks after initial documentation of response. Blood levels of CgA were assessed and percentage of participants with CgA response were reported.
Time Frame: Baseline until CgA response or death due to any cause (up to 1226 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
percentage of participants | 16.4 [9.6 to 32.5] | 11.1 [4.0 to 25.6]

12. Secondary Outcome: Quality of Life Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 is a cancer-specific instrument with 30 questions to assess the participant quality of life. First 28 questions used for evaluating 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea and vomiting, pain) and other single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Each question was assessed on 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much); high score represented high level of symptomatology/problem. Last 2 questions used for evaluating global health status (GHS)/quality of life. Each question was assessed on 7-point scale (1=very poor to 7=excellent). Scores averaged, transformed to 0-100 scale; higher score=better level of functioning.
Time Frame: Day 1 of Cycle 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 27, 28, 29, 30, 31, 32, 33, 34, 35, 36, 37, 38, 39, 40, 41, 42, 43, End of treatment (up to maximum duration of 1226 days)
Population: FAS included all participants who were enrolled into the study regardless of whether participants received study drug or not. Here, "0 participants" in the "number analyzed" field signifies none of the participants were evaluable in the given group at this time point, hence data was not reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
units on a scale
  Global health status:Cycle 1: number analyzed (Participants) | 61 | 43
  Global health status:Cycle 1 | 71.31 (21.111) | 66.09 (20.282)
  Global health status: Cycle 2: number analyzed (Participants) | 56 | 41
  Global health status: Cycle 2 | 69.94 (19.311) | 65.45 (20.880)
  Global health status: Cycle 3: number analyzed (Participants) | 55 | 40
  Global health status: Cycle 3 | 70.30 (21.502) | 60.83 (26.768)
  Global health status: Cycle 4: number analyzed (Participants) | 50 | 38
  Global health status: Cycle 4 | 70.00 (21.429) | 61.84 (25.010)
  Global health status: Cycle 5: number analyzed (Participants) | 47 | 34
  Global health status: Cycle 5 | 69.15 (19.421) | 65.93 (24.306)
  Global health status: Cycle 6: number analyzed (Participants) | 43 | 31
  Global health status: Cycle 6 | 68.41 (18.053) | 65.32 (20.310)
  Global health status: Cycle 7: number analyzed (Participants) | 39 | 29
  Global health status: Cycle 7 | 68.38 (21.132) | 61.21 (24.016)
  Global health status: Cycle 8: number analyzed (Participants) | 37 | 25
  Global health status: Cycle 8 | 70.05 (17.062) | 65.33 (20.649)
  Global health status: Cycle 9: number analyzed (Participants) | 35 | 26
  Global health status: Cycle 9 | 66.90 (20.058) | 65.71 (20.045)
  Global health status: Cycle 10: number analyzed (Participants) | 35 | 23
  Global health status: Cycle 10 | 68.10 (20.561) | 63.04 (18.434)
  Global health status: Cycle 11: number analyzed (Participants) | 35 | 24
  Global health status: Cycle 11 | 63.81 (21.384) | 66.67 (19.812)
  Global health status: Cycle 12: number analyzed (Participants) | 35 | 22
  Global health status: Cycle 12 | 65.71 (22.395) | 64.77 (22.848)
  Global health status: Cycle 13: number analyzed (Participants) | 34 | 21
  Global health status: Cycle 13 | 67.89 (20.733) | 66.67 (19.365)
  Global health status: Cycle 14: number analyzed (Participants) | 31 | 19
  Global health status: Cycle 14 | 68.28 (20.797) | 57.89 (18.937)
  Global health status: Cycle 15: number analyzed (Participants) | 30 | 17
  Global health status: Cycle 15 | 66.67 (22.318) | 64.71 (21.757)
  Global health status: Cycle 16: number analyzed (Participants) | 27 | 16
  Global health status: Cycle 16 | 64.51 (21.005) | 67.19 (17.339)
  Global health status: Cycle 17: number analyzed (Participants) | 22 | 15
  Global health status: Cycle 17 | 62.50 (23.110) | 67.78 (15.706)
  Global health status: Cycle 18: number analyzed (Participants) | 17 | 14
  Global health status: Cycle 18 | 58.33 (24.826) | 70.83 (18.125)
  Global health status: Cycle 19: number analyzed (Participants) | 12 | 14
  Global health status: Cycle 19 | 54.86 (24.736) | 66.67 (20.672)
  Global health status: Cycle 20: number analyzed (Participants) | 11 | 13
  Global health status: Cycle 20 | 55.30 (25.893) | 64.74 (17.398)
  Global health status: Cycle 21: number analyzed (Participants) | 11 | 12
  Global health status: Cycle 21 | 55.30 (23.650) | 65.28 (18.407)
  Global health status: Cycle 22: number analyzed (Participants) | 11 | 11
  Global health status: Cycle 22 | 56.06 (23.889) | 62.88 (27.224)
  Global health status: Cycle 23: number analyzed (Participants) | 11 | 10
  Global health status: Cycle 23 | 56.82 (24.386) | 59.17 (20.953)
  Global health status: Cycle 24: number analyzed (Participants) | 10 | 10
  Global health status: Cycle 24 | 50.00 (23.570) | 60.83 (19.265)
  Global health status: Cycle 25: number analyzed (Participants) | 10 | 8
  Global health status: Cycle 25 | 51.67 (19.954) | 61.46 (16.022)
  Global health status: Cycle 26: number analyzed (Participants) | 7 | 7
  Global health status: Cycle 26 | 50.00 (20.972) | 65.48 (13.968)
  Global health status: Cycle 27: number analyzed (Participants) | 6 | 8
  Global health status: Cycle 27 | 41.67 (12.910) | 61.46 (17.216)
  Global health status: Cycle 28: number analyzed (Participants) | 7 | 8
  Global health status: Cycle 28 | 44.05 (20.813) | 61.46 (16.022)
  Global health status: Cycle 29: number analyzed (Participants) | 5 | 7
  Global health status: Cycle 29 | 56.67 (19.003) | 63.10 (16.567)
  Global health status: Cycle 30: number analyzed (Participants) | 4 | 7
  Global health status: Cycle 30 | 52.08 (21.916) | 64.29 (14.996)
  Global health status: Cycle 31: number analyzed (Participants) | 2 | 7
  Global health status: Cycle 31 | 58.33 (11.785) | 60.71 (20.813)
  Global health status: Cycle 32: number analyzed (Participants) | 3 | 6
  Global health status: Cycle 32 | 61.11 (19.245) | 59.72 (15.290)
  Global health status: Cycle 33: number analyzed (Participants) | 3 | 6
  Global health status: Cycle 33 | 61.11 (12.729) | 55.56 (22.771)
  Global health status: Cycle 34: number analyzed (Participants) | 3 | 6
  Global health status: Cycle 34 | 58.33 (25.000) | 55.56 (20.861)
  Global health status: Cycle 35: number analyzed (Participants) | 2 | 6
  Global health status: Cycle 35 | 66.67 (23.570) | 61.11 (13.608)
  Global health status: Cycle 36: number analyzed (Participants) | 1 | 5
  Global health status: Cycle 36 | 83.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 58.33 (16.667)
  Global health status: Cycle 37: number analyzed (Participants) | 1 | 4
  Global health status: Cycle 37 | 83.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 58.33 (21.517)
  Global health status: Cycle 38: number analyzed (Participants) | 0 | 4
  Global health status: Cycle 38 |  | 58.33 (21.517)
  Global health status: Cycle 39: number analyzed (Participants) | 1 | 3
  Global health status: Cycle 39 | 83.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 50.00 (16.667)
  Global health status: Cycle 40: number analyzed (Participants) | 1 | 3
  Global health status: Cycle 40 | 83.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 50.00 (16.667)
  Global health status: Cycle 41: number analyzed (Participants) | 0 | 3
  Global health status: Cycle 41 |  | 50.00 (16.667)
  Global health status: Cycle 42: number analyzed (Participants) | 0 | 2
  Global health status: Cycle 42 |  | 45.83 (5.893)
  Global health status: Cycle 43: number analyzed (Participants) | 0 | 1
  Global health status: Cycle 43 |  | 50.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Global health status: EOT: number analyzed (Participants) | 33 | 30
  Global health status: EOT | 60.10 (22.318) | 50.00 (22.210)
  Physical Functioning: Cycle 1: number analyzed (Participants) | 61 | 44
  Physical Functioning: Cycle 1 | 90.38 (14.733) | 86.93 (12.677)
  Physical Functioning: Cycle 2: number analyzed (Participants) | 57 | 42
  Physical Functioning: Cycle 2 | 89.71 (10.988) | 86.51 (13.929)
  Physical Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Physical Functioning: Cycle 3 | 88.73 (12.886) | 85.00 (17.263)
  Physical Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Physical Functioning: Cycle 4 | 89.07 (10.412) | 83.68 (16.958)
  Physical Functioning: Cycle 5: number analyzed (Participants) | 47 | 34
  Physical Functioning: Cycle 5 | 88.23 (11.311) | 87.06 (17.519)
  Physical Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Physical Functioning: Cycle 6 | 87.91 (11.293) | 83.44 (18.924)
  Physical Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Physical Functioning: Cycle 7 | 86.24 (12.891) | 84.14 (15.473)
  Physical Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Physical Functioning: Cycle 8 | 85.23 (12.486) | 88.27 (11.102)
  Physical Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Physical Functioning: Cycle 9 | 84.00 (13.255) | 87.18 (14.474)
  Physical Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Physical Functioning: Cycle 10 | 86.67 (11.771) | 87.25 (15.943)
  Physical Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Physical Functioning: Cycle 11 | 84.19 (12.944) | 90.83 (10.552)
  Physical Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Physical Functioning: Cycle 12 | 84.38 (15.419) | 88.48 (11.489)
  Physical Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Physical Functioning: Cycle 13 | 87.45 (11.808) | 89.52 (10.016)
  Physical Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Physical Functioning: Cycle 14 | 86.67 (12.996) | 86.67 (10.423)
  Physical Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Physical Functioning: Cycle 15 | 85.33 (11.534) | 89.02 (11.041)
  Physical Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Physical Functioning: Cycle 16 | 83.70 (18.053) | 89.58 (10.319)
  Physical Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Physical Functioning: Cycle 17 | 82.42 (16.657) | 88.00 (9.155)
  Physical Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Physical Functioning: Cycle 18 | 82.35 (18.248) | 90.95 (8.516)
  Physical Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Physical Functioning: Cycle 19 | 75.00 (22.406) | 89.52 (9.324)
  Physical Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Physical Functioning: Cycle 20 | 74.55 (20.181) | 89.74 (8.439)
  Physical Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Physical Functioning: Cycle 21 | 75.15 (17.911) | 90.00 (7.785)
  Physical Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Physical Functioning: Cycle 22 | 77.58 (22.563) | 81.82 (24.782)
  Physical Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Physical Functioning: Cycle 23 | 77.73 (18.170) | 82.67 (14.470)
  Physical Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Physical Functioning: Cycle 24 | 72.67 (22.760) | 82.67 (14.807)
  Physical Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Physical Functioning: Cycle 25 | 74.67 (23.685) | 89.17 (10.653)
  Physical Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Physical Functioning: Cycle 26 | 66.67 (25.531) | 83.81 (13.801)
  Physical Functioning: Cycle 27): number analyzed (Participants) | 6 | 8
  Physical Functioning: Cycle 27) | 62.22 (27.217) | 85.83 (12.051)
  Physical Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Physical Functioning: Cycle 28 | 69.52 (21.381) | 87.50 (11.513)
  Physical Functioning: Cycle 29: number analyzed (Participants) | 6 | 7
  Physical Functioning: Cycle 29 | 80.00 (10.328) | 83.81 (15.803)
  Physical Functioning: Cycle 30: number analyzed (Participants) | 5 | 7
  Physical Functioning: Cycle 30 | 84.00 (3.651) | 84.76 (11.362)
  Physical Functioning: Cycle 31: number analyzed (Participants) | 3 | 7
  Physical Functioning: Cycle 31 | 77.78 (10.184) | 85.71 (13.569)
  Physical Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Physical Functioning: Cycle 32 | 84.44 (3.849) | 82.22 (10.037)
  Physical Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Physical Functioning: Cycle 33 | 73.33 (6.667) | 83.33 (10.954)
  Physical Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Physical Functioning: Cycle 34 | 64.44 (21.430) | 80.00 (12.649)
  Physical Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Physical Functioning: Cycle 35 | 70.00 (23.570) | 78.89 (12.939)
  Physical Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Physical Functioning: Cycle 36 | 86.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 80.00 (9.428)
  Physical Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Physical Functioning: Cycle 37 | 86.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 76.67 (3.849)
  Physical Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Physical Functioning: Cycle 38 |  | 75.00 (6.383)
  Physical Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Physical Functioning: Cycle 39 | 86.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 77.78 (3.849)
  Physical Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Physical Functioning: Cycle 40 | 93.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 71.11 (10.184)
  Physical Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Physical Functioning: Cycle 41 |  | 77.78 (10.184)
  Physical Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Physical Functioning: Cycle 42 |  | 80.00 (0.000)
  Physical Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Physical Functioning: Cycle 43 |  | 80.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Physical Functioning: EOT: number analyzed (Participants) | 33 | 30
  Physical Functioning: EOT | 76.16 (23.454) | 78.00 (19.191)
  Role Functioning: Cycle 1: number analyzed (Participants) | 60 | 44
  Role Functioning: Cycle 1 | 88.33 (20.424) | 85.61 (18.880)
  Role Functioning: Cycle 2: number analyzed (Participants) | 57 | 42
  Role Functioning: Cycle 2 | 85.67 (17.089) | 80.56 (25.214)
  Role Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Role Functioning: Cycle 3 | 85.15 (18.613) | 80.83 (25.473)
  Role Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Role Functioning: Cycle 4 | 84.67 (17.444) | 80.26 (23.841)
  Role Functioning: Cycle 5: number analyzed (Participants) | 47 | 34
  Role Functioning: Cycle 5 | 85.82 (19.343) | 82.35 (23.904)
  Role Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Role Functioning: Cycle 6 | 86.05 (16.639) | 79.57 (25.353)
  Role Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Role Functioning: Cycle 7 | 83.33 (21.965) | 81.03 (24.285)
  Role Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Role Functioning: Cycle 8 | 80.63 (19.049) | 85.33 (16.887)
  Role Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Role Functioning: Cycle 9 | 76.19 (22.968) | 80.77 (22.945)
  Role Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Role Functioning: Cycle 10 | 82.86 (18.737) | 83.33 (23.028)
  Role Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Role Functioning: Cycle 11 | 79.52 (22.537) | 86.11 (18.822)
  Role Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Role Functioning: Cycle 12 | 79.52 (20.246) | 84.85 (19.182)
  Role Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Role Functioning: Cycle 13 | 82.35 (19.219) | 84.13 (17.059)
  Role Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Role Functioning: Cycle 14 | 81.72 (20.346) | 79.82 (19.704)
  Role Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Role Functioning: Cycle 15 | 77.22 (22.946) | 77.45 (22.777)
  Role Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Role Functioning: Cycle 16 | 77.16 (24.956) | 84.38 (15.478)
  Role Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Role Functioning: Cycle 17 | 74.24 (24.520) | 82.22 (17.213)
  Role Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Role Functioning: Cycle 18 | 75.49 (28.332) | 84.52 (16.621)
  Role Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Role Functioning: Cycle 19 | 66.67 (26.591) | 79.76 (20.856)
  Role Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Role Functioning: Cycle 20 | 69.70 (27.707) | 80.77 (19.059)
  Role Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Role Functioning: Cycle 21 | 68.18 (27.340) | 79.17 (23.704)
  Role Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Role Functioning: Cycle 22 | 68.18 (29.302) | 71.21 (29.899)
  Role Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Role Functioning: Cycle 23 | 63.64 (30.567) | 71.67 (24.907)
  Role Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Role Functioning: Cycle 24 | 60.00 (27.442) | 76.67 (22.498)
  Role Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Role Functioning: Cycle 25 | 58.33 (30.682) | 77.08 (23.465)
  Role Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Role Functioning: Cycle 26 | 57.14 (30.211) | 83.33 (16.667)
  Role Functioning: Cycle 27: number analyzed (Participants) | 6 | 8
  Role Functioning: Cycle 27 | 58.33 (36.132) | 77.08 (23.465)
  Role Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Role Functioning: Cycle 28 | 59.52 (18.898) | 79.17 (24.801)
  Role Functioning: Cycle 29: number analyzed (Participants) | 6 | 7
  Role Functioning: Cycle 29 | 75.00 (13.944) | 78.57 (24.934)
  Role Functioning: Cycle 30: number analyzed (Participants) | 5 | 7
  Role Functioning: Cycle 30 | 90.00 (14.907) | 76.19 (25.198)
  Role Functioning: Cycle 31: number analyzed (Participants) | 3 | 7
  Role Functioning: Cycle 31 | 83.33 (16.667) | 78.57 (24.934)
  Role Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Role Functioning: Cycle 32 | 94.44 (9.623) | 77.78 (20.184)
  Role Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Role Functioning: Cycle 33 | 88.89 (19.245) | 72.22 (25.092)
  Role Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Role Functioning: Cycle 34 | 72.22 (34.694) | 69.44 (30.581)
  Role Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Role Functioning: Cycle 35 | 75.00 (35.355) | 72.22 (25.092)
  Role Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Role Functioning: Cycle 36 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 73.33 (19.003)
  Role Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Role Functioning: Cycle 37 | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 70.83 (28.464)
  Role Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Role Functioning: Cycle 38 |  | 66.67 (27.217)
  Role Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Role Functioning: Cycle 39 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 55.56 (19.245)
  Role Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Role Functioning: Cycle 40 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 55.56 (9.623)
  Role Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Role Functioning: Cycle 41 |  | 55.56 (19.245)
  Role Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Role Functioning: Cycle 42 |  | 66.67 (0.000)
  Role Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Role Functioning: Cycle 43 |  | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Role Functioning: EOT: number analyzed (Participants) | 33 | 30
  Role Functioning: EOT | 70.71 (26.031) | 65.56 (36.075)
  Emotional Functioning: Cycle 1: number analyzed (Participants) | 61 | 43
  Emotional Functioning: Cycle 1 | 80.19 (18.644) | 76.23 (18.238)
  Emotional Functioning: Cycle 2: number analyzed (Participants) | 57 | 41
  Emotional Functioning: Cycle 2 | 84.31 (17.619) | 77.64 (17.021)
  Emotional Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Emotional Functioning: Cycle 3 | 82.53 (18.792) | 73.96 (24.401)
  Emotional Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Emotional Functioning: Cycle 4 | 82.67 (16.906) | 77.41 (22.167)
  Emotional Functioning: Cycle 5: number analyzed (Participants) | 47 | 34
  Emotional Functioning: Cycle 5 | 82.09 (18.632) | 79.66 (21.141)
  Emotional Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Emotional Functioning: Cycle 6 | 82.17 (17.871) | 73.92 (24.696)
  Emotional Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Emotional Functioning: Cycle 7 | 80.56 (21.059) | 73.56 (26.075)
  Emotional Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Emotional Functioning: Cycle 8 | 80.63 (21.877) | 76.00 (18.991)
  Emotional Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Emotional Functioning: Cycle 9 | 80.24 (19.812) | 76.92 (18.304)
  Emotional Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Emotional Functioning: Cycle 10 | 81.27 (19.818) | 76.45 (21.998)
  Emotional Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Emotional Functioning: Cycle 11 | 79.76 (19.311) | 75.46 (20.587)
  Emotional Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Emotional Functioning: Cycle 12 | 78.10 (23.052) | 75.76 (22.700)
  Emotional Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Emotional Functioning: Cycle 13 | 77.45 (22.429) | 77.38 (19.211)
  Emotional Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Emotional Functioning: Cycle 14 | 78.49 (20.387) | 75.00 (24.375)
  Emotional Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Emotional Functioning: Cycle 15 | 80.00 (21.173) | 74.51 (23.839)
  Emotional Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Emotional Functioning: Cycle 16 | 82.10 (22.133) | 75.00 (24.343)
  Emotional Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Emotional Functioning: Cycle 17 | 79.92 (23.522) | 79.44 (19.382)
  Emotional Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Emotional Functioning: Cycle 18 | 78.92 (23.592) | 76.19 (25.499)
  Emotional Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Emotional Functioning: Cycle 19 | 73.61 (28.611) | 73.81 (25.288)
  Emotional Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Emotional Functioning: Cycle 20 | 71.21 (29.666) | 78.85 (25.823)
  Emotional Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Emotional Functioning: Cycle 21 | 76.52 (28.824) | 75.00 (25.624)
  Emotional Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Emotional Functioning: Cycle 22 | 75.76 (30.834) | 78.03 (22.445)
  Emotional Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Emotional Functioning: Cycle 23 | 74.24 (30.834) | 75.00 (27.778)
  Emotional Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Emotional Functioning: Cycle 24 | 71.67 (28.921) | 76.67 (22.153)
  Emotional Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Emotional Functioning: Cycle 25 | 65.83 (33.206) | 66.67 (29.881)
  Emotional Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Emotional Functioning: Cycle 26 | 71.43 (34.979) | 77.38 (17.156)
  Emotional Functioning: Cycle 27: number analyzed (Participants) | 6 | 8
  Emotional Functioning: Cycle 27 | 56.94 (32.667) | 68.75 (29.124)
  Emotional Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Emotional Functioning: Cycle 28 | 65.48 (34.166) | 68.75 (29.463)
  Emotional Functioning: Cycle 29: number analyzed (Participants) | 5 | 7
  Emotional Functioning: Cycle 29 | 68.33 (29.698) | 71.43 (31.127)
  Emotional Functioning: Cycle 30: number analyzed (Participants) | 4 | 7
  Emotional Functioning: Cycle 30 | 72.92 (29.950) | 70.24 (31.497)
  Emotional Functioning: Cycle 31: number analyzed (Participants) | 2 | 7
  Emotional Functioning: Cycle 31 | 45.83 (17.678) | 72.62 (26.227)
  Emotional Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Emotional Functioning: Cycle 32 | 69.44 (29.266) | 69.44 (33.610)
  Emotional Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Emotional Functioning: Cycle 33 | 77.78 (19.245) | 70.83 (27.764)
  Emotional Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Emotional Functioning: Cycle 34 | 66.67 (33.333) | 66.67 (34.561)
  Emotional Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Emotional Functioning: Cycle 35 | 83.33 (23.570) | 68.06 (33.918)
  Emotional Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Emotional Functioning: Cycle 36 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 71.67 (31.513)
  Emotional Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Emotional Functioning: Cycle 37 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 77.08 (35.600)
  Emotional Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Emotional Functioning: Cycle 38 |  | 70.83 (42.219)
  Emotional Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Emotional Functioning: Cycle 39 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 63.89 (48.829)
  Emotional Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Emotional Functioning: Cycle 40 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 66.67 (38.188)
  Emotional Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Emotional Functioning: Cycle 41 |  | 58.33 (41.667)
  Emotional Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Emotional Functioning: Cycle 42 |  | 54.17 (64.818)
  Emotional Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Emotional Functioning: Cycle 43 |  | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Emotional Functioning: EOT: number analyzed (Participants) | 33 | 30
  Emotional Functioning: EOT | 67.17 (23.748) | 66.94 (27.024)
  Cognitive Functioning: Cycle 1: number analyzed (Participants) | 61 | 43
  Cognitive Functioning: Cycle 1 | 90.16 (15.329) | 88.76 (15.310)
  Cognitive Functioning: Cycle 2: number analyzed (Participants) | 57 | 41
  Cognitive Functioning: Cycle 2 | 88.89 (15.537) | 89.43 (13.310)
  Cognitive Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Cognitive Functioning: Cycle 3 | 89.09 (15.119) | 87.50 (19.882)
  Cognitive Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Cognitive Functioning: Cycle 4 | 89.67 (12.993) | 87.72 (15.346)
  Cognitive Functioning: Cycle 5: number analyzed (Participants) | 47 | 34
  Cognitive Functioning: Cycle 5 | 88.65 (15.583) | 85.29 (22.385)
  Cognitive Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Cognitive Functioning: Cycle 6 | 89.53 (15.006) | 82.80 (25.993)
  Cognitive Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Cognitive Functioning: Cycle 7 | 89.74 (14.618) | 85.06 (20.091)
  Cognitive Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Cognitive Functioning: Cycle 8 | 87.39 (13.836) | 83.33 (21.517)
  Cognitive Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Cognitive Functioning: Cycle 9 | 88.10 (16.455) | 85.26 (20.181)
  Cognitive Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Cognitive Functioning: Cycle 10 | 88.10 (13.750) | 83.33 (21.320)
  Cognitive Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Cognitive Functioning: Cycle 11 | 86.67 (16.068) | 86.11 (17.492)
  Cognitive Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Cognitive Functioning: Cycle 12 | 86.67 (13.886) | 86.36 (18.993)
  Cognitive Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Cognitive Functioning: Cycle 13 | 87.25 (15.922) | 85.71 (19.211)
  Cognitive Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Cognitive Functioning: Cycle 14 | 88.71 (13.185) | 77.19 (22.368)
  Cognitive Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Cognitive Functioning: Cycle 15 | 88.33 (12.495) | 80.39 (27.154)
  Cognitive Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Cognitive Functioning: Cycle 16 | 88.27 (12.067) | 80.21 (24.509)
  Cognitive Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Cognitive Functioning: Cycle 17 | 89.39 (12.112) | 84.44 (20.380)
  Cognitive Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Cognitive Functioning: Cycle 18 | 88.24 (14.148) | 79.76 (24.615)
  Cognitive Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Cognitive Functioning: Cycle 19 | 88.89 (12.975) | 78.57 (24.832)
  Cognitive Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Cognitive Functioning: Cycle 20 | 90.91 (11.459) | 82.05 (24.964)
  Cognitive Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Cognitive Functioning: Cycle 21 | 89.39 (11.237) | 76.39 (26.071)
  Cognitive Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Cognitive Functioning: Cycle 22 | 86.36 (12.513) | 81.82 (20.350)
  Cognitive Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Cognitive Functioning: Cycle 23 | 84.85 (11.677) | 76.67 (27.442)
  Cognitive Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Cognitive Functioning: Cycle 24 | 85.00 (16.574) | 81.67 (19.954)
  Cognitive Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Cognitive Functioning: Cycle 25 | 81.67 (18.342) | 75.00 (25.198)
  Cognitive Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Cognitive Functioning: Cycle 26 | 85.71 (20.250) | 85.71 (17.817)
  Cognitive Functioning: Cycle 27: number analyzed (Participants) | 6 | 8
  Cognitive Functioning: Cycle 27 | 75.00 (20.412) | 77.08 (25.099)
  Cognitive Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Cognitive Functioning: Cycle 28 | 76.19 (18.898) | 72.92 (29.463)
  Cognitive Functioning: Cycle 29: number analyzed (Participants) | 5 | 7
  Cognitive Functioning: Cycle 29 | 76.67 (14.907) | 78.57 (26.726)
  Cognitive Functioning: Cycle 30: number analyzed (Participants) | 4 | 7
  Cognitive Functioning: Cycle 30 | 75.00 (16.667) | 76.19 (31.706)
  Cognitive Functioning: Cycle 31: number analyzed (Participants) | 2 | 7
  Cognitive Functioning: Cycle 31 | 83.33 (23.570) | 73.81 (31.706)
  Cognitive Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Cognitive Functioning: Cycle 32 | 83.33 (16.667) | 69.44 (32.347)
  Cognitive Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Cognitive Functioning: Cycle 33 | 88.89 (19.245) | 69.44 (26.701)
  Cognitive Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Cognitive Functioning: Cycle 34 | 77.78 (9.623) | 66.67 (34.960)
  Cognitive Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Cognitive Functioning: Cycle 35 | 100.00 (0.000) | 75.00 (27.386)
  Cognitive Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Cognitive Functioning: Cycle 36 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 73.33 (34.561)
  Cognitive Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Cognitive Functioning: Cycle 37 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 75.00 (39.675)
  Cognitive Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Cognitive Functioning: Cycle 38 |  | 70.83 (47.871)
  Cognitive Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Cognitive Functioning: Cycle 39 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 72.22 (34.694)
  Cognitive Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Cognitive Functioning: Cycle 40 | 83.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 61.11 (34.694)
  Cognitive Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Cognitive Functioning: Cycle 41 |  | 61.11 (41.944)
  Cognitive Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Cognitive Functioning: Cycle 42 |  | 50.00 (70.711)
  Cognitive Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Cognitive Functioning: Cycle 43 |  | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Cognitive Functioning: EOT: number analyzed (Participants) | 33 | 30
  Cognitive Functioning: EOT | 83.33 (17.180) | 78.33 (23.631)
  Social Functioning: Cycle 1: number analyzed (Participants) | 61 | 43
  Social Functioning: Cycle 1 | 80.87 (23.734) | 79.46 (25.675)
  Social Functioning: Cycle 2: number analyzed (Participants) | 57 | 41
  Social Functioning: Cycle 2 | 83.04 (20.288) | 82.93 (20.578)
  Social Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Social Functioning: Cycle 3 | 79.09 (23.399) | 77.08 (26.335)
  Social Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Social Functioning: Cycle 4 | 81.67 (21.626) | 79.82 (25.160)
  Social Functioning: Cycle 5: number analyzed (Participants) | 47 | 34
  Social Functioning: Cycle 5 | 80.85 (21.697) | 79.41 (26.291)
  Social Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Social Functioning: Cycle 6 | 80.23 (28.232) | 77.42 (28.398)
  Social Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Social Functioning: Cycle 7 | 80.34 (22.579) | 83.91 (27.271)
  Social Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Social Functioning: Cycle 8 | 78.83 (21.748) | 80.00 (25.909)
  Social Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Social Functioning: Cycle 9 | 77.62 (24.234) | 82.05 (23.534)
  Social Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Social Functioning: Cycle 10 | 81.43 (20.119) | 76.81 (26.939)
  Social Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Social Functioning: Cycle 11 | 76.19 (23.321) | 81.25 (26.151)
  Social Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Social Functioning: Cycle 12 | 75.71 (25.030) | 81.82 (27.172)
  Social Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Social Functioning: Cycle 13 | 77.94 (25.859) | 84.92 (21.670)
  Social Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Social Functioning: Cycle 14 | 81.18 (20.968) | 79.82 (29.700)
  Social Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Social Functioning: Cycle 15 | 76.67 (19.865) | 74.51 (31.797)
  Social Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Social Functioning: Cycle 16 | 75.93 (24.167) | 77.08 (25.000)
  Social Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Social Functioning: Cycle 17 | 75.00 (25.066) | 75.56 (25.871)
  Social Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Social Functioning: Cycle 18 | 76.47 (27.041) | 82.14 (28.090)
  Social Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Social Functioning: Cycle 19 | 72.22 (24.958) | 77.38 (26.640)
  Social Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Social Functioning: Cycle 20 | 75.76 (30.151) | 83.33 (21.517)
  Social Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Social Functioning: Cycle 21 | 71.21 (28.955) | 81.94 (26.071)
  Social Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Social Functioning: Cycle 22 | 69.70 (33.181) | 75.76 (30.151)
  Social Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Social Functioning: Cycle 23 | 71.21 (30.814) | 78.33 (31.476)
  Social Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Social Functioning: Cycle 24 | 63.33 (32.203) | 76.67 (30.631)
  Social Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Social Functioning: Cycle 25 | 70.00 (39.126) | 66.67 (34.503)
  Social Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Social Functioning: Cycle 26 | 61.90 (34.311) | 88.10 (15.853)
  Social Functioning: Cycle 27: number analyzed (Participants) | 6 | 8
  Social Functioning: Cycle 27 | 58.33 (32.914) | 70.83 (33.034)
  Social Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Social Functioning: Cycle 28 | 73.81 (38.318) | 77.08 (28.084)
  Social Functioning: Cycle 29: number analyzed (Participants) | 5 | 7
  Social Functioning: Cycle 29 | 80.00 (18.257) | 71.43 (34.311)
  Social Functioning: Cycle 30: number analyzed (Participants) | 4 | 7
  Social Functioning: Cycle 30 | 75.00 (31.914) | 69.05 (36.551)
  Social Functioning: Cycle 31: number analyzed (Participants) | 2 | 7
  Social Functioning: Cycle 31 | 66.67 (47.140) | 71.43 (35.635)
  Social Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 32 | 77.78 (19.245) | 66.67 (36.515)
  Social Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 33 | 66.67 (0.000) | 69.44 (30.581)
  Social Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 34 | 66.67 (0.000) | 63.89 (37.143)
  Social Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Social Functioning: Cycle 35 | 66.67 (23.570) | 72.22 (37.515)
  Social Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Social Functioning: Cycle 36 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 53.33 (36.132)
  Social Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Social Functioning: Cycle 37 | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 58.33 (41.944)
  Social Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Social Functioning: Cycle 38 |  | 66.67 (36.004)
  Social Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Social Functioning: Cycle 39 | 100.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.44 (38.490)
  Social Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Social Functioning: Cycle 40 | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 61.11 (38.490)
  Social Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Social Functioning: Cycle 41 |  | 44.44 (25.459)
  Social Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Social Functioning: Cycle 42 |  | 41.67 (35.355)
  Social Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Social Functioning: Cycle 43 |  | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Social Functioning: EOT: number analyzed (Participants) | 33 | 30
  Social Functioning: EOT | 73.74 (25.355) | 65.00 (29.148)
  Fatigue: Cycle 1: number analyzed (Participants) | 61 | 44
  Fatigue: Cycle 1 | 21.49 (20.374) | 29.42 (17.835)
  Fatigue: Cycle 2: number analyzed (Participants) | 57 | 42
  Fatigue: Cycle 2 | 24.37 (17.995) | 29.10 (19.001)
  Fatigue: Cycle 3: number analyzed (Participants) | 55 | 40
  Fatigue: Cycle 3 | 26.46 (19.303) | 30.28 (22.644)
  Fatigue: Cycle 4: number analyzed (Participants) | 50 | 38
  Fatigue: Cycle 4 | 24.00 (18.424) | 29.53 (24.133)
  Fatigue: Cycle 5: number analyzed (Participants) | 47 | 34
  Fatigue: Cycle 5 | 26.00 (17.069) | 27.61 (23.865)
  Fatigue: Cycle 6: number analyzed (Participants) | 43 | 31
  Fatigue: Cycle 6 | 25.32 (17.029) | 29.93 (25.526)
  Fatigue: Cycle 7: number analyzed (Participants) | 39 | 29
  Fatigue: Cycle 7 | 26.78 (21.284) | 28.35 (24.232)
  Fatigue: Cycle 8: number analyzed (Participants) | 37 | 25
  Fatigue: Cycle 8 | 27.63 (17.297) | 23.11 (18.681)
  Fatigue: Cycle 9: number analyzed (Participants) | 35 | 26
  Fatigue: Cycle 9 | 26.35 (20.182) | 22.22 (20.608)
  Fatigue: Cycle 10: number analyzed (Participants) | 35 | 23
  Fatigue: Cycle 10 | 26.03 (19.975) | 24.64 (23.914)
  Fatigue: Cycle 11: number analyzed (Participants) | 35 | 24
  Fatigue: Cycle 11 | 27.94 (18.548) | 22.45 (20.624)
  Fatigue: Cycle 12: number analyzed (Participants) | 35 | 22
  Fatigue: Cycle 12 | 26.35 (20.001) | 22.22 (23.256)
  Fatigue: Cycle 13: number analyzed (Participants) | 34 | 21
  Fatigue: Cycle 13 | 25.16 (19.012) | 18.52 (15.045)
  Fatigue: Cycle 14: number analyzed (Participants) | 31 | 19
  Fatigue: Cycle 14 | 24.73 (19.183) | 24.56 (20.813)
  Fatigue: Cycle 15: number analyzed (Participants) | 30 | 17
  Fatigue: Cycle 15 | 24.07 (20.443) | 24.84 (24.066)
  Fatigue: Cycle 16: number analyzed (Participants) | 27 | 16
  Fatigue: Cycle 16 | 27.16 (23.937) | 22.92 (17.902)
  Fatigue: Cycle 17: number analyzed (Participants) | 22 | 15
  Fatigue: Cycle 17 | 28.28 (22.150) | 18.52 (18.144)
  Fatigue: Cycle 18: number analyzed (Participants) | 17 | 14
  Fatigue: Cycle 18 | 26.80 (22.243) | 22.22 (17.433)
  Fatigue: Cycle 19: number analyzed (Participants) | 12 | 14
  Fatigue: Cycle 19 | 34.26 (31.944) | 23.02 (20.191)
  Fatigue: Cycle 20: number analyzed (Participants) | 11 | 13
  Fatigue: Cycle 20 | 34.34 (26.036) | 22.22 (18.144)
  Fatigue: Cycle 21: number analyzed (Participants) | 11 | 12
  Fatigue: Cycle 21 | 34.34 (32.377) | 28.70 (21.429)
  Fatigue: Cycle 22: number analyzed (Participants) | 11 | 11
  Fatigue: Cycle 22 | 31.31 (28.029) | 30.30 (27.707)
  Fatigue: Cycle 23: number analyzed (Participants) | 11 | 10
  Fatigue: Cycle 23 | 39.39 (28.702) | 28.89 (25.229)
  Fatigue: Cycle 24: number analyzed (Participants) | 10 | 10
  Fatigue: Cycle 24 | 36.67 (32.309) | 28.89 (26.294)
  Fatigue: Cycle 25: number analyzed (Participants) | 10 | 8
  Fatigue: Cycle 25 | 40.00 (30.180) | 27.78 (21.414)
  Fatigue: Cycle 26: number analyzed (Participants) | 7 | 7
  Fatigue: Cycle 26 | 44.44 (27.962) | 22.22 (14.344)
  Fatigue: Cycle 27: number analyzed (Participants) | 6 | 8
  Fatigue: Cycle 27 | 50.00 (30.429) | 26.39 (22.954)
  Fatigue: Cycle 28: number analyzed (Participants) | 7 | 8
  Fatigue: Cycle 28 | 42.86 (28.276) | 30.56 (26.394)
  Fatigue: Cycle 29: number analyzed (Participants) | 6 | 7
  Fatigue: Cycle 29 | 35.19 (23.744) | 28.57 (21.138)
  Fatigue: Cycle 30: number analyzed (Participants) | 5 | 7
  Fatigue: Cycle 30 | 24.44 (18.257) | 31.75 (27.539)
  Fatigue: Cycle 31: number analyzed (Participants) | 3 | 7
  Fatigue: Cycle 31 | 22.22 (29.397) | 31.75 (29.696)
  Fatigue: Cycle 32: number analyzed (Participants) | 3 | 6
  Fatigue: Cycle 32 | 18.52 (23.130) | 35.19 (12.989)
  Fatigue: Cycle 33: number analyzed (Participants) | 3 | 6
  Fatigue: Cycle 33 | 22.22 (29.397) | 40.74 (20.688)
  Fatigue: Cycle 34: number analyzed (Participants) | 3 | 6
  Fatigue: Cycle 34 | 37.04 (35.717) | 40.74 (16.728)
  Fatigue: Cycle 35: number analyzed (Participants) | 2 | 6
  Fatigue: Cycle 35 | 33.33 (47.140) | 35.19 (16.355)
  Fatigue: Cycle 36: number analyzed (Participants) | 1 | 5
  Fatigue: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 40.00 (14.907)
  Fatigue: Cycle 37: number analyzed (Participants) | 1 | 4
  Fatigue: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 36.11 (21.033)
  Fatigue: Cycle 38: number analyzed (Participants) | 0 | 4
  Fatigue: Cycle 38 |  | 44.44 (27.217)
  Fatigue: Cycle 39: number analyzed (Participants) | 1 | 3
  Fatigue: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 51.85 (33.945)
  Fatigue: Cycle 40: number analyzed (Participants) | 1 | 3
  Fatigue: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 59.26 (33.945)
  Fatigue: Cycle 41: number analyzed (Participants) | 0 | 3
  Fatigue: Cycle 41 |  | 48.15 (23.130)
  Fatigue: Cycle 42: number analyzed (Participants) | 0 | 2
  Fatigue: Cycle 42 |  | 44.44 (31.427)
  Fatigue: Cycle 43: number analyzed (Participants) | 0 | 1
  Fatigue: Cycle 43 |  | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Fatigue: EOT: number analyzed (Participants) | 33 | 30
  Fatigue: EOT | 33.00 (23.812) | 40.56 (28.632)
  Nausea and Vomiting: Cycle 1: number analyzed (Participants) | 61 | 44
  Nausea and Vomiting: Cycle 1 | 6.56 (13.010) | 7.95 (17.420)
  Nausea and Vomiting: Cycle 2: number analyzed (Participants) | 57 | 42
  Nausea and Vomiting: Cycle 2 | 7.31 (12.206) | 7.14 (9.123)
  Nausea and Vomiting: Cycle 3: number analyzed (Participants) | 55 | 40
  Nausea and Vomiting: Cycle 3 | 7.27 (12.735) | 12.08 (19.967)
  Nausea and Vomiting: Cycle 4: number analyzed (Participants) | 50 | 38
  Nausea and Vomiting: Cycle 4 | 8.00 (13.569) | 4.39 (9.238)
  Nausea and Vomiting: Cycle 5: number analyzed (Participants) | 47 | 34
  Nausea and Vomiting: Cycle 5 | 6.38 (12.794) | 8.33 (14.935)
  Nausea and Vomiting: Cycle 6: number analyzed (Participants) | 43 | 31
  Nausea and Vomiting: Cycle 6 | 6.98 (12.189) | 6.99 (11.200)
  Nausea and Vomiting: Cycle 7: number analyzed (Participants) | 39 | 29
  Nausea and Vomiting: Cycle 7 | 6.41 (12.458) | 6.90 (15.117)
  Nausea and Vomiting: Cycle 8: number analyzed (Participants) | 37 | 25
  Nausea and Vomiting: Cycle 8 | 7.66 (15.513) | 3.33 (6.804)
  Nausea and Vomiting: Cycle 9: number analyzed (Participants) | 35 | 26
  Nausea and Vomiting: Cycle 9 | 9.05 (14.766) | 4.49 (10.064)
  Nausea and Vomiting: Cycle 10: number analyzed (Participants) | 35 | 23
  Nausea and Vomiting: Cycle 10 | 5.71 (12.088) | 4.35 (9.014)
  Nausea and Vomiting: Cycle 11: number analyzed (Participants) | 35 | 24
  Nausea and Vomiting: Cycle 11 | 4.76 (10.362) | 4.86 (9.167)
  Nausea and Vomiting: Cycle 12: number analyzed (Participants) | 35 | 22
  Nausea and Vomiting: Cycle 12 | 4.76 (11.835) | 6.06 (8.206)
  Nausea and Vomiting: Cycle 13: number analyzed (Participants) | 34 | 21
  Nausea and Vomiting: Cycle 13 | 3.43 (8.970) | 2.38 (5.976)
  Nausea and Vomiting: Cycle 14: number analyzed (Participants) | 31 | 19
  Nausea and Vomiting: Cycle 14 | 5.38 (9.988) | 6.14 (12.681)
  Nausea and Vomiting: Cycle 15: number analyzed (Participants) | 30 | 17
  Nausea and Vomiting: Cycle 15 | 7.22 (12.132) | 5.88 (16.605)
  Nausea and Vomiting: Cycle 16: number analyzed (Participants) | 27 | 16
  Nausea and Vomiting: Cycle 16 | 4.32 (9.906) | 3.13 (9.065)
  Nausea and Vomiting: Cycle 17: number analyzed (Participants) | 22 | 15
  Nausea and Vomiting: Cycle 17 | 3.03 (8.351) | 4.44 (9.894)
  Nausea and Vomiting: Cycle 18: number analyzed (Participants) | 17 | 14
  Nausea and Vomiting: Cycle 18 | 4.90 (11.433) | 1.19 (4.454)
  Nausea and Vomiting: Cycle 19: number analyzed (Participants) | 12 | 14
  Nausea and Vomiting: Cycle 19 | 4.17 (10.360) | 4.76 (12.105)
  Nausea and Vomiting: Cycle 20: number analyzed (Participants) | 11 | 13
  Nausea and Vomiting: Cycle 20 | 6.06 (15.407) | 1.28 (4.623)
  Nausea and Vomiting: Cycle 21: number analyzed (Participants) | 11 | 12
  Nausea and Vomiting: Cycle 21 | 4.55 (15.076) | 6.94 (19.408)
  Nausea and Vomiting: Cycle 22: number analyzed (Participants) | 11 | 11
  Nausea and Vomiting: Cycle 22 | 4.55 (15.076) | 9.09 (30.151)
  Nausea and Vomiting: Cycle 23: number analyzed (Participants) | 11 | 10
  Nausea and Vomiting: Cycle 23 | 6.06 (15.407) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 24: number analyzed (Participants) | 10 | 10
  Nausea and Vomiting: Cycle 24 | 6.67 (11.653) | 3.33 (7.027)
  Nausea and Vomiting: Cycle 25: number analyzed (Participants) | 10 | 8
  Nausea and Vomiting: Cycle 25 | 8.33 (14.164) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 26: number analyzed (Participants) | 7 | 7
  Nausea and Vomiting: Cycle 26 | 7.14 (8.909) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 27: number analyzed (Participants) | 6 | 8
  Nausea and Vomiting: Cycle 27 | 11.11 (20.184) | 4.17 (11.785)
  Nausea and Vomiting: Cycle 28: number analyzed (Participants) | 7 | 8
  Nausea and Vomiting: Cycle 28 | 9.52 (18.898) | 2.08 (5.893)
  Nausea and Vomiting: Cycle 29: number analyzed (Participants) | 6 | 7
  Nausea and Vomiting: Cycle 29 | 2.78 (6.804) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 30: number analyzed (Participants) | 5 | 7
  Nausea and Vomiting: Cycle 30 | 0.00 (0.000) | 2.38 (6.299)
  Nausea and Vomiting: Cycle 31: number analyzed (Participants) | 3 | 7
  Nausea and Vomiting: Cycle 31 | 0.00 (0.000) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 32: number analyzed (Participants) | 3 | 6
  Nausea and Vomiting: Cycle 32 | 5.56 (9.623) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 33: number analyzed (Participants) | 3 | 6
  Nausea and Vomiting: Cycle 33 | 22.22 (38.490) | 2.78 (6.804)
  Nausea and Vomiting: Cycle 34: number analyzed (Participants) | 3 | 6
  Nausea and Vomiting: Cycle 34 | 22.22 (38.490) | 8.33 (13.944)
  Nausea and Vomiting: Cycle 35: number analyzed (Participants) | 2 | 6
  Nausea and Vomiting: Cycle 35 | 16.67 (23.570) | 0.00 (0.000)
  Nausea and Vomiting: Cycle 36: number analyzed (Participants) | 1 | 5
  Nausea and Vomiting: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Nausea and Vomiting: Cycle 37: number analyzed (Participants) | 1 | 4
  Nausea and Vomiting: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 4.17 (8.333)
  Nausea and Vomiting: Cycle 38: number analyzed (Participants) | 0 | 4
  Nausea and Vomiting: Cycle 38 |  | 0.00 (0.000)
  Nausea and Vomiting: Cycle 39: number analyzed (Participants) | 1 | 3
  Nausea and Vomiting: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Nausea and Vomiting: Cycle 40: number analyzed (Participants) | 1 | 3
  Nausea and Vomiting: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Nausea and Vomiting: Cycle 41: number analyzed (Participants) | 0 | 3
  Nausea and Vomiting: Cycle 41 |  | 0.00 (0.000)
  Nausea and Vomiting: Cycle 42: number analyzed (Participants) | 0 | 2
  Nausea and Vomiting: Cycle 42 |  | 0.00 (0.000)
  Nausea and Vomiting: Cycle 43: number analyzed (Participants) | 0 | 1
  Nausea and Vomiting: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Nausea and Vomiting: EOT: number analyzed (Participants) | 33 | 30
  Nausea and Vomiting: EOT | 16.16 (21.844) | 12.78 (20.846)
  Pain: Cycle 1: number analyzed (Participants) | 61 | 44
  Pain: Cycle 1 | 16.39 (20.067) | 18.18 (18.958)
  Pain: Cycle 2: number analyzed (Participants) | 57 | 42
  Pain: Cycle 2 | 16.67 (18.094) | 19.05 (20.353)
  Pain: Cycle 3: number analyzed (Participants) | 55 | 40
  Pain: Cycle 3 | 15.76 (18.542) | 22.50 (27.099)
  Pain: Cycle 4: number analyzed (Participants) | 50 | 38
  Pain: Cycle 4 | 14.00 (15.922) | 23.25 (24.056)
  Pain: Cycle 5: number analyzed (Participants) | 47 | 34
  Pain: Cycle 5 | 15.96 (16.651) | 18.14 (22.235)
  Pain: Cycle 6: number analyzed (Participants) | 43 | 31
  Pain: Cycle 6 | 15.89 (17.041) | 20.43 (26.073)
  Pain: Cycle 7: number analyzed (Participants) | 39 | 29
  Pain: Cycle 7 | 20.09 (21.690) | 22.99 (22.893)
  Pain: Cycle 8: number analyzed (Participants) | 37 | 25
  Pain: Cycle 8 | 17.57 (17.099) | 14.67 (16.887)
  Pain: Cycle 9: number analyzed (Participants) | 35 | 26
  Pain: Cycle 9 | 20.48 (19.838) | 19.87 (19.447)
  Pain: Cycle 10: number analyzed (Participants) | 35 | 23
  Pain: Cycle 10 | 19.52 (22.682) | 18.84 (22.079)
  Pain: Cycle 11: number analyzed (Participants) | 35 | 24
  Pain: Cycle 11 | 19.05 (19.446) | 13.89 (18.169)
  Pain: Cycle 12: number analyzed (Participants) | 35 | 22
  Pain: Cycle 12 | 20.48 (22.172) | 16.67 (17.817)
  Pain: Cycle 13: number analyzed (Participants) | 34 | 21
  Pain: Cycle 13 | 17.16 (15.616) | 15.87 (20.053)
  Pain: Cycle 14: number analyzed (Participants) | 31 | 19
  Pain: Cycle 14 | 14.52 (17.074) | 21.05 (19.909)
  Pain: Cycle 15: number analyzed (Participants) | 30 | 17
  Pain: Cycle 15 | 15.00 (23.305) | 21.57 (24.127)
  Pain: Cycle 16: number analyzed (Participants) | 27 | 16
  Pain: Cycle 16 | 17.28 (21.917) | 15.63 (14.232)
  Pain: Cycle 17: number analyzed (Participants) | 22 | 15
  Pain: Cycle 17 | 18.94 (23.171) | 15.56 (17.213)
  Pain: Cycle 18: number analyzed (Participants) | 17 | 14
  Pain: Cycle 18 | 16.67 (22.048) | 10.71 (16.803)
  Pain: Cycle 19: number analyzed (Participants) | 12 | 14
  Pain: Cycle 19 | 26.39 (27.941) | 13.10 (16.249)
  Pain: Cycle 20: number analyzed (Participants) | 11 | 13
  Pain: Cycle 20 | 25.76 (27.247) | 12.82 (15.447)
  Pain: Cycle 21: number analyzed (Participants) | 11 | 12
  Pain: Cycle 21 | 25.76 (29.215) | 16.67 (21.320)
  Pain: Cycle 22: number analyzed (Participants) | 11 | 11
  Pain: Cycle 22 | 18.18 (26.304) | 21.21 (21.201)
  Pain: Cycle 23: number analyzed (Participants) | 11 | 10
  Pain: Cycle 23 | 21.21 (27.979) | 15.00 (22.839)
  Pain: Cycle 24: number analyzed (Participants) | 10 | 10
  Pain: Cycle 24 | 28.33 (26.117) | 20.00 (24.595)
  Pain: Cycle 25: number analyzed (Participants) | 10 | 8
  Pain: Cycle 25 | 26.67 (30.631) | 16.67 (19.920)
  Pain: Cycle 26: number analyzed (Participants) | 7 | 7
  Pain: Cycle 26 | 38.10 (40.500) | 16.67 (19.245)
  Pain: Cycle 27: number analyzed (Participants) | 6 | 8
  Pain: Cycle 27 | 47.22 (35.616) | 20.83 (21.362)
  Pain: Cycle 28: number analyzed (Participants) | 7 | 8
  Pain: Cycle 28 | 35.71 (33.923) | 22.92 (25.099)
  Pain: Cycle 29: number analyzed (Participants) | 6 | 7
  Pain: Cycle 29 | 19.44 (19.484) | 23.81 (26.972)
  Pain: Cycle 30: number analyzed (Participants) | 5 | 7
  Pain: Cycle 30 | 20.00 (21.731) | 19.05 (24.398)
  Pain: Cycle 31: number analyzed (Participants) | 3 | 7
  Pain: Cycle 31 | 16.67 (28.868) | 26.19 (23.288)
  Pain: Cycle 32: number analyzed (Participants) | 3 | 6
  Pain: Cycle 32 | 16.67 (28.868) | 27.78 (31.032)
  Pain: Cycle 33: number analyzed (Participants) | 3 | 6
  Pain: Cycle 33 | 16.67 (28.868) | 25.00 (25.276)
  Pain: Cycle 34: number analyzed (Participants) | 3 | 6
  Pain: Cycle 34 | 22.22 (38.490) | 27.78 (25.092)
  Pain: Cycle 35: number analyzed (Participants) | 2 | 6
  Pain: Cycle 35 | 25.00 (35.355) | 22.22 (13.608)
  Pain: Cycle 36: number analyzed (Participants) | 1 | 5
  Pain: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 20.00 (13.944)
  Pain: Cycle 37: number analyzed (Participants) | 1 | 4
  Pain: Cycle 37 | 16.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 29.17 (28.464)
  Pain: Cycle 38: number analyzed (Participants) | 0 | 4
  Pain: Cycle 38 |  | 29.17 (28.464)
  Pain: Cycle 39: number analyzed (Participants) | 1 | 3
  Pain: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 38.89 (25.459)
  Pain: Cycle 40: number analyzed (Participants) | 1 | 3
  Pain: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.44 (19.245)
  Pain: Cycle 41: number analyzed (Participants) | 0 | 3
  Pain: Cycle 41 |  | 55.56 (41.944)
  Pain: Cycle 42: number analyzed (Participants) | 0 | 2
  Pain: Cycle 42 |  | 33.33 (47.140)
  Pain: Cycle 43: number analyzed (Participants) | 0 | 1
  Pain: Cycle 43 |  | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Pain: EOT: number analyzed (Participants) | 33 | 30
  Pain: EOT | 23.74 (25.695) | 33.89 (32.009)
  Dyspnoea: Cycle 1: number analyzed (Participants) | 60 | 44
  Dyspnoea: Cycle 1 | 5.00 (12.003) | 7.58 (15.854)
  Dyspnoea: Cycle 2: number analyzed (Participants) | 57 | 42
  Dyspnoea: Cycle 2 | 7.02 (15.088) | 8.73 (18.123)
  Dyspnoea: Cycle 3: number analyzed (Participants) | 55 | 40
  Dyspnoea: Cycle 3 | 6.06 (12.975) | 9.17 (21.334)
  Dyspnoea: Cycle 4: number analyzed (Participants) | 50 | 38
  Dyspnoea: Cycle 4 | 6.00 (12.936) | 13.16 (21.280)
  Dyspnoea: Cycle 5: number analyzed (Participants) | 47 | 34
  Dyspnoea: Cycle 5 | 5.67 (14.445) | 10.78 (22.801)
  Dyspnoea: Cycle 6: number analyzed (Participants) | 43 | 31
  Dyspnoea: Cycle 6 | 6.98 (15.530) | 10.75 (24.925)
  Dyspnoea: Cycle 7: number analyzed (Participants) | 39 | 29
  Dyspnoea: Cycle 7 | 11.11 (22.076) | 10.34 (20.125)
  Dyspnoea: Cycle 8: number analyzed (Participants) | 37 | 25
  Dyspnoea: Cycle 8 | 15.32 (21.652) | 6.67 (13.608)
  Dyspnoea: Cycle 9: number analyzed (Participants) | 35 | 26
  Dyspnoea: Cycle 9 | 9.52 (20.725) | 5.13 (12.265)
  Dyspnoea: Cycle 10: number analyzed (Participants) | 35 | 23
  Dyspnoea: Cycle 10 | 9.52 (15.278) | 10.14 (21.165)
  Dyspnoea: Cycle 11: number analyzed (Participants) | 35 | 24
  Dyspnoea: Cycle 11 | 5.71 (12.746) | 9.72 (15.477)
  Dyspnoea: Cycle 12: number analyzed (Participants) | 35 | 22
  Dyspnoea: Cycle 12 | 8.57 (14.781) | 6.06 (13.159)
  Dyspnoea: Cycle 13: number analyzed (Participants) | 34 | 21
  Dyspnoea: Cycle 13 | 10.78 (15.829) | 12.70 (19.653)
  Dyspnoea: Cycle 14: number analyzed (Participants) | 31 | 19
  Dyspnoea: Cycle 14 | 9.68 (15.380) | 8.77 (15.080)
  Dyspnoea: Cycle 15: number analyzed (Participants) | 30 | 17
  Dyspnoea: Cycle 15 | 8.89 (14.993) | 9.80 (15.656)
  Dyspnoea: Cycle 16: number analyzed (Participants) | 27 | 16
  Dyspnoea: Cycle 16 | 6.17 (13.195) | 6.25 (13.437)
  Dyspnoea: Cycle 17: number analyzed (Participants) | 22 | 15
  Dyspnoea: Cycle 17 | 10.61 (15.891) | 6.67 (13.801)
  Dyspnoea: Cycle 18: number analyzed (Participants) | 17 | 14
  Dyspnoea: Cycle 18 | 7.84 (14.575) | 4.76 (12.105)
  Dyspnoea: Cycle 19: number analyzed (Participants) | 12 | 14
  Dyspnoea: Cycle 19 | 13.89 (17.164) | 4.76 (12.105)
  Dyspnoea: Cycle 20: number analyzed (Participants) | 11 | 13
  Dyspnoea: Cycle 20 | 6.06 (13.484) | 5.13 (12.518)
  Dyspnoea: Cycle 21: number analyzed (Participants) | 11 | 12
  Dyspnoea: Cycle 21 | 12.12 (16.817) | 8.33 (15.076)
  Dyspnoea: Cycle 22: number analyzed (Participants) | 11 | 11
  Dyspnoea: Cycle 22 | 9.09 (15.570) | 9.09 (15.570)
  Dyspnoea: Cycle 23: number analyzed (Participants) | 11 | 10
  Dyspnoea: Cycle 23 | 6.06 (13.484) | 13.33 (17.213)
  Dyspnoea: Cycle 24: number analyzed (Participants) | 10 | 10
  Dyspnoea: Cycle 24 | 6.67 (14.055) | 13.33 (17.213)
  Dyspnoea: Cycle 25: number analyzed (Participants) | 10 | 8
  Dyspnoea: Cycle 25 | 13.33 (23.307) | 8.33 (15.430)
  Dyspnoea: Cycle 26: number analyzed (Participants) | 7 | 7
  Dyspnoea: Cycle 26 | 9.52 (16.265) | 9.52 (16.265)
  Dyspnoea: Cycle 27: number analyzed (Participants) | 6 | 8
  Dyspnoea: Cycle 27 | 11.11 (27.217) | 8.33 (15.430)
  Dyspnoea: Cycle 28: number analyzed (Participants) | 7 | 8
  Dyspnoea: Cycle 28 | 19.05 (17.817) | 12.50 (17.252)
  Dyspnoea: Cycle 29: number analyzed (Participants) | 6 | 7
  Dyspnoea: Cycle 29 | 11.11 (27.217) | 19.05 (17.817)
  Dyspnoea: Cycle 30: number analyzed (Participants) | 5 | 7
  Dyspnoea: Cycle 30 | 6.67 (14.907) | 14.29 (17.817)
  Dyspnoea: Cycle 31: number analyzed (Participants) | 3 | 7
  Dyspnoea: Cycle 31 | 0.00 (0.000) | 9.52 (16.265)
  Dyspnoea: Cycle 32: number analyzed (Participants) | 3 | 6
  Dyspnoea: Cycle 32 | 11.11 (19.245) | 16.67 (27.889)
  Dyspnoea: Cycle 33: number analyzed (Participants) | 3 | 6
  Dyspnoea: Cycle 33 | 22.22 (38.490) | 11.11 (17.213)
  Dyspnoea: Cycle 34: number analyzed (Participants) | 3 | 6
  Dyspnoea: Cycle 34 | 11.11 (19.245) | 16.67 (27.889)
  Dyspnoea: Cycle 35: number analyzed (Participants) | 2 | 6
  Dyspnoea: Cycle 35 | 16.67 (23.570) | 11.11 (17.213)
  Dyspnoea: Cycle 36: number analyzed (Participants) | 1 | 5
  Dyspnoea: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 26.67 (27.889)
  Dyspnoea: Cycle 37: number analyzed (Participants) | 1 | 4
  Dyspnoea: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 8.33 (16.667)
  Dyspnoea: Cycle 38: number analyzed (Participants) | 0 | 4
  Dyspnoea: Cycle 38 |  | 8.33 (16.667)
  Dyspnoea: Cycle 39: number analyzed (Participants) | 1 | 3
  Dyspnoea: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Dyspnoea: Cycle 40: number analyzed (Participants) | 1 | 3
  Dyspnoea: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Dyspnoea: Cycle 41: number analyzed (Participants) | 0 | 3
  Dyspnoea: Cycle 41 |  | 0.00 (0.000)
  Dyspnoea: Cycle 42: number analyzed (Participants) | 0 | 2
  Dyspnoea: Cycle 42 |  | 16.67 (23.570)
  Dyspnoea: Cycle 43: number analyzed (Participants) | 0 | 1
  Dyspnoea: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Dyspnoea: EOT: number analyzed (Participants) | 33 | 30
  Dyspnoea: EOT | 14.14 (16.730) | 13.33 (24.132)
  Insomnia: Cycle 1: number analyzed (Participants) | 61 | 44
  Insomnia: Cycle 1 | 13.11 (20.438) | 25.76 (27.715)
  Insomnia: Cycle 2: number analyzed (Participants) | 57 | 42
  Insomnia: Cycle 2 | 9.36 (16.372) | 19.84 (23.350)
  Insomnia: Cycle 3: number analyzed (Participants) | 55 | 40
  Insomnia: Cycle 3 | 12.12 (17.408) | 26.67 (26.366)
  Insomnia: Cycle 4: number analyzed (Participants) | 50 | 38
  Insomnia: Cycle 4 | 11.33 (19.760) | 24.56 (27.601)
  Insomnia: Cycle 5: number analyzed (Participants) | 47 | 34
  Insomnia: Cycle 5 | 9.22 (19.289) | 17.65 (26.253)
  Insomnia: Cycle 6: number analyzed (Participants) | 43 | 31
  Insomnia: Cycle 6 | 10.85 (18.857) | 20.43 (26.774)
  Insomnia: Cycle 7: number analyzed (Participants) | 39 | 29
  Insomnia: Cycle 7 | 9.40 (18.651) | 21.84 (28.558)
  Insomnia: Cycle 8: number analyzed (Participants) | 37 | 25
  Insomnia: Cycle 8 | 10.81 (20.867) | 21.33 (21.257)
  Insomnia: Cycle 9: number analyzed (Participants) | 35 | 26
  Insomnia: Cycle 9 | 11.43 (19.708) | 20.51 (23.242)
  Insomnia: Cycle 10: number analyzed (Participants) | 35 | 23
  Insomnia: Cycle 10 | 12.38 (18.232) | 21.74 (21.576)
  Insomnia: Cycle 11: number analyzed (Participants) | 35 | 24
  Insomnia: Cycle 11 | 12.38 (18.232) | 22.22 (27.217)
  Insomnia: Cycle 12: number analyzed (Participants) | 35 | 22
  Insomnia: Cycle 12 | 6.67 (15.760) | 22.73 (27.958)
  Insomnia: Cycle 13: number analyzed (Participants) | 34 | 21
  Insomnia: Cycle 13 | 9.80 (15.417) | 23.81 (21.455)
  Insomnia: Cycle 14: number analyzed (Participants) | 31 | 19
  Insomnia: Cycle 14 | 8.60 (17.144) | 22.81 (19.413)
  Insomnia: Cycle 15: number analyzed (Participants) | 29 | 17
  Insomnia: Cycle 15 | 9.20 (17.586) | 25.49 (25.082)
  Insomnia: Cycle 16: number analyzed (Participants) | 27 | 16
  Insomnia: Cycle 16 | 9.88 (20.286) | 25.00 (28.545)
  Insomnia: Cycle 17: number analyzed (Participants) | 22 | 15
  Insomnia: Cycle 17 | 6.06 (16.703) | 22.22 (24.125)
  Insomnia: Cycle 18: number analyzed (Participants) | 17 | 14
  Insomnia: Cycle 18 | 11.76 (16.420) | 23.81 (24.209)
  Insomnia: Cycle 19: number analyzed (Participants) | 12 | 14
  Insomnia: Cycle 19 | 13.89 (22.285) | 23.81 (24.209)
  Insomnia: Cycle 20: number analyzed (Participants) | 11 | 13
  Insomnia: Cycle 20 | 9.09 (15.570) | 25.64 (24.167)
  Insomnia: Cycle 21: number analyzed (Participants) | 11 | 12
  Insomnia: Cycle 21 | 18.18 (22.918) | 30.56 (26.432)
  Insomnia: Cycle 22: number analyzed (Participants) | 11 | 11
  Insomnia: Cycle 22 | 15.15 (22.918) | 30.30 (27.707)
  Insomnia: Cycle 23: number analyzed (Participants) | 11 | 10
  Insomnia: Cycle 23 | 15.15 (17.408) | 30.00 (33.148)
  Insomnia: Cycle 24: number analyzed (Participants) | 10 | 10
  Insomnia: Cycle 24 | 10.00 (22.498) | 33.33 (27.217)
  Insomnia: Cycle 25: number analyzed (Participants) | 10 | 8
  Insomnia: Cycle 25 | 23.33 (27.442) | 29.17 (27.817)
  Insomnia: Cycle 26: number analyzed (Participants) | 7 | 7
  Insomnia: Cycle 26 | 9.52 (16.265) | 23.81 (25.198)
  Insomnia: Cycle 27: number analyzed (Participants) | 6 | 8
  Insomnia: Cycle 27 | 27.78 (38.968) | 33.33 (25.198)
  Insomnia: Cycle 28: number analyzed (Participants) | 7 | 8
  Insomnia: Cycle 28 | 23.81 (25.198) | 25.00 (29.547)
  Insomnia: Cycle 29: number analyzed (Participants) | 6 | 7
  Insomnia: Cycle 29 | 22.22 (27.217) | 38.10 (35.635)
  Insomnia: Cycle 30: number analyzed (Participants) | 5 | 7
  Insomnia: Cycle 30 | 6.67 (14.907) | 28.57 (29.991)
  Insomnia: Cycle 31: number analyzed (Participants) | 3 | 7
  Insomnia: Cycle 31 | 11.11 (19.245) | 19.05 (26.227)
  Insomnia: Cycle 32: number analyzed (Participants) | 3 | 6
  Insomnia: Cycle 32 | 22.22 (19.245) | 27.78 (25.092)
  Insomnia: Cycle 33: number analyzed (Participants) | 3 | 6
  Insomnia: Cycle 33 | 22.22 (19.245) | 22.22 (27.217)
  Insomnia: Cycle 34: number analyzed (Participants) | 3 | 6
  Insomnia: Cycle 34 | 22.22 (38.490) | 27.78 (25.092)
  Insomnia: Cycle 35: number analyzed (Participants) | 2 | 6
  Insomnia: Cycle 35 | 16.67 (23.570) | 27.78 (25.092)
  Insomnia: Cycle 36: number analyzed (Participants) | 1 | 5
  Insomnia: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 26.67 (27.889)
  Insomnia: Cycle 37: number analyzed (Participants) | 1 | 4
  Insomnia: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (19.245)
  Insomnia: Cycle 38: number analyzed (Participants) | 0 | 4
  Insomnia: Cycle 38 |  | 33.33 (27.217)
  Insomnia: Cycle 39: number analyzed (Participants) | 1 | 3
  Insomnia: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 22.22 (19.245)
  Insomnia: Cycle 40: number analyzed (Participants) | 1 | 3
  Insomnia: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 33.33 (0.000)
  Insomnia: Cycle 41: number analyzed (Participants) | 0 | 3
  Insomnia: Cycle 41 |  | 22.22 (19.245)
  Insomnia: Cycle 42: number analyzed (Participants) | 0 | 2
  Insomnia: Cycle 42 |  | 16.67 (23.570)
  Insomnia: Cycle 43: number analyzed (Participants) | 0 | 1
  Insomnia: Cycle 43 |  | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Insomnia: EOT: number analyzed (Participants) | 33 | 30
  Insomnia: EOT | 16.16 (26.512) | 25.56 (33.543)
  Appetite Loss: Cycle 1: number analyzed (Participants) | 61 | 44
  Appetite Loss: Cycle 1 | 12.57 (21.225) | 15.91 (23.282)
  Appetite Loss: Cycle 2: number analyzed (Participants) | 57 | 42
  Appetite Loss: Cycle 2 | 16.96 (21.009) | 18.25 (22.333)
  Appetite Loss: Cycle 3: number analyzed (Participants) | 55 | 40
  Appetite Loss: Cycle 3 | 13.94 (18.912) | 20.83 (28.929)
  Appetite Loss: Cycle 4: number analyzed (Participants) | 50 | 38
  Appetite Loss: Cycle 4 | 14.00 (24.365) | 16.67 (26.565)
  Appetite Loss: Cycle 5: number analyzed (Participants) | 47 | 34
  Appetite Loss: Cycle 5 | 10.64 (20.974) | 15.69 (28.704)
  Appetite Loss: Cycle 6: number analyzed (Participants) | 43 | 31
  Appetite Loss: Cycle 6 | 10.85 (20.212) | 18.28 (30.839)
  Appetite Loss: Cycle 7: number analyzed (Participants) | 39 | 29
  Appetite Loss: Cycle 7 | 14.53 (22.679) | 14.94 (28.986)
  Appetite Loss: Cycle 8: number analyzed (Participants) | 37 | 25
  Appetite Loss: Cycle 8 | 16.22 (25.606) | 14.67 (25.604)
  Appetite Loss: Cycle 9: number analyzed (Participants) | 35 | 26
  Appetite Loss: Cycle 9 | 14.29 (18.587) | 14.10 (26.954)
  Appetite Loss: Cycle 10: number analyzed (Participants) | 35 | 23
  Appetite Loss: Cycle 10 | 13.33 (21.693) | 17.39 (28.194)
  Appetite Loss: Cycle 11: number analyzed (Participants) | 35 | 24
  Appetite Loss: Cycle 11 | 15.24 (21.907) | 8.33 (22.522)
  Appetite Loss: Cycle 12: number analyzed (Participants) | 35 | 22
  Appetite Loss: Cycle 12 | 13.33 (25.820) | 12.12 (24.224)
  Appetite Loss: Cycle 13: number analyzed (Participants) | 34 | 21
  Appetite Loss: Cycle 13 | 13.73 (21.893) | 7.94 (14.548)
  Appetite Loss: Cycle 14: number analyzed (Participants) | 31 | 19
  Appetite Loss: Cycle 14 | 10.75 (21.751) | 10.53 (19.413)
  Appetite Loss: Cycle 15: number analyzed (Participants) | 30 | 17
  Appetite Loss: Cycle 15 | 13.33 (24.132) | 15.69 (29.149)
  Appetite Loss: Cycle 16: number analyzed (Participants) | 27 | 16
  Appetite Loss: Cycle 16 | 13.58 (23.130) | 8.33 (19.245)
  Appetite Loss: Cycle 17: number analyzed (Participants) | 22 | 15
  Appetite Loss: Cycle 17 | 10.61 (23.874) | 6.67 (18.687)
  Appetite Loss: Cycle 18: number analyzed (Participants) | 17 | 14
  Appetite Loss: Cycle 18 | 17.65 (29.149) | 9.52 (20.375)
  Appetite Loss: Cycle 19: number analyzed (Participants) | 12 | 14
  Appetite Loss: Cycle 19 | 19.44 (33.207) | 9.52 (27.514)
  Appetite Loss: Cycle 20: number analyzed (Participants) | 11 | 13
  Appetite Loss: Cycle 20 | 21.21 (34.230) | 5.13 (12.518)
  Appetite Loss: Cycle 21: number analyzed (Participants) | 11 | 12
  Appetite Loss: Cycle 21 | 21.21 (34.230) | 16.67 (22.473)
  Appetite Loss: Cycle 22: number analyzed (Participants) | 11 | 11
  Appetite Loss: Cycle 22 | 18.18 (31.140) | 15.15 (22.918)
  Appetite Loss: Cycle 23: number analyzed (Participants) | 11 | 10
  Appetite Loss: Cycle 23 | 18.18 (31.140) | 10.00 (22.498)
  Appetite Loss: Cycle 24: number analyzed (Participants) | 10 | 10
  Appetite Loss: Cycle 24 | 23.33 (35.312) | 13.33 (23.307)
  Appetite Loss: Cycle 25: number analyzed (Participants) | 10 | 8
  Appetite Loss: Cycle 25 | 23.33 (41.722) | 8.33 (23.570)
  Appetite Loss: Cycle 26: number analyzed (Participants) | 7 | 7
  Appetite Loss: Cycle 26 | 38.10 (48.795) | 4.76 (12.599)
  Appetite Loss: Cycle 27: number analyzed (Participants) | 6 | 8
  Appetite Loss: Cycle 27 | 33.33 (42.164) | 12.50 (35.355)
  Appetite Loss: Cycle 28: number analyzed (Participants) | 7 | 8
  Appetite Loss: Cycle 28 | 28.57 (40.500) | 16.67 (35.635)
  Appetite Loss: Cycle 29: number analyzed (Participants) | 6 | 7
  Appetite Loss: Cycle 29 | 11.11 (27.217) | 4.76 (12.599)
  Appetite Loss: Cycle 30: number analyzed (Participants) | 5 | 7
  Appetite Loss: Cycle 30 | 0.00 (0.000) | 4.76 (12.599)
  Appetite Loss: Cycle 31: number analyzed (Participants) | 3 | 7
  Appetite Loss: Cycle 31 | 0.00 (0.000) | 9.52 (25.198)
  Appetite Loss: Cycle 32: number analyzed (Participants) | 3 | 6
  Appetite Loss: Cycle 32 | 11.11 (19.245) | 16.67 (27.889)
  Appetite Loss: Cycle 33: number analyzed (Participants) | 3 | 6
  Appetite Loss: Cycle 33 | 22.22 (38.490) | 16.67 (27.889)
  Appetite Loss: Cycle 34: number analyzed (Participants) | 3 | 6
  Appetite Loss: Cycle 34 | 33.33 (57.735) | 27.78 (32.773)
  Appetite Loss: Cycle 35: number analyzed (Participants) | 2 | 6
  Appetite Loss: Cycle 35 | 33.33 (47.140) | 11.11 (27.217)
  Appetite Loss: Cycle 36: number analyzed (Participants) | 1 | 5
  Appetite Loss: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Appetite Loss: Cycle 37: number analyzed (Participants) | 1 | 4
  Appetite Loss: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (19.245)
  Appetite Loss: Cycle 38: number analyzed (Participants) | 0 | 4
  Appetite Loss: Cycle 38 |  | 16.67 (19.245)
  Appetite Loss: Cycle 39: number analyzed (Participants) | 1 | 3
  Appetite Loss: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Appetite Loss: Cycle 40: number analyzed (Participants) | 1 | 3
  Appetite Loss: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Appetite Loss: Cycle 41: number analyzed (Participants) | 0 | 3
  Appetite Loss: Cycle 41 |  | 22.22 (38.490)
  Appetite Loss: Cycle 42: number analyzed (Participants) | 0 | 2
  Appetite Loss: Cycle 42 |  | 16.67 (23.570)
  Appetite Loss: Cycle 43: number analyzed (Participants) | 0 | 1
  Appetite Loss: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Appetite Loss: EOT: number analyzed (Participants) | 33 | 30
  Appetite Loss: EOT | 27.27 (34.816) | 26.67 (32.044)
  Constipation: Cycle 1: number analyzed (Participants) | 61 | 44
  Constipation: Cycle 1 | 7.10 (17.336) | 9.09 (18.135)
  Constipation: Cycle 2: number analyzed (Participants) | 57 | 42
  Constipation: Cycle 2 | 3.51 (10.321) | 13.49 (26.605)
  Constipation: Cycle 3: number analyzed (Participants) | 55 | 40
  Constipation: Cycle 3 | 7.27 (15.303) | 4.17 (13.477)
  Constipation: Cycle 4: number analyzed (Participants) | 50 | 38
  Constipation: Cycle 4 | 6.67 (15.058) | 5.26 (12.318)
  Constipation: Cycle 5: number analyzed (Participants) | 47 | 34
  Constipation: Cycle 5 | 3.55 (12.499) | 2.94 (12.627)
  Constipation: Cycle 6: number analyzed (Participants) | 43 | 31
  Constipation: Cycle 6 | 3.88 (10.812) | 2.15 (8.324)
  Constipation: Cycle 7: number analyzed (Participants) | 39 | 29
  Constipation: Cycle 7 | 3.42 (10.245) | 5.75 (17.970)
  Constipation: Cycle 8: number analyzed (Participants) | 37 | 25
  Constipation: Cycle 8 | 3.60 (13.109) | 4.00 (14.657)
  Constipation: Cycle 9: number analyzed (Participants) | 35 | 26
  Constipation: Cycle 9 | 6.67 (15.760) | 3.85 (14.382)
  Constipation: Cycle 10: number analyzed (Participants) | 35 | 23
  Constipation: Cycle 10 | 2.86 (9.468) | 5.80 (16.368)
  Constipation: Cycle 11: number analyzed (Participants) | 35 | 24
  Constipation: Cycle 11 | 3.81 (13.459) | 2.78 (9.411)
  Constipation: Cycle 12: number analyzed (Participants) | 35 | 22
  Constipation: Cycle 12 | 5.71 (12.746) | 4.55 (11.708)
  Constipation: Cycle 13: number analyzed (Participants) | 34 | 21
  Constipation: Cycle 13 | 2.94 (9.597) | 1.59 (7.274)
  Constipation: Cycle 14: number analyzed (Participants) | 31 | 19
  Constipation: Cycle 14 | 1.08 (5.987) | 3.51 (10.510)
  Constipation: Cycle 15: number analyzed (Participants) | 30 | 17
  Constipation: Cycle 15 | 2.22 (8.457) | 3.92 (16.169)
  Constipation: Cycle 16: number analyzed (Participants) | 27 | 16
  Constipation: Cycle 16 | 2.47 (8.896) | 6.25 (13.437)
  Constipation: Cycle 17: number analyzed (Participants) | 22 | 15
  Constipation: Cycle 17 | 6.06 (13.159) | 2.22 (8.607)
  Constipation: Cycle 18: number analyzed (Participants) | 17 | 14
  Constipation: Cycle 18 | 3.92 (11.070) | 4.76 (12.105)
  Constipation: Cycle 19: number analyzed (Participants) | 12 | 14
  Constipation: Cycle 19 | 0.00 (0.000) | 9.52 (20.375)
  Constipation: Cycle 20: number analyzed (Participants) | 11 | 13
  Constipation: Cycle 20 | 0.00 (0.000) | 0.00 (0.000)
  Constipation: Cycle 21: number analyzed (Participants) | 11 | 12
  Constipation: Cycle 21 | 0.00 (0.000) | 2.78 (9.623)
  Constipation: Cycle 22: number analyzed (Participants) | 11 | 11
  Constipation: Cycle 22 | 0.00 (0.000) | 12.12 (30.814)
  Constipation: Cycle 23: number analyzed (Participants) | 11 | 10
  Constipation: Cycle 23 | 0.00 (0.000) | 3.33 (10.541)
  Constipation: Cycle 24: number analyzed (Participants) | 10 | 10
  Constipation: Cycle 24 | 0.00 (0.000) | 6.67 (14.055)
  Constipation: Cycle 25: number analyzed (Participants) | 10 | 8
  Constipation: Cycle 25 | 3.33 (10.541) | 0.00 (0.000)
  Constipation: Cycle 26: number analyzed (Participants) | 7 | 7
  Constipation: Cycle 26 | 0.00 (0.000) | 4.76 (12.599)
  Constipation: Cycle 27: number analyzed (Participants) | 6 | 8
  Constipation: Cycle 27 | 5.56 (13.608) | 4.17 (11.785)
  Constipation: Cycle 28: number analyzed (Participants) | 7 | 8
  Constipation: Cycle 28 | 4.76 (12.599) | 4.17 (11.785)
  Constipation: Cycle 29: number analyzed (Participants) | 5 | 7
  Constipation: Cycle 29 | 0.00 (0.000) | 4.76 (12.599)
  Constipation: Cycle 30: number analyzed (Participants) | 4 | 7
  Constipation: Cycle 30 | 0.00 (0.000) | 4.76 (12.599)
  Constipation: Cycle 31: number analyzed (Participants) | 2 | 7
  Constipation: Cycle 31 | 0.00 (0.000) | 4.76 (12.599)
  Constipation: Cycle 32: number analyzed (Participants) | 3 | 6
  Constipation: Cycle 32 | 0.00 (0.000) | 0.00 (0.000)
  Constipation: Cycle 33: number analyzed (Participants) | 3 | 6
  Constipation: Cycle 33 | 0.00 (0.000) | 5.56 (13.608)
  Constipation: Cycle 34: number analyzed (Participants) | 3 | 6
  Constipation: Cycle 34 | 0.00 (0.000) | 5.56 (13.608)
  Constipation: Cycle 35: number analyzed (Participants) | 2 | 6
  Constipation: Cycle 35 | 0.00 (0.000) | 5.56 (13.608)
  Constipation: Cycle 36: number analyzed (Participants) | 1 | 5
  Constipation: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 13.33 (29.814)
  Constipation: Cycle 37: number analyzed (Participants) | 1 | 4
  Constipation: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Constipation: Cycle 38: number analyzed (Participants) | 0 | 4
  Constipation: Cycle 38 |  | 0.00 (0.000)
  Constipation: Cycle 39: number analyzed (Participants) | 1 | 3
  Constipation: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Constipation: Cycle 40: number analyzed (Participants) | 1 | 3
  Constipation: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Constipation: Cycle 41: number analyzed (Participants) | 0 | 3
  Constipation: Cycle 41 |  | 0.00 (0.000)
  Constipation: Cycle 42: number analyzed (Participants) | 0 | 2
  Constipation: Cycle 42 |  | 0.00 (0.000)
  Constipation: Cycle 43: number analyzed (Participants) | 0 | 1
  Constipation: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Constipation: EOT: number analyzed (Participants) | 33 | 30
  Constipation: EOT | 10.10 (19.516) | 3.33 (10.171)
  Diarrhoea: Cycle 1: number analyzed (Participants) | 61 | 43
  Diarrhoea: Cycle 1 | 14.21 (22.327) | 11.63 (17.644)
  Diarrhoea: Cycle 2: number analyzed (Participants) | 57 | 41
  Diarrhoea: Cycle 2 | 18.13 (26.027) | 17.07 (25.951)
  Diarrhoea: Cycle 3: number analyzed (Participants) | 55 | 40
  Diarrhoea: Cycle 3 | 16.36 (24.740) | 24.17 (25.021)
  Diarrhoea: Cycle 4: number analyzed (Participants) | 50 | 38
  Diarrhoea: Cycle 4 | 22.00 (27.446) | 15.79 (21.556)
  Diarrhoea: Cycle 5: number analyzed (Participants) | 47 | 34
  Diarrhoea: Cycle 5 | 22.70 (26.105) | 21.57 (23.039)
  Diarrhoea: Cycle 6: number analyzed (Participants) | 43 | 31
  Diarrhoea: Cycle 6 | 24.03 (29.390) | 22.58 (21.751)
  Diarrhoea: Cycle 7: number analyzed (Participants) | 39 | 29
  Diarrhoea: Cycle 7 | 29.06 (27.762) | 25.29 (29.080)
  Diarrhoea: Cycle 8: number analyzed (Participants) | 37 | 25
  Diarrhoea: Cycle 8 | 26.13 (27.369) | 20.00 (28.868)
  Diarrhoea: Cycle 9: number analyzed (Participants) | 35 | 26
  Diarrhoea: Cycle 9 | 30.48 (30.648) | 29.49 (33.102)
  Diarrhoea: Cycle 10: number analyzed (Participants) | 35 | 23
  Diarrhoea: Cycle 10 | 24.76 (26.000) | 27.54 (29.563)
  Diarrhoea: Cycle 11: number analyzed (Participants) | 35 | 24
  Diarrhoea: Cycle 11 | 23.81 (25.012) | 23.61 (23.008)
  Diarrhoea: Cycle 12: number analyzed (Participants) | 35 | 22
  Diarrhoea: Cycle 12 | 21.90 (22.785) | 18.18 (22.366)
  Diarrhoea: Cycle 13: number analyzed (Participants) | 34 | 21
  Diarrhoea: Cycle 13 | 21.57 (21.528) | 19.05 (27.021)
  Diarrhoea: Cycle 14: number analyzed (Participants) | 31 | 19
  Diarrhoea: Cycle 14 | 23.66 (23.084) | 19.30 (20.233)
  Diarrhoea: Cycle 15: number analyzed (Participants) | 30 | 17
  Diarrhoea: Cycle 15 | 21.11 (23.947) | 25.49 (22.140)
  Diarrhoea: Cycle 16: number analyzed (Participants) | 27 | 16
  Diarrhoea: Cycle 16 | 18.52 (25.036) | 20.83 (20.638)
  Diarrhoea: Cycle 17: number analyzed (Participants) | 22 | 15
  Diarrhoea: Cycle 17 | 21.21 (19.370) | 15.56 (24.774)
  Diarrhoea: Cycle 18: number analyzed (Participants) | 17 | 14
  Diarrhoea: Cycle 18 | 25.49 (27.712) | 19.05 (25.198)
  Diarrhoea: Cycle 19: number analyzed (Participants) | 12 | 14
  Diarrhoea: Cycle 19 | 13.89 (17.164) | 19.05 (21.540)
  Diarrhoea: Cycle 20: number analyzed (Participants) | 11 | 13
  Diarrhoea: Cycle 20 | 27.27 (20.101) | 23.08 (25.036)
  Diarrhoea: Cycle 21: number analyzed (Participants) | 11 | 12
  Diarrhoea: Cycle 21 | 33.33 (29.814) | 25.00 (28.868)
  Diarrhoea: Cycle 22: number analyzed (Participants) | 11 | 11
  Diarrhoea: Cycle 22 | 18.18 (31.140) | 21.21 (26.968)
  Diarrhoea: Cycle 23: number analyzed (Participants) | 11 | 10
  Diarrhoea: Cycle 23 | 24.24 (33.635) | 26.67 (30.631)
  Diarrhoea: Cycle 24: number analyzed (Participants) | 10 | 10
  Diarrhoea: Cycle 24 | 23.33 (22.498) | 23.33 (31.623)
  Diarrhoea: Cycle 25: number analyzed (Participants) | 10 | 8
  Diarrhoea: Cycle 25 | 16.67 (17.568) | 29.17 (27.817)
  Diarrhoea: Cycle 26: number analyzed (Participants) | 7 | 7
  Diarrhoea: Cycle 26 | 19.05 (26.227) | 28.57 (29.991)
  Diarrhoea: Cycle 27: number analyzed (Participants) | 6 | 8
  Diarrhoea: Cycle 27 | 22.22 (17.213) | 37.50 (33.034)
  Diarrhoea: Cycle 28: number analyzed (Participants) | 7 | 8
  Diarrhoea: Cycle 28 | 14.29 (17.817) | 29.17 (27.817)
  Diarrhoea: Cycle 29: number analyzed (Participants) | 5 | 7
  Diarrhoea: Cycle 29 | 0.00 (0.000) | 28.57 (29.991)
  Diarrhoea: Cycle 30: number analyzed (Participants) | 4 | 7
  Diarrhoea: Cycle 30 | 0.00 (0.000) | 38.10 (23.002)
  Diarrhoea: Cycle 31: number analyzed (Participants) | 2 | 7
  Diarrhoea: Cycle 31 | 0.00 (0.000) | 33.33 (27.217)
  Diarrhoea: Cycle 32: number analyzed (Participants) | 3 | 6
  Diarrhoea: Cycle 32 | 22.22 (19.245) | 50.00 (27.889)
  Diarrhoea: Cycle 33: number analyzed (Participants) | 3 | 6
  Diarrhoea: Cycle 33 | 11.11 (19.245) | 50.00 (27.889)
  Diarrhoea: Cycle 34: number analyzed (Participants) | 3 | 6
  Diarrhoea: Cycle 34 | 33.33 (33.333) | 44.44 (27.217)
  Diarrhoea: Cycle 35: number analyzed (Participants) | 2 | 6
  Diarrhoea: Cycle 35 | 16.67 (23.570) | 38.89 (32.773)
  Diarrhoea: Cycle 36: number analyzed (Participants) | 1 | 5
  Diarrhoea: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 40.00 (43.461)
  Diarrhoea: Cycle 37: number analyzed (Participants) | 1 | 4
  Diarrhoea: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 25.00 (31.914)
  Diarrhoea: Cycle 38: number analyzed (Participants) | 0 | 4
  Diarrhoea: Cycle 38 |  | 41.67 (31.914)
  Diarrhoea: Cycle 39: number analyzed (Participants) | 1 | 3
  Diarrhoea: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 33.33 (33.333)
  Diarrhoea: Cycle 40: number analyzed (Participants) | 1 | 3
  Diarrhoea: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.44 (38.490)
  Diarrhoea: Cycle 41: number analyzed (Participants) | 0 | 3
  Diarrhoea: Cycle 41 |  | 44.44 (38.490)
  Diarrhoea: Cycle 42: number analyzed (Participants) | 0 | 2
  Diarrhoea: Cycle 42 |  | 50.00 (23.570)
  Diarrhoea: Cycle 43: number analyzed (Participants) | 0 | 1
  Diarrhoea: Cycle 43 |  | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Diarrhoea: EOT: number analyzed (Participants) | 33 | 30
  Diarrhoea: EOT | 24.24 (29.194) | 17.78 (24.343)
  Financial Difficulties: Cycle 1: number analyzed (Participants) | 61 | 43
  Financial Difficulties: Cycle 1 | 25.68 (35.691) | 31.01 (33.646)
  Financial Difficulties: Cycle 2: number analyzed (Participants) | 57 | 41
  Financial Difficulties: Cycle 2 | 23.39 (28.843) | 21.95 (26.468)
  Financial Difficulties: Cycle 3: number analyzed (Participants) | 55 | 40
  Financial Difficulties: Cycle 3 | 23.03 (30.002) | 30.00 (34.427)
  Financial Difficulties: Cycle 4: number analyzed (Participants) | 50 | 38
  Financial Difficulties: Cycle 4 | 24.00 (30.147) | 28.95 (27.037)
  Financial Difficulties: Cycle 5: number analyzed (Participants) | 47 | 34
  Financial Difficulties: Cycle 5 | 26.24 (34.005) | 25.49 (29.654)
  Financial Difficulties: Cycle 6: number analyzed (Participants) | 43 | 31
  Financial Difficulties: Cycle 6 | 27.13 (35.078) | 26.88 (31.528)
  Financial Difficulties: Cycle 7: number analyzed (Participants) | 39 | 29
  Financial Difficulties: Cycle 7 | 29.06 (31.696) | 27.59 (32.206)
  Financial Difficulties: Cycle 8: number analyzed (Participants) | 37 | 25
  Financial Difficulties: Cycle 8 | 30.63 (32.753) | 25.33 (29.313)
  Financial Difficulties: Cycle 9: number analyzed (Participants) | 35 | 26
  Financial Difficulties: Cycle 9 | 22.86 (28.892) | 20.51 (29.929)
  Financial Difficulties: Cycle 10: number analyzed (Participants) | 35 | 23
  Financial Difficulties: Cycle 10 | 25.71 (28.105) | 24.64 (30.513)
  Financial Difficulties: Cycle 11: number analyzed (Participants) | 35 | 24
  Financial Difficulties: Cycle 11 | 26.67 (27.771) | 23.61 (28.622)
  Financial Difficulties: Cycle 12: number analyzed (Participants) | 35 | 22
  Financial Difficulties: Cycle 12 | 26.67 (30.033) | 19.70 (26.546)
  Financial Difficulties: Cycle 13: number analyzed (Participants) | 34 | 21
  Financial Difficulties: Cycle 13 | 23.53 (27.864) | 19.05 (30.861)
  Financial Difficulties: Cycle 14: number analyzed (Participants) | 31 | 19
  Financial Difficulties: Cycle 14 | 23.66 (28.795) | 17.54 (28.040)
  Financial Difficulties: Cycle 15: number analyzed (Participants) | 30 | 17
  Financial Difficulties: Cycle 15 | 21.11 (22.289) | 19.61 (29.009)
  Financial Difficulties: Cycle 16: number analyzed (Participants) | 27 | 16
  Financial Difficulties: Cycle 16 | 22.22 (22.646) | 18.75 (29.736)
  Financial Difficulties: Cycle 17: number analyzed (Participants) | 22 | 15
  Financial Difficulties: Cycle 17 | 19.70 (24.471) | 15.56 (27.794)
  Financial Difficulties: Cycle 18: number analyzed (Participants) | 17 | 14
  Financial Difficulties: Cycle 18 | 17.65 (29.149) | 16.67 (21.681)
  Financial Difficulties: Cycle 19: number analyzed (Participants) | 12 | 14
  Financial Difficulties: Cycle 19 | 22.22 (32.824) | 14.29 (17.118)
  Financial Difficulties: Cycle 20: number analyzed (Participants) | 11 | 13
  Financial Difficulties: Cycle 20 | 15.15 (22.918) | 15.38 (29.235)
  Financial Difficulties: Cycle 21: number analyzed (Participants) | 11 | 12
  Financial Difficulties: Cycle 21 | 24.24 (33.635) | 16.67 (30.151)
  Financial Difficulties: Cycle 22: number analyzed (Participants) | 11 | 11
  Financial Difficulties: Cycle 22 | 18.18 (27.340) | 15.15 (22.918)
  Financial Difficulties: Cycle 23: number analyzed (Participants) | 11 | 10
  Financial Difficulties: Cycle 23 | 15.15 (22.918) | 20.00 (32.203)
  Financial Difficulties: Cycle 24: number analyzed (Participants) | 10 | 10
  Financial Difficulties: Cycle 24 | 20.00 (28.109) | 16.67 (32.394)
  Financial Difficulties: Cycle 25: number analyzed (Participants) | 10 | 8
  Financial Difficulties: Cycle 25 | 16.67 (28.328) | 29.17 (37.533)
  Financial Difficulties: Cycle 26: number analyzed (Participants) | 7 | 7
  Financial Difficulties: Cycle 26 | 23.81 (31.706) | 28.57 (40.500)
  Financial Difficulties: Cycle 27: number analyzed (Participants) | 6 | 8
  Financial Difficulties: Cycle 27 | 16.67 (27.889) | 20.83 (35.355)
  Financial Difficulties: Cycle 28: number analyzed (Participants) | 7 | 8
  Financial Difficulties: Cycle 28 | 19.05 (26.227) | 20.83 (35.355)
  Financial Difficulties: Cycle 29: number analyzed (Participants) | 5 | 7
  Financial Difficulties: Cycle 29 | 13.33 (29.814) | 19.05 (37.796)
  Financial Difficulties: Cycle 30: number analyzed (Participants) | 4 | 7
  Financial Difficulties: Cycle 30 | 16.67 (33.333) | 19.05 (37.796)
  Financial Difficulties: Cycle 31: number analyzed (Participants) | 2 | 7
  Financial Difficulties: Cycle 31 | 33.33 (47.140) | 19.05 (37.796)
  Financial Difficulties: Cycle 32: number analyzed (Participants) | 3 | 6
  Financial Difficulties: Cycle 32 | 22.22 (38.490) | 22.22 (40.369)
  Financial Difficulties: Cycle 33: number analyzed (Participants) | 3 | 6
  Financial Difficulties: Cycle 33 | 33.33 (33.333) | 22.22 (40.369)
  Financial Difficulties: Cycle 34: number analyzed (Participants) | 3 | 6
  Financial Difficulties: Cycle 34 | 22.22 (19.245) | 22.22 (40.369)
  Financial Difficulties: Cycle 35: number analyzed (Participants) | 2 | 6
  Financial Difficulties: Cycle 35 | 50.00 (23.570) | 22.22 (40.369)
  Financial Difficulties: Cycle 36: number analyzed (Participants) | 1 | 5
  Financial Difficulties: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 20.00 (44.721)
  Financial Difficulties: Cycle 37: number analyzed (Participants) | 1 | 4
  Financial Difficulties: Cycle 37 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 8.33 (16.667)
  Financial Difficulties: Cycle 38: number analyzed (Participants) | 0 | 4
  Financial Difficulties: Cycle 38 |  | 8.33 (16.667)
  Financial Difficulties: Cycle 39: number analyzed (Participants) | 1 | 3
  Financial Difficulties: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Financial Difficulties: Cycle 40: number analyzed (Participants) | 1 | 3
  Financial Difficulties: Cycle 40 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Financial Difficulties: Cycle 41: number analyzed (Participants) | 0 | 3
  Financial Difficulties: Cycle 41 |  | 22.22 (19.245)
  Financial Difficulties: Cycle 42: number analyzed (Participants) | 0 | 2
  Financial Difficulties: Cycle 42 |  | 0.00 (0.000)
  Financial Difficulties: Cycle 43: number analyzed (Participants) | 0 | 1
  Financial Difficulties: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Financial Difficulties: EOT: number analyzed (Participants) | 33 | 30
  Financial Difficulties: EOT | 30.30 (29.302) | 23.33 (26.479)

13. Secondary Outcome: Quality of Life Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Gastrointestinal Related Neuroendocrine Tumours-21 (EORTC QLQ-GI NET 21)
Description: EORTC QLQ-GI-NET 21 was a 21-item questionnaire. These 21 questions assesses endocrine symptoms, gastrointestinal (G.I.) symptoms, treatment related symptoms, social functioning, disease related worries, muscle/bone pain, sexual function, information/communication function and body image. Each item was answered on a 4-point scale: 1 =not at all, 2 =a little, 3 =quite a bit, 4 =very much; where higher scores indicated more severe symptoms/problems. Scores averaged, transformed to 0-100 scale; higher score=more severe symptoms.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
units on a scale
  Endocrine Symptoms: Cycle 1: number analyzed (Participants) | 61 | 44
  Endocrine Symptoms: Cycle 1 | 9.47 (14.746) | 15.66 (20.378)
  Endocrine Symptoms: Cycle 2: number analyzed (Participants) | 57 | 41
  Endocrine Symptoms: Cycle 2 | 9.94 (14.347) | 14.91 (16.407)
  Endocrine Symptoms: Cycle 3: number analyzed (Participants) | 55 | 40
  Endocrine Symptoms: Cycle 3 | 14.75 (20.066) | 11.67 (14.443)
  Endocrine Symptoms: Cycle 4: number analyzed (Participants) | 50 | 37
  Endocrine Symptoms: Cycle 4 | 12.67 (15.227) | 12.31 (14.531)
  Endocrine Symptoms: Cycle 5: number analyzed (Participants) | 47 | 33
  Endocrine Symptoms: Cycle 5 | 12.29 (13.752) | 8.08 (12.507)
  Endocrine Symptoms: Cycle 6: number analyzed (Participants) | 43 | 31
  Endocrine Symptoms: Cycle 6 | 13.18 (16.490) | 9.32 (13.788)
  Endocrine Symptoms: Cycle 7: number analyzed (Participants) | 39 | 29
  Endocrine Symptoms: Cycle 7 | 12.82 (14.315) | 12.07 (16.538)
  Endocrine Symptoms: Cycle 8: number analyzed (Participants) | 37 | 25
  Endocrine Symptoms: Cycle 8 | 13.81 (18.408) | 10.67 (14.515)
  Endocrine Symptoms: Cycle 9: number analyzed (Participants) | 35 | 26
  Endocrine Symptoms: Cycle 9 | 10.16 (14.851) | 11.11 (14.741)
  Endocrine Symptoms: Cycle 10: number analyzed (Participants) | 35 | 23
  Endocrine Symptoms: Cycle 10 | 10.16 (13.304) | 14.01 (18.416)
  Endocrine Symptoms: Cycle 11: number analyzed (Participants) | 35 | 24
  Endocrine Symptoms: Cycle 11 | 13.02 (16.934) | 13.43 (19.653)
  Endocrine Symptoms: Cycle 12: number analyzed (Participants) | 35 | 22
  Endocrine Symptoms: Cycle 12 | 12.06 (16.693) | 11.62 (17.644)
  Endocrine Symptoms: Cycle 13: number analyzed (Participants) | 34 | 21
  Endocrine Symptoms: Cycle 13 | 10.46 (14.459) | 11.64 (15.899)
  Endocrine Symptoms: Cycle 14: number analyzed (Participants) | 31 | 19
  Endocrine Symptoms: Cycle 14 | 12.19 (16.815) | 14.62 (18.538)
  Endocrine Symptoms: Cycle 15: number analyzed (Participants) | 30 | 17
  Endocrine Symptoms: Cycle 15 | 13.33 (18.082) | 15.69 (18.864)
  Endocrine Symptoms: Cycle 16: number analyzed (Participants) | 27 | 16
  Endocrine Symptoms: Cycle 16 | 10.70 (16.155) | 9.03 (11.631)
  Endocrine Symptoms: Cycle 17: number analyzed (Participants) | 22 | 15
  Endocrine Symptoms: Cycle 17 | 12.12 (18.753) | 8.89 (10.457)
  Endocrine Symptoms: Cycle 18: number analyzed (Participants) | 17 | 14
  Endocrine Symptoms: Cycle 18 | 11.11 (18.840) | 11.90 (14.756)
  Endocrine Symptoms: Cycle 19: number analyzed (Participants) | 12 | 14
  Endocrine Symptoms: Cycle 19 | 14.81 (21.364) | 6.35 (11.293)
  Endocrine Symptoms: Cycle 20: number analyzed (Participants) | 11 | 13
  Endocrine Symptoms: Cycle 20 | 15.15 (20.045) | 11.11 (17.568)
  Endocrine Symptoms: Cycle 21: number analyzed (Participants) | 11 | 12
  Endocrine Symptoms: Cycle 21 | 20.20 (20.975) | 9.26 (12.385)
  Endocrine Symptoms: Cycle 22: number analyzed (Participants) | 11 | 11
  Endocrine Symptoms: Cycle 22 | 14.14 (19.303) | 16.16 (21.294)
  Endocrine Symptoms: Cycle 23: number analyzed (Participants) | 11 | 10
  Endocrine Symptoms: Cycle 23 | 18.18 (15.131) | 13.33 (16.397)
  Endocrine Symptoms: Cycle 24: number analyzed (Participants) | 10 | 10
  Endocrine Symptoms: Cycle 24 | 22.22 (31.427) | 13.33 (14.628)
  Endocrine Symptoms: Cycle 25: number analyzed (Participants) | 10 | 8
  Endocrine Symptoms: Cycle 25 | 16.67 (23.570) | 8.33 (12.944)
  Endocrine Symptoms: Cycle 26: number analyzed (Participants) | 7 | 7
  Endocrine Symptoms: Cycle 26 | 22.22 (27.962) | 7.94 (13.929)
  Endocrine Symptoms: Cycle 27: number analyzed (Participants) | 6 | 8
  Endocrine Symptoms: Cycle 27 | 22.22 (28.109) | 9.72 (12.511)
  Endocrine Symptoms: Cycle 28: number analyzed (Participants) | 7 | 8
  Endocrine Symptoms: Cycle 28 | 19.05 (29.197) | 12.50 (18.245)
  Endocrine Symptoms: Cycle 29: number analyzed (Participants) | 6 | 7
  Endocrine Symptoms: Cycle 29 | 12.96 (12.989) | 11.11 (12.830)
  Endocrine Symptoms: Cycle 30: number analyzed (Participants) | 5 | 7
  Endocrine Symptoms: Cycle 30 | 8.89 (9.296) | 14.29 (13.929)
  Endocrine Symptoms: Cycle 31: number analyzed (Participants) | 3 | 7
  Endocrine Symptoms: Cycle 31 | 14.81 (6.415) | 12.70 (11.878)
  Endocrine Symptoms: Cycle 32: number analyzed (Participants) | 3 | 6
  Endocrine Symptoms: Cycle 32 | 7.41 (12.830) | 14.81 (13.456)
  Endocrine Symptoms: Cycle 33: number analyzed (Participants) | 3 | 6
  Endocrine Symptoms: Cycle 33 | 11.11 (0.000) | 16.67 (11.653)
  Endocrine Symptoms: Cycle 34: number analyzed (Participants) | 3 | 6
  Endocrine Symptoms: Cycle 34 | 18.52 (6.415) | 20.37 (23.744)
  Endocrine Symptoms: Cycle 35: number analyzed (Participants) | 2 | 6
  Endocrine Symptoms: Cycle 35 | 22.22 (0.000) | 16.67 (16.851)
  Endocrine Symptoms: Cycle 36: number analyzed (Participants) | 1 | 5
  Endocrine Symptoms: Cycle 36 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 17.78 (18.592)
  Endocrine Symptoms: Cycle 37: number analyzed (Participants) | 1 | 4
  Endocrine Symptoms: Cycle 37 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 5.56 (11.111)
  Endocrine Symptoms: Cycle 38: number analyzed (Participants) | 0 | 4
  Endocrine Symptoms: Cycle 38 |  | 8.33 (10.638)
  Endocrine Symptoms: Cycle 39: number analyzed (Participants) | 1 | 3
  Endocrine Symptoms: Cycle 39 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (11.111)
  Endocrine Symptoms: Cycle 40: number analyzed (Participants) | 1 | 3
  Endocrine Symptoms: Cycle 40 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (11.111)
  Endocrine Symptoms: Cycle 41: number analyzed (Participants) | 0 | 3
  Endocrine Symptoms: Cycle 41 |  | 11.11 (11.111)
  Endocrine Symptoms: Cycle 42: number analyzed (Participants) | 0 | 2
  Endocrine Symptoms: Cycle 42 |  | 0.00 (0.000)
  Endocrine Symptoms: Cycle 43: number analyzed (Participants) | 0 | 1
  Endocrine Symptoms: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Endocrine Symptoms: EOT: number analyzed (Participants) | 33 | 29
  Endocrine Symptoms: EOT | 13.80 (15.474) | 11.11 (16.534)
  Gastrointestinal Symptoms: Cycle 1: number analyzed (Participants) | 61 | 44
  Gastrointestinal Symptoms: Cycle 1 | 15.41 (14.633) | 15.30 (13.301)
  Gastrointestinal Symptoms: Cycle 2: number analyzed (Participants) | 57 | 41
  Gastrointestinal Symptoms: Cycle 2 | 17.66 (14.057) | 17.72 (13.631)
  Gastrointestinal Symptoms: Cycle 3: number analyzed (Participants) | 55 | 40
  Gastrointestinal Symptoms: Cycle 3 | 20.24 (17.543) | 19.50 (16.702)
  Gastrointestinal Symptoms: Cycle 4: number analyzed (Participants) | 50 | 38
  Gastrointestinal Symptoms: Cycle 4 | 19.47 (16.814) | 19.30 (17.315)
  Gastrointestinal Symptoms: Cycle 5: number analyzed (Participants) | 47 | 33
  Gastrointestinal Symptoms: Cycle 5 | 15.18 (13.528) | 21.01 (17.569)
  Gastrointestinal Symptoms: Cycle 6: number analyzed (Participants) | 43 | 31
  Gastrointestinal Symptoms: Cycle 6 | 18.76 (16.982) | 21.51 (20.273)
  Gastrointestinal Symptoms: Cycle 7: number analyzed (Participants) | 39 | 29
  Gastrointestinal Symptoms: Cycle 7 | 18.63 (19.114) | 20.23 (18.728)
  Gastrointestinal Symptoms: Cycle 8: number analyzed (Participants) | 37 | 25
  Gastrointestinal Symptoms: Cycle 8 | 20.72 (19.359) | 19.47 (15.743)
  Gastrointestinal Symptoms: Cycle 9: number analyzed (Participants) | 35 | 26
  Gastrointestinal Symptoms: Cycle 9 | 18.86 (18.040) | 19.49 (17.681)
  Gastrointestinal Symptoms: Cycle 10: number analyzed (Participants) | 35 | 23
  Gastrointestinal Symptoms: Cycle 10 | 18.38 (17.916) | 19.78 (18.315)
  Gastrointestinal Symptoms: Cycle 11: number analyzed (Participants) | 35 | 24
  Gastrointestinal Symptoms: Cycle 11 | 18.86 (15.295) | 16.94 (17.360)
  Gastrointestinal Symptoms: Cycle 12: number analyzed (Participants) | 35 | 22
  Gastrointestinal Symptoms: Cycle 12 | 18.86 (18.040) | 18.79 (20.741)
  Gastrointestinal Symptoms: Cycle 13: number analyzed (Participants) | 34 | 21
  Gastrointestinal Symptoms: Cycle 13 | 18.04 (17.641) | 14.60 (13.600)
  Gastrointestinal Symptoms: Cycle 14: number analyzed (Participants) | 31 | 19
  Gastrointestinal Symptoms: Cycle 14 | 18.06 (18.871) | 16.49 (13.943)
  Gastrointestinal Symptoms: Cycle 15: number analyzed (Participants) | 30 | 17
  Gastrointestinal Symptoms: Cycle 15 | 19.56 (17.934) | 22.35 (22.966)
  Gastrointestinal Symptoms: Cycle 16: number analyzed (Participants) | 27 | 16
  Gastrointestinal Symptoms: Cycle 16 | 17.53 (17.458) | 17.50 (14.782)
  Gastrointestinal Symptoms: Cycle 17: number analyzed (Participants) | 22 | 15
  Gastrointestinal Symptoms: Cycle 17 | 18.18 (19.099) | 13.78 (12.206)
  Gastrointestinal Symptoms: Cycle 18: number analyzed (Participants) | 17 | 14
  Gastrointestinal Symptoms: Cycle 18 | 24.31 (20.942) | 15.71 (12.433)
  Gastrointestinal Symptoms: Cycle 19: number analyzed (Participants) | 12 | 14
  Gastrointestinal Symptoms: Cycle 19 | 23.89 (21.360) | 20.48 (20.500)
  Gastrointestinal Symptoms: Cycle 20: number analyzed (Participants) | 11 | 13
  Gastrointestinal Symptoms: Cycle 20 | 25.45 (22.473) | 16.41 (15.303)
  Gastrointestinal Symptoms: Cycle 21: number analyzed (Participants) | 11 | 12
  Gastrointestinal Symptoms: Cycle 21 | 29.09 (22.759) | 17.22 (16.927)
  Gastrointestinal Symptoms: Cycle 22: number analyzed (Participants) | 11 | 11
  Gastrointestinal Symptoms: Cycle 22 | 23.03 (21.574) | 18.18 (18.641)
  Gastrointestinal Symptoms: Cycle 23: number analyzed (Participants) | 11 | 10
  Gastrointestinal Symptoms: Cycle 23 | 27.27 (26.408) | 20.00 (18.856)
  Gastrointestinal Symptoms: Cycle 24: number analyzed (Participants) | 10 | 10
  Gastrointestinal Symptoms: Cycle 24 | 26.00 (20.476) | 21.33 (18.539)
  Gastrointestinal Symptoms: Cycle 25: number analyzed (Participants) | 10 | 8
  Gastrointestinal Symptoms: Cycle 25 | 24.67 (19.386) | 23.33 (17.090)
  Gastrointestinal Symptoms: Cycle 26: number analyzed (Participants) | 7 | 7
  Gastrointestinal Symptoms: Cycle 26 | 30.48 (17.152) | 20.95 (15.601)
  Gastrointestinal Symptoms: Cycle 27: number analyzed (Participants) | 6 | 8
  Gastrointestinal Symptoms: Cycle 27 | 34.44 (28.415) | 25.83 (20.912)
  Gastrointestinal Symptoms: Cycle 28: number analyzed (Participants) | 7 | 8
  Gastrointestinal Symptoms: Cycle 28 | 28.57 (23.637) | 23.96 (20.967)
  Gastrointestinal Symptoms: Cycle 29: number analyzed (Participants) | 6 | 7
  Gastrointestinal Symptoms: Cycle 29 | 22.22 (5.443) | 28.57 (17.090)
  Gastrointestinal Symptoms: Cycle 30: number analyzed (Participants) | 5 | 7
  Gastrointestinal Symptoms: Cycle 30 | 18.67 (15.202) | 21.90 (17.518)
  Gastrointestinal Symptoms: Cycle 31: number analyzed (Participants) | 3 | 7
  Gastrointestinal Symptoms: Cycle 31 | 24.44 (26.943) | 22.86 (19.572)
  Gastrointestinal Symptoms: Cycle 32: number analyzed (Participants) | 3 | 6
  Gastrointestinal Symptoms: Cycle 32 | 22.22 (27.756) | 27.78 (19.052)
  Gastrointestinal Symptoms: Cycle 33: number analyzed (Participants) | 3 | 6
  Gastrointestinal Symptoms: Cycle 33 | 26.67 (35.277) | 23.33 (17.256)
  Gastrointestinal Symptoms: Cycle 34: number analyzed (Participants) | 3 | 6
  Gastrointestinal Symptoms: Cycle 34 | 20.00 (29.059) | 28.89 (15.587)
  Gastrointestinal Symptoms: Cycle 35: number analyzed (Participants) | 2 | 6
  Gastrointestinal Symptoms: Cycle 35 | 23.33 (32.998) | 20.00 (15.202)
  Gastrointestinal Symptoms: Cycle 36: number analyzed (Participants) | 1 | 5
  Gastrointestinal Symptoms: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 17.33 (15.348)
  Gastrointestinal Symptoms: Cycle 37: number analyzed (Participants) | 1 | 4
  Gastrointestinal Symptoms: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 21.67 (13.744)
  Gastrointestinal Symptoms: Cycle 38: number analyzed (Participants) | 0 | 4
  Gastrointestinal Symptoms: Cycle 38 |  | 27.92 (20.520)
  Gastrointestinal Symptoms: Cycle 39: number analyzed (Participants) | 1 | 3
  Gastrointestinal Symptoms: Cycle 39 | 6.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 31.11 (19.245)
  Gastrointestinal Symptoms: Cycle 40: number analyzed (Participants) | 1 | 3
  Gastrointestinal Symptoms: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 26.67 (17.638)
  Gastrointestinal Symptoms: Cycle 41: number analyzed (Participants) | 0 | 3
  Gastrointestinal Symptoms: Cycle 41 |  | 35.56 (21.430)
  Gastrointestinal Symptoms: Cycle 42: number analyzed (Participants) | 0 | 2
  Gastrointestinal Symptoms: Cycle 42 |  | 33.33 (18.856)
  Gastrointestinal Symptoms: Cycle 43: number analyzed (Participants) | 0 | 1
  Gastrointestinal Symptoms: Cycle 43 |  | 20.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Gastrointestinal Symptoms:EOT: number analyzed (Participants) | 33 | 29
  Gastrointestinal Symptoms:EOT | 23.23 (18.568) | 18.85 (19.766)
  Treatment Related Symptoms: Cycle 1: number analyzed (Participants) | 19 | 13
  Treatment Related Symptoms: Cycle 1 | 12.57 (14.797) | 16.24 (19.038)
  Treatment Related Symptoms: Cycle 2: number analyzed (Participants) | 56 | 36
  Treatment Related Symptoms: Cycle 2 | 14.48 (11.686) | 16.20 (14.141)
  Treatment Related Symptoms: Cycle 3: number analyzed (Participants) | 49 | 39
  Treatment Related Symptoms: Cycle 3 | 15.42 (12.280) | 17.09 (18.574)
  Treatment Related Symptoms: Cycle 4: number analyzed (Participants) | 45 | 36
  Treatment Related Symptoms: Cycle 4 | 17.53 (15.622) | 13.89 (16.074)
  Treatment Related Symptoms: Cycle 5: number analyzed (Participants) | 45 | 31
  Treatment Related Symptoms: Cycle 5 | 15.06 (11.522) | 14.52 (15.361)
  Treatment Related Symptoms: Cycle 6: number analyzed (Participants) | 41 | 30
  Treatment Related Symptoms: Cycle 6 | 15.45 (13.293) | 15.00 (17.577)
  Treatment Related Symptoms: Cycle 7: number analyzed (Participants) | 37 | 27
  Treatment Related Symptoms: Cycle 7 | 18.77 (16.216) | 15.84 (17.207)
  Treatment Related Symptoms: Cycle 8: number analyzed (Participants) | 35 | 24
  Treatment Related Symptoms: Cycle 8 | 20.48 (19.930) | 14.12 (17.870)
  Treatment Related Symptoms: Cycle 9: number analyzed (Participants) | 32 | 23
  Treatment Related Symptoms: Cycle 9 | 18.23 (15.917) | 14.01 (17.558)
  Treatment Related Symptoms: Cycle 10: number analyzed (Participants) | 33 | 23
  Treatment Related Symptoms: Cycle 10 | 15.99 (15.760) | 16.91 (17.446)
  Treatment Related Symptoms: Cycle 11: number analyzed (Participants) | 35 | 24
  Treatment Related Symptoms: Cycle 11 | 16.83 (16.196) | 15.05 (21.453)
  Treatment Related Symptoms: Cycle 12: number analyzed (Participants) | 34 | 21
  Treatment Related Symptoms: Cycle 12 | 16.01 (18.989) | 11.11 (13.494)
  Treatment Related Symptoms: Cycle 13: number analyzed (Participants) | 32 | 19
  Treatment Related Symptoms: Cycle 13 | 15.45 (12.441) | 7.89 (8.942)
  Treatment Related Symptoms: Cycle 14: number analyzed (Participants) | 29 | 19
  Treatment Related Symptoms: Cycle 14 | 13.60 (12.386) | 11.70 (13.968)
  Treatment Related Symptoms: Cycle 15: number analyzed (Participants) | 28 | 16
  Treatment Related Symptoms: Cycle 15 | 15.48 (12.950) | 8.68 (12.664)
  Treatment Related Symptoms: Cycle 16: number analyzed (Participants) | 25 | 15
  Treatment Related Symptoms: Cycle 16 | 13.78 (13.714) | 10.74 (14.467)
  Treatment Related Symptoms: Cycle 17: number analyzed (Participants) | 21 | 15
  Treatment Related Symptoms: Cycle 17 | 14.81 (15.941) | 7.41 (8.572)
  Treatment Related Symptoms: Cycle 18: number analyzed (Participants) | 16 | 14
  Treatment Related Symptoms: Cycle 18 | 17.71 (16.999) | 10.71 (11.828)
  Treatment Related Symptoms: Cycle 19: number analyzed (Participants) | 10 | 14
  Treatment Related Symptoms: Cycle 19 | 20.00 (17.013) | 12.30 (13.287)
  Treatment Related Symptoms: Cycle 20: number analyzed (Participants) | 10 | 12
  Treatment Related Symptoms: Cycle 20 | 18.33 (17.382) | 9.72 (11.392)
  Treatment Related Symptoms: Cycle 21: number analyzed (Participants) | 11 | 12
  Treatment Related Symptoms: Cycle 21 | 18.18 (18.608) | 14.81 (14.279)
  Treatment Related Symptoms: Cycle 22: number analyzed (Participants) | 10 | 11
  Treatment Related Symptoms: Cycle 22 | 24.44 (22.253) | 12.63 (12.691)
  Treatment Related Symptoms: Cycle 23: number analyzed (Participants) | 10 | 10
  Treatment Related Symptoms: Cycle 23 | 22.22 (23.570) | 13.89 (13.671)
  Treatment Related Symptoms: Cycle 24: number analyzed (Participants) | 9 | 10
  Treatment Related Symptoms: Cycle 24 | 22.84 (24.602) | 11.67 (13.969)
  Treatment Related Symptoms: Cycle 25: number analyzed (Participants) | 8 | 8
  Treatment Related Symptoms: Cycle 25 | 21.53 (21.504) | 15.28 (14.164)
  Treatment Related Symptoms: Cycle 26: number analyzed (Participants) | 7 | 7
  Treatment Related Symptoms: Cycle 26 | 26.19 (21.448) | 12.70 (11.437)
  Treatment Related Symptoms: Cycle 27: number analyzed (Participants) | 6 | 8
  Treatment Related Symptoms: Cycle 27 | 37.96 (16.636) | 19.44 (18.306)
  Treatment Related Symptoms: Cycle 28: number analyzed (Participants) | 5 | 8
  Treatment Related Symptoms: Cycle 28 | 35.56 (21.009) | 17.36 (15.555)
  Treatment Related Symptoms: Cycle 29: number analyzed (Participants) | 4 | 7
  Treatment Related Symptoms: Cycle 29 | 16.67 (4.536) | 15.87 (12.184)
  Treatment Related Symptoms: Cycle 30: number analyzed (Participants) | 3 | 7
  Treatment Related Symptoms: Cycle 30 | 20.37 (3.208) | 15.87 (14.138)
  Treatment Related Symptoms: Cycle 31: number analyzed (Participants) | 3 | 7
  Treatment Related Symptoms: Cycle 31 | 22.22 (11.111) | 20.63 (17.484)
  Treatment Related Symptoms: Cycle 32: number analyzed (Participants) | 3 | 6
  Treatment Related Symptoms: Cycle 32 | 16.67 (5.556) | 20.37 (7.590)
  Treatment Related Symptoms: Cycle 33: number analyzed (Participants) | 3 | 6
  Treatment Related Symptoms: Cycle 33 | 22.22 (11.111) | 20.37 (7.590)
  Treatment Related Symptoms: Cycle 34: number analyzed (Participants) | 3 | 6
  Treatment Related Symptoms: Cycle 34 | 27.78 (9.623) | 20.37 (12.989)
  Treatment Related Symptoms: Cycle 35: number analyzed (Participants) | 2 | 6
  Treatment Related Symptoms: Cycle 35 | 11.11 (15.713) | 17.59 (11.340)
  Treatment Related Symptoms: Cycle 36: number analyzed (Participants) | 1 | 5
  Treatment Related Symptoms: Cycle 36 | 16.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 25.56 (7.454)
  Treatment Related Symptoms: Cycle 37: number analyzed (Participants) | 1 | 4
  Treatment Related Symptoms: Cycle 37 | 16.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 26.39 (8.333)
  Treatment Related Symptoms: Cycle 38: number analyzed (Participants) | 0 | 3
  Treatment Related Symptoms: Cycle 38 |  | 22.22 (11.111)
  Treatment Related Symptoms: Cycle 39: number analyzed (Participants) | 1 | 3
  Treatment Related Symptoms: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 29.63 (6.415)
  Treatment Related Symptoms: Cycle 40: number analyzed (Participants) | 1 | 3
  Treatment Related Symptoms: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 25.93 (6.415)
  Treatment Related Symptoms: Cycle 41: number analyzed (Participants) | 0 | 3
  Treatment Related Symptoms: Cycle 41 |  | 24.07 (8.486)
  Treatment Related Symptoms: Cycle 42: number analyzed (Participants) | 0 | 2
  Treatment Related Symptoms: Cycle 42 |  | 27.78 (7.857)
  Treatment Related Symptoms: Cycle 43: number analyzed (Participants) | 0 | 1
  Treatment Related Symptoms: Cycle 43 |  | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Treatment Related Symptoms: EOT: number analyzed (Participants) | 29 | 27
  Treatment Related Symptoms: EOT | 24.33 (20.542) | 20.78 (24.969)
  Social Functioning: Cycle 1: number analyzed (Participants) | 61 | 44
  Social Functioning: Cycle 1 | 35.34 (22.907) | 31.06 (20.132)
  Social Functioning: Cycle 2: number analyzed (Participants) | 57 | 41
  Social Functioning: Cycle 2 | 30.99 (21.490) | 29.81 (22.695)
  Social Functioning: Cycle 3: number analyzed (Participants) | 55 | 40
  Social Functioning: Cycle 3 | 29.49 (20.534) | 30.00 (25.061)
  Social Functioning: Cycle 4: number analyzed (Participants) | 50 | 38
  Social Functioning: Cycle 4 | 27.00 (19.441) | 26.17 (22.331)
  Social Functioning: Cycle 5: number analyzed (Participants) | 47 | 33
  Social Functioning: Cycle 5 | 27.90 (19.087) | 24.24 (22.473)
  Social Functioning: Cycle 6: number analyzed (Participants) | 43 | 31
  Social Functioning: Cycle 6 | 25.71 (21.138) | 28.32 (23.101)
  Social Functioning: Cycle 7: number analyzed (Participants) | 39 | 29
  Social Functioning: Cycle 7 | 29.06 (20.171) | 27.20 (26.157)
  Social Functioning: Cycle 8: number analyzed (Participants) | 37 | 25
  Social Functioning: Cycle 8 | 30.63 (20.015) | 27.11 (20.051)
  Social Functioning: Cycle 9: number analyzed (Participants) | 35 | 26
  Social Functioning: Cycle 9 | 29.84 (27.715) | 23.08 (19.607)
  Social Functioning: Cycle 10: number analyzed (Participants) | 35 | 23
  Social Functioning: Cycle 10 | 28.89 (22.579) | 24.64 (24.835)
  Social Functioning: Cycle 11: number analyzed (Participants) | 35 | 24
  Social Functioning: Cycle 11 | 29.21 (21.573) | 24.07 (22.383)
  Social Functioning: Cycle 12: number analyzed (Participants) | 35 | 22
  Social Functioning: Cycle 12 | 28.25 (24.454) | 23.74 (22.562)
  Social Functioning: Cycle 13: number analyzed (Participants) | 34 | 21
  Social Functioning: Cycle 13 | 24.84 (23.380) | 23.81 (23.382)
  Social Functioning: Cycle 14: number analyzed (Participants) | 31 | 19
  Social Functioning: Cycle 14 | 27.96 (20.056) | 25.73 (24.018)
  Social Functioning: Cycle 15: number analyzed (Participants) | 30 | 17
  Social Functioning: Cycle 15 | 28.52 (20.149) | 28.76 (28.070)
  Social Functioning: Cycle 16: number analyzed (Participants) | 27 | 16
  Social Functioning: Cycle 16 | 27.16 (20.286) | 27.78 (23.307)
  Social Functioning: Cycle 17: number analyzed (Participants) | 22 | 15
  Social Functioning: Cycle 17 | 28.79 (21.320) | 23.70 (22.564)
  Social Functioning: Cycle 18: number analyzed (Participants) | 17 | 14
  Social Functioning: Cycle 18 | 29.41 (26.040) | 26.98 (21.666)
  Social Functioning: Cycle 19: number analyzed (Participants) | 12 | 14
  Social Functioning: Cycle 19 | 29.63 (25.219) | 28.57 (22.943)
  Social Functioning: Cycle 20: number analyzed (Participants) | 11 | 13
  Social Functioning: Cycle 20 | 31.82 (28.119) | 29.06 (28.160)
  Social Functioning: Cycle 21: number analyzed (Participants) | 11 | 12
  Social Functioning: Cycle 21 | 35.35 (30.151) | 24.07 (23.130)
  Social Functioning: Cycle 22: number analyzed (Participants) | 11 | 11
  Social Functioning: Cycle 22 | 31.31 (28.029) | 27.27 (24.527)
  Social Functioning: Cycle 23: number analyzed (Participants) | 11 | 10
  Social Functioning: Cycle 23 | 30.30 (28.149) | 26.67 (27.317)
  Social Functioning: Cycle 24: number analyzed (Participants) | 10 | 10
  Social Functioning: Cycle 24 | 38.89 (28.328) | 24.44 (24.456)
  Social Functioning: Cycle 25: number analyzed (Participants) | 10 | 8
  Social Functioning: Cycle 25 | 35.56 (27.116) | 31.94 (26.184)
  Social Functioning: Cycle 26: number analyzed (Participants) | 7 | 7
  Social Functioning: Cycle 26 | 46.03 (28.276) | 22.22 (11.111)
  Social Functioning: Cycle 27: number analyzed (Participants) | 6 | 8
  Social Functioning: Cycle 27 | 51.85 (28.689) | 33.33 (28.483)
  Social Functioning: Cycle 28: number analyzed (Participants) | 7 | 8
  Social Functioning: Cycle 28 | 46.03 (33.597) | 31.94 (29.360)
  Social Functioning: Cycle 29: number analyzed (Participants) | 6 | 7
  Social Functioning: Cycle 29 | 35.19 (25.740) | 28.57 (27.857)
  Social Functioning: Cycle 30: number analyzed (Participants) | 5 | 7
  Social Functioning: Cycle 30 | 35.56 (26.527) | 30.16 (29.893)
  Social Functioning: Cycle 31: number analyzed (Participants) | 3 | 7
  Social Functioning: Cycle 31 | 44.44 (22.222) | 30.16 (29.197)
  Social Functioning: Cycle 32: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 32 | 33.33 (11.111) | 31.48 (30.965)
  Social Functioning: Cycle 33: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 33 | 40.74 (23.130) | 40.74 (31.164)
  Social Functioning: Cycle 34: number analyzed (Participants) | 3 | 6
  Social Functioning: Cycle 34 | 44.44 (22.222) | 35.19 (29.327)
  Social Functioning: Cycle 35: number analyzed (Participants) | 2 | 6
  Social Functioning: Cycle 35 | 38.89 (23.570) | 33.33 (24.343)
  Social Functioning: Cycle 36: number analyzed (Participants) | 1 | 5
  Social Functioning: Cycle 36 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 31.11 (27.666)
  Social Functioning: Cycle 37: number analyzed (Participants) | 1 | 4
  Social Functioning: Cycle 37 | 22.22 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 30.56 (39.933)
  Social Functioning: Cycle 38: number analyzed (Participants) | 0 | 4
  Social Functioning: Cycle 38 |  | 41.67 (41.944)
  Social Functioning: Cycle 39: number analyzed (Participants) | 1 | 3
  Social Functioning: Cycle 39 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 51.85 (44.905)
  Social Functioning: Cycle 40: number analyzed (Participants) | 1 | 3
  Social Functioning: Cycle 40 | 11.11 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 42.59 (36.991)
  Social Functioning: Cycle 41: number analyzed (Participants) | 0 | 3
  Social Functioning: Cycle 41 |  | 44.44 (40.062)
  Social Functioning: Cycle 42: number analyzed (Participants) | 0 | 2
  Social Functioning: Cycle 42 |  | 38.89 (39.284)
  Social Functioning: Cycle 43: number analyzed (Participants) | 0 | 1
  Social Functioning: Cycle 43 |  | 11.11 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Social Functioning: EOT: number analyzed (Participants) | 33 | 29
  Social Functioning: EOT | 39.73 (25.914) | 41.38 (26.874)
  Disease Related Worries: Cycle 1: number analyzed (Participants) | 61 | 43
  Disease Related Worries: Cycle 1 | 49.27 (26.381) | 42.89 (23.108)
  Disease Related Worries: Cycle 2: number analyzed (Participants) | 57 | 41
  Disease Related Worries: Cycle 2 | 38.01 (24.550) | 36.04 (24.942)
  Disease Related Worries: Cycle 3: number analyzed (Participants) | 55 | 40
  Disease Related Worries: Cycle 3 | 36.46 (23.074) | 34.58 (23.853)
  Disease Related Worries: Cycle 4: number analyzed (Participants) | 50 | 38
  Disease Related Worries: Cycle 4 | 31.89 (22.075) | 33.19 (23.904)
  Disease Related Worries: Cycle 5: number analyzed (Participants) | 47 | 33
  Disease Related Worries: Cycle 5 | 37.12 (25.619) | 30.64 (22.742)
  Disease Related Worries: Cycle 6: number analyzed (Participants) | 43 | 31
  Disease Related Worries: Cycle 6 | 36.43 (25.148) | 34.05 (25.000)
  Disease Related Worries: Cycle 7: number analyzed (Participants) | 39 | 29
  Disease Related Worries: Cycle 7 | 39.32 (24.825) | 32.18 (26.618)
  Disease Related Worries: Cycle 8: number analyzed (Participants) | 37 | 25
  Disease Related Worries: Cycle 8 | 38.29 (25.653) | 32.00 (22.753)
  Disease Related Worries: Cycle 9: number analyzed (Participants) | 35 | 26
  Disease Related Worries: Cycle 9 | 35.71 (31.116) | 32.05 (22.072)
  Disease Related Worries: Cycle 10: number analyzed (Participants) | 35 | 23
  Disease Related Worries: Cycle 10 | 37.30 (26.458) | 28.02 (26.563)
  Disease Related Worries: Cycle 11: number analyzed (Participants) | 35 | 24
  Disease Related Worries: Cycle 11 | 35.87 (25.292) | 27.78 (22.700)
  Disease Related Worries: Cycle 12: number analyzed (Participants) | 35 | 22
  Disease Related Worries: Cycle 12 | 35.56 (28.621) | 29.29 (25.325)
  Disease Related Worries: Cycle 13: number analyzed (Participants) | 34 | 21
  Disease Related Worries: Cycle 13 | 34.64 (27.046) | 30.16 (24.881)
  Disease Related Worries: Cycle 14: number analyzed (Participants) | 31 | 19
  Disease Related Worries: Cycle 14 | 32.97 (22.312) | 31.87 (22.055)
  Disease Related Worries: Cycle 15: number analyzed (Participants) | 30 | 17
  Disease Related Worries: Cycle 15 | 34.44 (25.160) | 33.66 (27.250)
  Disease Related Worries: Cycle 16: number analyzed (Participants) | 27 | 16
  Disease Related Worries: Cycle 16 | 34.16 (25.022) | 37.85 (23.589)
  Disease Related Worries: Cycle 17: number analyzed (Participants) | 22 | 15
  Disease Related Worries: Cycle 17 | 29.80 (22.059) | 34.07 (27.043)
  Disease Related Worries: Cycle 18: number analyzed (Participants) | 17 | 14
  Disease Related Worries: Cycle 18 | 30.07 (28.805) | 32.14 (27.232)
  Disease Related Worries: Cycle 19: number analyzed (Participants) | 12 | 14
  Disease Related Worries: Cycle 19 | 37.50 (29.504) | 31.75 (28.862)
  Disease Related Worries: Cycle 20: number analyzed (Participants) | 11 | 13
  Disease Related Worries: Cycle 20 | 40.40 (32.687) | 29.91 (31.877)
  Disease Related Worries: Cycle 21: number analyzed (Participants) | 11 | 12
  Disease Related Worries: Cycle 21 | 39.90 (30.512) | 27.78 (30.887)
  Disease Related Worries: Cycle 22: number analyzed (Participants) | 11 | 11
  Disease Related Worries: Cycle 22 | 33.33 (31.032) | 30.30 (34.816)
  Disease Related Worries: Cycle 23: number analyzed (Participants) | 11 | 10
  Disease Related Worries: Cycle 23 | 36.36 (35.168) | 26.11 (29.403)
  Disease Related Worries: Cycle 24: number analyzed (Participants) | 10 | 10
  Disease Related Worries: Cycle 24 | 41.11 (32.309) | 27.78 (28.328)
  Disease Related Worries: Cycle 25: number analyzed (Participants) | 10 | 8
  Disease Related Worries: Cycle 25 | 38.33 (32.547) | 38.89 (31.983)
  Disease Related Worries: Cycle 26: number analyzed (Participants) | 7 | 7
  Disease Related Worries: Cycle 26 | 42.86 (33.597) | 31.75 (33.597)
  Disease Related Worries: Cycle 27: number analyzed (Participants) | 6 | 8
  Disease Related Worries: Cycle 27 | 52.78 (40.023) | 34.72 (28.133)
  Disease Related Worries: Cycle 28: number analyzed (Participants) | 7 | 8
  Disease Related Worries: Cycle 28 | 50.79 (38.946) | 40.28 (39.368)
  Disease Related Worries: Cycle 29: number analyzed (Participants) | 6 | 7
  Disease Related Worries: Cycle 29 | 37.96 (35.210) | 38.10 (35.635)
  Disease Related Worries: Cycle 30: number analyzed (Participants) | 5 | 7
  Disease Related Worries: Cycle 30 | 35.56 (38.809) | 34.92 (29.696)
  Disease Related Worries: Cycle 31: number analyzed (Participants) | 3 | 7
  Disease Related Worries: Cycle 31 | 48.15 (46.259) | 36.51 (32.530)
  Disease Related Worries: Cycle 32: number analyzed (Participants) | 3 | 6
  Disease Related Worries: Cycle 32 | 25.93 (23.130) | 37.04 (38.276)
  Disease Related Worries: Cycle 33: number analyzed (Participants) | 3 | 6
  Disease Related Worries: Cycle 33 | 51.85 (42.066) | 35.19 (36.118)
  Disease Related Worries: Cycle 34: number analyzed (Participants) | 3 | 6
  Disease Related Worries: Cycle 34 | 55.56 (40.062) | 35.19 (36.796)
  Disease Related Worries: Cycle 35: number analyzed (Participants) | 2 | 6
  Disease Related Worries: Cycle 35 | 16.67 (23.570) | 35.19 (34.006)
  Disease Related Worries: Cycle 36: number analyzed (Participants) | 1 | 5
  Disease Related Worries: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 31.11 (36.345)
  Disease Related Worries: Cycle 37: number analyzed (Participants) | 1 | 4
  Disease Related Worries: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 22.22 (31.427)
  Disease Related Worries: Cycle 38: number analyzed (Participants) | 0 | 4
  Disease Related Worries: Cycle 38 |  | 33.33 (45.361)
  Disease Related Worries: Cycle 39: number analyzed (Participants) | 1 | 3
  Disease Related Worries: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.44 (50.918)
  Disease Related Worries: Cycle 40: number analyzed (Participants) | 1 | 3
  Disease Related Worries: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 37.04 (35.717)
  Disease Related Worries: Cycle 41: number analyzed (Participants) | 0 | 3
  Disease Related Worries: Cycle 41 |  | 44.44 (50.918)
  Disease Related Worries: Cycle 42: number analyzed (Participants) | 0 | 2
  Disease Related Worries: Cycle 42 |  | 50.00 (54.997)
  Disease Related Worries: Cycle 43: number analyzed (Participants) | 0 | 1
  Disease Related Worries: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Disease Related Worries: EOT: number analyzed (Participants) | 33 | 29
  Disease Related Worries: EOT | 50.84 (27.079) | 41.38 (30.123)
  Muscle/Bone Pain Symptom: Cycle 1: number analyzed (Participants) | 59 | 44
  Muscle/Bone Pain Symptom: Cycle 1 | 13.56 (20.640) | 13.64 (20.734)
  Muscle/Bone Pain Symptom: Cycle 2: number analyzed (Participants) | 57 | 41
  Muscle/Bone Pain Symptom: Cycle 2 | 20.47 (24.197) | 17.89 (23.685)
  Muscle/Bone Pain Symptom: Cycle 3: number analyzed (Participants) | 55 | 40
  Muscle/Bone Pain Symptom: Cycle 3 | 16.36 (19.108) | 23.33 (24.108)
  Muscle/Bone Pain Symptom: Cycle 4: number analyzed (Participants) | 50 | 38
  Muscle/Bone Pain Symptom: Cycle 4 | 16.00 (20.471) | 21.93 (26.024)
  Muscle/Bone Pain Symptom: Cycle 5: number analyzed (Participants) | 47 | 33
  Muscle/Bone Pain Symptom: Cycle 5 | 17.02 (18.221) | 22.22 (27.217)
  Muscle/Bone Pain Symptom: Cycle 6: number analyzed (Participants) | 43 | 31
  Muscle/Bone Pain Symptom: Cycle 6 | 18.60 (20.959) | 20.43 (23.847)
  Muscle/Bone Pain Symptom: Cycle 7: number analyzed (Participants) | 39 | 29
  Muscle/Bone Pain Symptom: Cycle 7 | 20.51 (22.446) | 21.84 (29.915)
  Muscle/Bone Pain Symptom: Cycle 8: number analyzed (Participants) | 37 | 25
  Muscle/Bone Pain Symptom: Cycle 8 | 20.72 (22.705) | 20.00 (23.570)
  Muscle/Bone Pain Symptom: Cycle 9: number analyzed (Participants) | 35 | 26
  Muscle/Bone Pain Symptom: Cycle 9 | 16.19 (18.737) | 20.51 (21.243)
  Muscle/Bone Pain Symptom: Cycle 10: number analyzed (Participants) | 35 | 23
  Muscle/Bone Pain Symptom: Cycle 10 | 20.00 (25.820) | 24.64 (28.810)
  Muscle/Bone Pain Symptom: Cycle 11: number analyzed (Participants) | 35 | 24
  Muscle/Bone Pain Symptom: Cycle 11 | 21.90 (25.492) | 22.22 (25.380)
  Muscle/Bone Pain Symptom: Cycle 12: number analyzed (Participants) | 35 | 22
  Muscle/Bone Pain Symptom: Cycle 12 | 20.95 (26.918) | 19.70 (24.471)
  Muscle/Bone Pain Symptom: Cycle 13: number analyzed (Participants) | 34 | 21
  Muscle/Bone Pain Symptom: Cycle 13 | 20.59 (24.638) | 23.81 (28.172)
  Muscle/Bone Pain Symptom: Cycle 14: number analyzed (Participants) | 31 | 19
  Muscle/Bone Pain Symptom: Cycle 14 | 12.90 (22.240) | 22.81 (27.336)
  Muscle/Bone Pain Symptom: Cycle 15: number analyzed (Participants) | 29 | 17
  Muscle/Bone Pain Symptom: Cycle 15 | 11.49 (18.422) | 25.49 (32.338)
  Muscle/Bone Pain Symptom: Cycle 16: number analyzed (Participants) | 27 | 16
  Muscle/Bone Pain Symptom: Cycle 16 | 19.75 (24.909) | 16.67 (24.343)
  Muscle/Bone Pain Symptom: Cycle 17: number analyzed (Participants) | 22 | 15
  Muscle/Bone Pain Symptom: Cycle 17 | 22.73 (25.996) | 15.56 (24.774)
  Muscle/Bone Pain Symptom: Cycle 18: number analyzed (Participants) | 17 | 14
  Muscle/Bone Pain Symptom: Cycle 18 | 15.69 (20.809) | 14.29 (25.198)
  Muscle/Bone Pain Symptom: Cycle 19: number analyzed (Participants) | 12 | 14
  Muscle/Bone Pain Symptom: Cycle 19 | 25.00 (20.719) | 16.67 (25.318)
  Muscle/Bone Pain Symptom: Cycle 20: number analyzed (Participants) | 11 | 13
  Muscle/Bone Pain Symptom: Cycle 20 | 27.27 (25.025) | 12.82 (21.681)
  Muscle/Bone Pain Symptom: Cycle 21: number analyzed (Participants) | 11 | 12
  Muscle/Bone Pain Symptom: Cycle 21 | 21.21 (22.473) | 13.89 (22.285)
  Muscle/Bone Pain Symptom: Cycle 22: number analyzed (Participants) | 11 | 11
  Muscle/Bone Pain Symptom: Cycle 22 | 15.15 (22.918) | 24.24 (26.208)
  Muscle/Bone Pain Symptom: Cycle 23: number analyzed (Participants) | 11 | 10
  Muscle/Bone Pain Symptom: Cycle 23 | 21.21 (26.968) | 23.33 (22.498)
  Muscle/Bone Pain Symptom: Cycle 24: number analyzed (Participants) | 10 | 10
  Muscle/Bone Pain Symptom: Cycle 24 | 20.00 (23.307) | 30.00 (29.187)
  Muscle/Bone Pain Symptom: Cycle 25: number analyzed (Participants) | 10 | 8
  Muscle/Bone Pain Symptom: Cycle 25 | 23.33 (27.442) | 33.33 (30.861)
  Muscle/Bone Pain Symptom: Cycle 26: number analyzed (Participants) | 7 | 7
  Muscle/Bone Pain Symptom: Cycle 26 | 33.33 (27.217) | 28.57 (29.991)
  Muscle/Bone Pain Symptom: Cycle 27: number analyzed (Participants) | 6 | 8
  Muscle/Bone Pain Symptom: Cycle 27 | 50.00 (18.257) | 29.17 (27.817)
  Muscle/Bone Pain Symptom: Cycle 28: number analyzed (Participants) | 7 | 8
  Muscle/Bone Pain Symptom: Cycle 28 | 38.10 (23.002) | 33.33 (35.635)
  Muscle/Bone Pain Symptom: Cycle 29: number analyzed (Participants) | 6 | 7
  Muscle/Bone Pain Symptom: Cycle 29 | 22.22 (27.217) | 33.33 (27.217)
  Muscle/Bone Pain Symptom: Cycle 30: number analyzed (Participants) | 5 | 7
  Muscle/Bone Pain Symptom: Cycle 30 | 26.67 (27.889) | 28.57 (35.635)
  Muscle/Bone Pain Symptom: Cycle 31: number analyzed (Participants) | 3 | 7
  Muscle/Bone Pain Symptom: Cycle 31 | 22.22 (38.490) | 38.10 (29.991)
  Muscle/Bone Pain Symptom: Cycle 32: number analyzed (Participants) | 3 | 6
  Muscle/Bone Pain Symptom: Cycle 32 | 22.22 (38.490) | 38.89 (13.608)
  Muscle/Bone Pain Symptom: Cycle 33: number analyzed (Participants) | 3 | 6
  Muscle/Bone Pain Symptom: Cycle 33 | 33.33 (33.333) | 33.33 (29.814)
  Muscle/Bone Pain Symptom: Cycle 34: number analyzed (Participants) | 3 | 6
  Muscle/Bone Pain Symptom: Cycle 34 | 11.11 (19.245) | 44.44 (17.213)
  Muscle/Bone Pain Symptom: Cycle 35: number analyzed (Participants) | 2 | 6
  Muscle/Bone Pain Symptom: Cycle 35 | 33.33 (47.140) | 38.89 (13.608)
  Muscle/Bone Pain Symptom: Cycle 36: number analyzed (Participants) | 1 | 5
  Muscle/Bone Pain Symptom: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 53.33 (18.257)
  Muscle/Bone Pain Symptom: Cycle 37: number analyzed (Participants) | 1 | 4
  Muscle/Bone Pain Symptom: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 50.00 (19.245)
  Muscle/Bone Pain Symptom: Cycle 38: number analyzed (Participants) | 0 | 4
  Muscle/Bone Pain Symptom: Cycle 38 |  | 58.33 (16.667)
  Muscle/Bone Pain Symptom: Cycle 39: number analyzed (Participants) | 1 | 3
  Muscle/Bone Pain Symptom: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 44.44 (19.245)
  Muscle/Bone Pain Symptom: Cycle 40: number analyzed (Participants) | 1 | 3
  Muscle/Bone Pain Symptom: Cycle 40 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 55.56 (19.245)
  Muscle/Bone Pain Symptom: Cycle 41: number analyzed (Participants) | 0 | 3
  Muscle/Bone Pain Symptom: Cycle 41 |  | 55.56 (19.245)
  Muscle/Bone Pain Symptom: Cycle 42: number analyzed (Participants) | 0 | 2
  Muscle/Bone Pain Symptom: Cycle 42 |  | 50.00 (23.570)
  Muscle/Bone Pain Symptom: Cycle 43: number analyzed (Participants) | 0 | 1
  Muscle/Bone Pain Symptom: Cycle 43 |  | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Muscle/Bone Pain Symptom: EOT: number analyzed (Participants) | 33 | 29
  Muscle/Bone Pain Symptom: EOT | 25.25 (27.677) | 26.44 (30.052)
  Sexual Function: Cycle 1: number analyzed (Participants) | 34 | 29
  Sexual Function: Cycle 1 | 22.55 (31.485) | 34.48 (35.054)
  Sexual Function: Cycle 2: number analyzed (Participants) | 43 | 30
  Sexual Function: Cycle 2 | 17.83 (25.561) | 30.00 (30.763)
  Sexual Function: Cycle 3: number analyzed (Participants) | 39 | 29
  Sexual Function: Cycle 3 | 17.95 (25.185) | 36.78 (32.544)
  Sexual Function: Cycle 4: number analyzed (Participants) | 34 | 27
  Sexual Function: Cycle 4 | 18.63 (24.878) | 22.22 (30.662)
  Sexual Function: Cycle 5: number analyzed (Participants) | 32 | 27
  Sexual Function: Cycle 5 | 18.75 (25.312) | 28.40 (35.450)
  Sexual Function: Cycle 6: number analyzed (Participants) | 30 | 23
  Sexual Function: Cycle 6 | 14.44 (20.869) | 31.88 (35.503)
  Sexual Function: Cycle 7: number analyzed (Participants) | 28 | 23
  Sexual Function: Cycle 7 | 19.05 (24.727) | 30.43 (37.488)
  Sexual Function: Cycle 8: number analyzed (Participants) | 26 | 16
  Sexual Function: Cycle 8 | 23.08 (27.919) | 27.08 (27.806)
  Sexual Function: Cycle 9: number analyzed (Participants) | 25 | 19
  Sexual Function: Cycle 9 | 13.33 (27.217) | 28.07 (31.940)
  Sexual Function: Cycle 10: number analyzed (Participants) | 25 | 16
  Sexual Function: Cycle 10 | 17.33 (29.059) | 27.08 (32.702)
  Sexual Function: Cycle 11: number analyzed (Participants) | 25 | 16
  Sexual Function: Cycle 11 | 16.00 (25.676) | 20.83 (26.874)
  Sexual Function: Cycle 12: number analyzed (Participants) | 26 | 14
  Sexual Function: Cycle 12 | 20.51 (29.929) | 19.05 (25.198)
  Sexual Function: Cycle 13: number analyzed (Participants) | 24 | 15
  Sexual Function: Cycle 13 | 16.67 (26.006) | 22.22 (32.530)
  Sexual Function: Cycle 14: number analyzed (Participants) | 25 | 14
  Sexual Function: Cycle 14 | 20.00 (27.217) | 26.19 (26.726)
  Sexual Function: Cycle 15: number analyzed (Participants) | 21 | 12
  Sexual Function: Cycle 15 | 17.46 (27.119) | 19.44 (26.432)
  Sexual Function: Cycle 16: number analyzed (Participants) | 19 | 13
  Sexual Function: Cycle 16 | 22.81 (33.431) | 25.64 (27.735)
  Sexual Function: Cycle 17: number analyzed (Participants) | 15 | 12
  Sexual Function: Cycle 17 | 20.00 (27.603) | 22.22 (25.950)
  Sexual Function: Cycle 18: number analyzed (Participants) | 12 | 11
  Sexual Function: Cycle 18 | 22.22 (21.711) | 18.18 (27.340)
  Sexual Function: Cycle 19: number analyzed (Participants) | 7 | 10
  Sexual Function: Cycle 19 | 19.05 (26.227) | 20.00 (28.109)
  Sexual Function: Cycle 20: number analyzed (Participants) | 8 | 10
  Sexual Function: Cycle 20 | 25.00 (29.547) | 13.33 (23.307)
  Sexual Function: Cycle 21: number analyzed (Participants) | 7 | 9
  Sexual Function: Cycle 21 | 23.81 (25.198) | 14.81 (24.216)
  Sexual Function: Cycle 22: number analyzed (Participants) | 8 | 9
  Sexual Function: Cycle 22 | 33.33 (30.861) | 14.81 (24.216)
  Sexual Function: Cycle 23: number analyzed (Participants) | 7 | 8
  Sexual Function: Cycle 23 | 23.81 (31.706) | 20.83 (24.801)
  Sexual Function: Cycle 24: number analyzed (Participants) | 5 | 8
  Sexual Function: Cycle 24 | 26.67 (27.889) | 16.67 (25.198)
  Sexual Function: Cycle 25: number analyzed (Participants) | 5 | 6
  Sexual Function: Cycle 25 | 26.67 (36.515) | 16.67 (27.889)
  Sexual Function: Cycle 26: number analyzed (Participants) | 4 | 6
  Sexual Function: Cycle 26 | 25.00 (31.914) | 16.67 (27.889)
  Sexual Function: Cycle 27: number analyzed (Participants) | 1 | 6
  Sexual Function: Cycle 27 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (27.889)
  Sexual Function: Cycle 28: number analyzed (Participants) | 3 | 6
  Sexual Function: Cycle 28 | 33.33 (33.333) | 16.67 (27.889)
  Sexual Function: Cycle 29: number analyzed (Participants) | 1 | 6
  Sexual Function: Cycle 29 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (27.889)
  Sexual Function: Cycle 30: number analyzed (Participants) | 1 | 6
  Sexual Function: Cycle 30 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (27.889)
  Sexual Function: Cycle 31: number analyzed (Participants) | 1 | 6
  Sexual Function: Cycle 31 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (27.889)
  Sexual Function: Cycle 32: number analyzed (Participants) | 3 | 5
  Sexual Function: Cycle 32 | 22.22 (38.490) | 20.00 (29.814)
  Sexual Function: Cycle 33: number analyzed (Participants) | 1 | 5
  Sexual Function: Cycle 33 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 20.00 (29.814)
  Sexual Function: Cycle 34: number analyzed (Participants) | 1 | 5
  Sexual Function: Cycle 34 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 33.33 (33.333)
  Sexual Function: Cycle 35: number analyzed (Participants) | 1 | 5
  Sexual Function: Cycle 35 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 20.00 (29.814)
  Sexual Function: Cycle 36: number analyzed (Participants) | 1 | 4
  Sexual Function: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 25.00 (31.914)
  Sexual Function: Cycle 37: number analyzed (Participants) | 1 | 3
  Sexual Function: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 33.33 (33.333)
  Sexual Function: Cycle 38: number analyzed (Participants) | 0 | 3
  Sexual Function: Cycle 38 |  | 33.33 (33.333)
  Sexual Function: Cycle 39: number analyzed (Participants) | 1 | 2
  Sexual Function: Cycle 39 | 33.33 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 16.67 (23.570)
  Sexual Function: Cycle 40: number analyzed (Participants) | 1 | 2
  Sexual Function: Cycle 40 | 66.67 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Sexual Function: Cycle 41: number analyzed (Participants) | 0 | 2
  Sexual Function: Cycle 41 |  | 16.67 (23.570)
  Sexual Function: Cycle 42: number analyzed (Participants) | 0 | 1
  Sexual Function: Cycle 42 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Sexual Function: Cycle 43: number analyzed (Participants) | 0 | 1
  Sexual Function: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Sexual Function: EOT: number analyzed (Participants) | 22 | 19
  Sexual Function: EOT | 25.76 (27.084) | 49.12 (37.463)
  Information/Communication: Cycle 1: number analyzed (Participants) | 61 | 44
  Information/Communication: Cycle 1 | 8.74 (21.860) | 6.82 (15.384)
  Information/Communication: Cycle 2: number analyzed (Participants) | 57 | 41
  Information/Communication: Cycle 2 | 5.85 (12.791) | 5.69 (14.724)
  Information/Communication: Cycle 3: number analyzed (Participants) | 55 | 40
  Information/Communication: Cycle 3 | 5.45 (14.001) | 5.00 (14.222)
  Information/Communication: Cycle 4: number analyzed (Participants) | 50 | 38
  Information/Communication: Cycle 4 | 4.67 (11.684) | 5.26 (12.318)
  Information/Communication: Cycle 5: number analyzed (Participants) | 47 | 33
  Information/Communication: Cycle 5 | 3.55 (10.389) | 7.07 (18.177)
  Information/Communication: Cycle 6: number analyzed (Participants) | 43 | 31
  Information/Communication: Cycle 6 | 4.65 (11.687) | 5.38 (15.146)
  Information/Communication: Cycle 7: number analyzed (Participants) | 39 | 29
  Information/Communication: Cycle 7 | 6.84 (13.636) | 9.20 (23.395)
  Information/Communication: Cycle 8: number analyzed (Participants) | 37 | 25
  Information/Communication: Cycle 8 | 8.11 (16.491) | 5.33 (15.753)
  Information/Communication: Cycle 9: number analyzed (Participants) | 35 | 26
  Information/Communication: Cycle 9 | 5.71 (12.746) | 3.85 (10.860)
  Information/Communication: Cycle 10: number analyzed (Participants) | 35 | 23
  Information/Communication: Cycle 10 | 8.57 (16.848) | 7.25 (17.281)
  Information/Communication: Cycle 11: number analyzed (Participants) | 35 | 24
  Information/Communication: Cycle 11 | 7.62 (18.232) | 5.56 (16.051)
  Information/Communication: Cycle 12: number analyzed (Participants) | 35 | 22
  Information/Communication: Cycle 12 | 10.48 (22.537) | 1.52 (7.107)
  Information/Communication: Cycle 13: number analyzed (Participants) | 34 | 21
  Information/Communication: Cycle 13 | 3.92 (10.901) | 4.76 (11.952)
  Information/Communication: Cycle 14: number analyzed (Participants) | 31 | 19
  Information/Communication: Cycle 14 | 6.45 (13.387) | 3.51 (10.510)
  Information/Communication: Cycle 15: number analyzed (Participants) | 30 | 17
  Information/Communication: Cycle 15 | 4.44 (11.525) | 7.84 (18.743)
  Information/Communication: Cycle 16: number analyzed (Participants) | 27 | 16
  Information/Communication: Cycle 16 | 2.47 (8.896) | 8.33 (14.907)
  Information/Communication: Cycle 17: number analyzed (Participants) | 22 | 15
  Information/Communication: Cycle 17 | 4.55 (11.708) | 2.22 (8.607)
  Information/Communication: Cycle 18: number analyzed (Participants) | 17 | 14
  Information/Communication: Cycle 18 | 7.84 (14.575) | 7.14 (19.298)
  Information/Communication: Cycle 19: number analyzed (Participants) | 12 | 14
  Information/Communication: Cycle 19 | 0.00 (0.000) | 2.38 (8.909)
  Information/Communication: Cycle 20: number analyzed (Participants) | 11 | 13
  Information/Communication: Cycle 20 | 3.03 (10.050) | 2.56 (9.245)
  Information/Communication: Cycle 21: number analyzed (Participants) | 11 | 12
  Information/Communication: Cycle 21 | 6.06 (13.484) | 2.78 (9.623)
  Information/Communication: Cycle 22: number analyzed (Participants) | 11 | 11
  Information/Communication: Cycle 22 | 6.06 (13.484) | 3.03 (10.050)
  Information/Communication: Cycle 23: number analyzed (Participants) | 11 | 10
  Information/Communication: Cycle 23 | 9.09 (21.556) | 3.33 (10.541)
  Information/Communication: Cycle 24: number analyzed (Participants) | 10 | 10
  Information/Communication: Cycle 24 | 10.00 (22.498) | 3.33 (10.541)
  Information/Communication: Cycle 25: number analyzed (Participants) | 10 | 8
  Information/Communication: Cycle 25 | 6.67 (14.055) | 4.17 (11.785)
  Information/Communication: Cycle 26: number analyzed (Participants) | 6 | 7
  Information/Communication: Cycle 26 | 11.11 (17.213) | 4.76 (12.599)
  Information/Communication: Cycle 27: number analyzed (Participants) | 6 | 8
  Information/Communication: Cycle 27 | 0.00 (0.000) | 4.17 (11.785)
  Information/Communication: Cycle 28: number analyzed (Participants) | 7 | 8
  Information/Communication: Cycle 28 | 9.52 (16.265) | 4.17 (11.785)
  Information/Communication: Cycle 29: number analyzed (Participants) | 6 | 7
  Information/Communication: Cycle 29 | 5.56 (13.608) | 4.76 (12.599)
  Information/Communication: Cycle 30: number analyzed (Participants) | 5 | 7
  Information/Communication: Cycle 30 | 0.00 (0.000) | 4.76 (12.599)
  Information/Communication: Cycle 31: number analyzed (Participants) | 3 | 7
  Information/Communication: Cycle 31 | 0.00 (0.000) | 4.76 (12.599)
  Information/Communication: Cycle 32: number analyzed (Participants) | 3 | 6
  Information/Communication: Cycle 32 | 0.00 (0.000) | 5.56 (13.608)
  Information/Communication: Cycle 33: number analyzed (Participants) | 3 | 6
  Information/Communication: Cycle 33 | 11.11 (19.245) | 0.00 (0.000)
  Information/Communication: Cycle 34: number analyzed (Participants) | 3 | 6
  Information/Communication: Cycle 34 | 11.11 (19.245) | 5.56 (13.608)
  Information/Communication: Cycle 35: number analyzed (Participants) | 2 | 6
  Information/Communication: Cycle 35 | 0.00 (0.000) | 5.56 (13.608)
  Information/Communication: Cycle 36: number analyzed (Participants) | 1 | 5
  Information/Communication: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Information/Communication: Cycle 37: number analyzed (Participants) | 1 | 4
  Information/Communication: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Information/Communication: Cycle 38: number analyzed (Participants) | 0 | 4
  Information/Communication: Cycle 38 |  | 8.33 (16.667)
  Information/Communication: Cycle 39: number analyzed (Participants) | 1 | 3
  Information/Communication: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Information/Communication: Cycle 40: number analyzed (Participants) | 1 | 3
  Information/Communication: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 11.11 (19.245)
  Information/Communication: Cycle 41: number analyzed (Participants) | 0 | 3
  Information/Communication: Cycle 41 |  | 11.11 (19.245)
  Information/Communication: Cycle 42: number analyzed (Participants) | 0 | 2
  Information/Communication: Cycle 42 |  | 0.00 (0.000)
  Information/Communication: Cycle 43: number analyzed (Participants) | 0 | 1
  Information/Communication: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Information/Communication: EOT: number analyzed (Participants) | 33 | 29
  Information/Communication: EOT | 10.10 (19.516) | 5.75 (20.057)
  Body Image: Cycle 1: number analyzed (Participants) | 60 | 44
  Body Image: Cycle 1 | 21.67 (32.950) | 24.24 (24.234)
  Body Image: Cycle 2: number analyzed (Participants) | 57 | 41
  Body Image: Cycle 2 | 12.87 (19.674) | 15.45 (25.925)
  Body Image: Cycle 3: number analyzed (Participants) | 52 | 40
  Body Image: Cycle 3 | 10.90 (21.614) | 19.17 (31.020)
  Body Image: Cycle 4: number analyzed (Participants) | 49 | 38
  Body Image: Cycle 4 | 10.88 (17.197) | 16.67 (24.199)
  Body Image: Cycle 5: number analyzed (Participants) | 46 | 33
  Body Image: Cycle 5 | 8.70 (17.826) | 15.15 (25.126)
  Body Image: Cycle 6: number analyzed (Participants) | 42 | 30
  Body Image: Cycle 6 | 11.90 (21.866) | 21.11 (29.664)
  Body Image: Cycle 7: number analyzed (Participants) | 38 | 28
  Body Image: Cycle 7 | 14.91 (25.347) | 21.43 (31.706)
  Body Image: Cycle 8: number analyzed (Participants) | 37 | 24
  Body Image: Cycle 8 | 13.51 (24.164) | 15.28 (24.035)
  Body Image: Cycle 9: number analyzed (Participants) | 35 | 25
  Body Image: Cycle 9 | 14.29 (28.337) | 14.67 (23.727)
  Body Image: Cycle 10: number analyzed (Participants) | 34 | 23
  Body Image: Cycle 10 | 13.73 (24.779) | 18.84 (26.258)
  Body Image: Cycle 11: number analyzed (Participants) | 35 | 24
  Body Image: Cycle 11 | 12.38 (19.944) | 15.28 (24.035)
  Body Image: Cycle 12: number analyzed (Participants) | 35 | 22
  Body Image: Cycle 12 | 10.48 (21.038) | 9.09 (23.417)
  Body Image: Cycle 13: number analyzed (Participants) | 34 | 21
  Body Image: Cycle 13 | 7.84 (20.199) | 7.94 (17.965)
  Body Image: Cycle 14: number analyzed (Participants) | 31 | 19
  Body Image: Cycle 14 | 12.90 (23.847) | 7.02 (13.962)
  Body Image: Cycle 15: number analyzed (Participants) | 29 | 17
  Body Image: Cycle 15 | 9.20 (21.633) | 9.80 (19.596)
  Body Image: Cycle 16: number analyzed (Participants) | 27 | 16
  Body Image: Cycle 16 | 16.05 (28.300) | 10.42 (23.472)
  Body Image: Cycle 17: number analyzed (Participants) | 22 | 15
  Body Image: Cycle 17 | 12.12 (26.318) | 8.89 (15.258)
  Body Image: Cycle 18: number analyzed (Participants) | 17 | 14
  Body Image: Cycle 18 | 15.69 (31.441) | 7.14 (14.194)
  Body Image: Cycle 19: number analyzed (Participants) | 12 | 14
  Body Image: Cycle 19 | 11.11 (25.950) | 2.38 (8.909)
  Body Image: Cycle 20: number analyzed (Participants) | 11 | 12
  Body Image: Cycle 20 | 9.09 (30.151) | 8.33 (15.076)
  Body Image: Cycle 21: number analyzed (Participants) | 11 | 12
  Body Image: Cycle 21 | 9.09 (30.151) | 2.78 (9.623)
  Body Image: Cycle 22: number analyzed (Participants) | 11 | 11
  Body Image: Cycle 22 | 15.15 (31.140) | 6.06 (13.484)
  Body Image: Cycle 23: number analyzed (Participants) | 11 | 10
  Body Image: Cycle 23 | 9.09 (21.556) | 6.67 (14.055)
  Body Image: Cycle 24: number analyzed (Participants) | 10 | 10
  Body Image: Cycle 24 | 16.67 (36.004) | 3.33 (10.541)
  Body Image: Cycle 25: number analyzed (Participants) | 10 | 8
  Body Image: Cycle 25 | 16.67 (36.004) | 8.33 (15.430)
  Body Image: Cycle 26: number analyzed (Participants) | 7 | 7
  Body Image: Cycle 26 | 23.81 (41.786) | 4.76 (12.599)
  Body Image: Cycle 27: number analyzed (Participants) | 6 | 8
  Body Image: Cycle 27 | 22.22 (40.369) | 4.17 (11.785)
  Body Image: Cycle 28: number analyzed (Participants) | 6 | 8
  Body Image: Cycle 28 | 22.22 (40.369) | 12.50 (17.252)
  Body Image: Cycle 29: number analyzed (Participants) | 6 | 7
  Body Image: Cycle 29 | 11.11 (27.217) | 0.00 (0.000)
  Body Image: Cycle 30: number analyzed (Participants) | 5 | 7
  Body Image: Cycle 30 | 0.00 (0.000) | 0.00 (0.000)
  Body Image: Cycle 31: number analyzed (Participants) | 3 | 7
  Body Image: Cycle 31 | 0.00 (0.000) | 0.00 (0.000)
  Body Image: Cycle 32: number analyzed (Participants) | 3 | 6
  Body Image: Cycle 32 | 0.00 (0.000) | 0.00 (0.000)
  Body Image: Cycle 33: number analyzed (Participants) | 3 | 6
  Body Image: Cycle 33 | 0.00 (0.000) | 5.56 (13.608)
  Body Image: Cycle 34: number analyzed (Participants) | 3 | 6
  Body Image: Cycle 34 | 22.22 (38.490) | 5.56 (13.608)
  Body Image: Cycle 35: number analyzed (Participants) | 2 | 6
  Body Image: Cycle 35 | 16.67 (23.570) | 11.11 (17.213)
  Body Image: Cycle 36: number analyzed (Participants) | 1 | 5
  Body Image: Cycle 36 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Body Image: Cycle 37: number analyzed (Participants) | 1 | 4
  Body Image: Cycle 37 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 8.33 (16.667)
  Body Image: Cycle 38: number analyzed (Participants) | 0 | 4
  Body Image: Cycle 38 |  | 8.33 (16.667)
  Body Image: Cycle 39: number analyzed (Participants) | 1 | 3
  Body Image: Cycle 39 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 22.22 (38.490)
  Body Image: Cycle 40: number analyzed (Participants) | 1 | 3
  Body Image: Cycle 40 | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 0.00 (0.000)
  Body Image: Cycle 41: number analyzed (Participants) | 0 | 3
  Body Image: Cycle 41 |  | 11.11 (19.245)
  Body Image: Cycle 42: number analyzed (Participants) | 0 | 2
  Body Image: Cycle 42 |  | 0.00 (0.000)
  Body Image: Cycle 43: number analyzed (Participants) | 0 | 1
  Body Image: Cycle 43 |  | 0.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  Body Image: EOT: number analyzed (Participants) | 33 | 29
  Body Image: EOT | 23.23 (32.792) | 18.39 (31.605)

14. Secondary Outcome: Plasma Concentration of Soluble Protein Biomarker (sKIT)
Time Frame: Pre-dose on Day 1 and 15 of Cycle 1, Day 1 of Cycle 2, 3 and every 2 cycles thereafter (Cycle 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, 39, 41, 43), End of Treatment (up to maximum duration of 1226 days)
Population: sKIT analysis set: enrolled participants who received at least 1 dose of study drug, had at least 1 biomarker parameter from corresponding assay sample with both baseline and post-treatment assessment. Here, "0 participants" in "number analyzed" field=none of the participants were evaluable in given group at this time point, hence data not reported
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pcg/mL)
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 58 | 45
picogram per milliliter (pcg/mL)
  Cycle1/Day1 | 58218.8 (18406.35) | 62267.7 (17298.53)
  Cycle1/Day15: number analyzed (Participants) | 58 | 44
  Cycle1/Day15 | 51614.2 (18638.21) | 48946.4 (15189.15)
  Cycle2/Day1: number analyzed (Participants) | 56 | 44
  Cycle2/Day1 | 37705.1 (14128.27) | 40334.8 (14304.02)
  Cycle3/Day1: number analyzed (Participants) | 52 | 41
  Cycle3/Day1 | 26939.9 (10839.77) | 30224.0 (13709.28)
  Cycle5/Day1: number analyzed (Participants) | 46 | 35
  Cycle5/Day1 | 20596.1 (7331.69) | 23892.6 (11355.85)
  Cycle7/Day1: number analyzed (Participants) | 38 | 29
  Cycle7/Day1 | 18222.9 (8010.89) | 19786.4 (10564.09)
  Cycle9/Day1: number analyzed (Participants) | 32 | 24
  Cycle9/Day1 | 17677.0 (6179.43) | 19761.3 (12429.49)
  Cycle11/Day1: number analyzed (Participants) | 33 | 23
  Cycle11/Day1 | 16689.8 (7452.02) | 21091.1 (13222.55)
  Cycle13/Day1: number analyzed (Participants) | 30 | 20
  Cycle13/Day1 | 16657.7 (8876.97) | 18103.0 (7763.15)
  Cycle15/Day1: number analyzed (Participants) | 28 | 14
  Cycle15/Day1 | 15675.0 (6591.98) | 16222.5 (4939.29)
  Cycle17/Day1: number analyzed (Participants) | 21 | 15
  Cycle17/Day1 | 15705.5 (5665.32) | 15769.0 (7628.43)
  Cycle19/Day1: number analyzed (Participants) | 12 | 13
  Cycle19/Day1 | 14600.0 (4537.41) | 15811.2 (7297.71)
  Cycle21/Day1: number analyzed (Participants) | 11 | 10
  Cycle21/Day1 | 14809.5 (4395.74) | 15577.0 (5782.28)
  Cycle23/Day1: number analyzed (Participants) | 11 | 8
  Cycle23/Day1 | 13332.3 (3670.43) | 12238.8 (4252.01)
  Cycle25/Day1: number analyzed (Participants) | 10 | 7
  Cycle25/Day1 | 13674.0 (5440.63) | 13112.1 (5057.35)
  Cycle27/Day1: number analyzed (Participants) | 5 | 8
  Cycle27/Day1 | 12616.0 (3513.31) | 16553.1 (8092.47)
  Cycle29/Day1: number analyzed (Participants) | 4 | 7
  Cycle29/Day1 | 13638.8 (3555.38) | 16261.4 (10057.56)
  Cycle31/Day1: number analyzed (Participants) | 2 | 6
  Cycle31/Day1 | 9567.5 (1644.02) | 10950.8 (4149.34)
  Cycle33/Day1: number analyzed (Participants) | 2 | 6
  Cycle33/Day1 | 9440.0 (1541.49) | 10590.0 (4008.65)
  Cycle35/Day1: number analyzed (Participants) | 1 | 6
  Cycle35/Day1 | 11255.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 10241.7 (2748.91)
  Cycle37/Day1: number analyzed (Participants) | 0 | 4
  Cycle37/Day1 |  | 9038.8 (3243.45)
  Cycle39/Day1: number analyzed (Participants) | 0 | 2
  Cycle39/Day1 |  | 8672.5 (477.30)
  Cycle41/Day1: number analyzed (Participants) | 0 | 3
  Cycle41/Day1 |  | 7023.3 (1849.00)
  Cycle43/Day1: number analyzed (Participants) | 0 | 1
  Cycle43/Day1 |  | 9360.0 (NA) — Standard deviation was not estimable since only 1 participant was evaluable.
  EOT: number analyzed (Participants) | 30 | 28
  EOT | 21680.3 (10358.35) | 22605.5 (10953.00)

15. Secondary Outcome: Minimum Observed Plasma Concentration (Ctrough) of Sunitinib and Its Metabolite SU012662
Description: Ctrough is the minimum observed plasma concentration of drug. SU012662 is the metabolite of sunitinib.
Time Frame: Pre-dose on Day 15 of Cycle 1, Day 1 of Cycle 2, 3 and 5
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study medication, had baseline and at least 1 post-baseline value for each parameters.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
nanogram per milliliter (ng/mL)
  Sunitinib: Cycle1/Day15: number analyzed (Participants) | 60 | 44
  Sunitinib: Cycle1/Day15 | 52.78 (27.361) | 41.93 (21.707)
  Sunitinib: Cycle2/Day1: number analyzed (Participants) | 57 | 44
  Sunitinib: Cycle2/Day1 | 42.68 (20.320) | 38.38 (22.765)
  Sunitinib: Cycle3/Day1: number analyzed (Participants) | 54 | 41
  Sunitinib: Cycle3/Day1 | 41.79 (21.517) | 38.49 (18.750)
  Sunitinib: Cycle5/Day1: number analyzed (Participants) | 48 | 35
  Sunitinib: Cycle5/Day1 | 35.57 (15.221) | 33.60 (15.010)
  SU012662: Cycle1/Day15: number analyzed (Participants) | 60 | 44
  SU012662: Cycle1/Day15 | 18.03 (11.169) | 14.26 (9.264)
  SU012662: Cycle2/Day1: number analyzed (Participants) | 57 | 44
  SU012662: Cycle2/Day1 | 15.94 (9.059) | 12.53 (8.000)
  SU012662: Cycle3/Day1: number analyzed (Participants) | 54 | 41
  SU012662: Cycle3/Day1 | 15.85 (9.444) | 13.64 (6.983)
  SU012662: Cycle5/Day1: number analyzed (Participants) | 48 | 35
  SU012662: Cycle5/Day1 | 12.78 (6.375) | 12.61 (6.735)

16. Secondary Outcome: Dose-Corrected Trough Plasma Concentration of Sunitinib and Its Metabolite SU012662
Description: Dose-corrected plasma trough concentration is calculated as: trough plasma concentration*(intended dose divided by actual dose). Intended dose was defined as the starting dose in the study and actual dose was defined as the last dose which the participant had received. SU012662 is the metabolite of sunitinib.
Time Frame: Pre dose on Day 15 of Cycle 1, Day 1 of Cycle 2, 3 and 5
Population: PK population included all participants who received at least 1 dose of study medication, had baseline and at least 1 post-baseline value for each parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
ng/mL
  Sunitinib: Cycle1/Day15: number analyzed (Participants) | 59 | 40
  Sunitinib: Cycle1/Day15 | 52.66 (27.136) | 43.38 (21.520)
  Sunitinib: Cycle2/Day1: number analyzed (Participants) | 55 | 36
  Sunitinib: Cycle2/Day1 | 42.89 (20.607) | 39.52 (19.833)
  Sunitinib: Cycle3/Day1: number analyzed (Participants) | 49 | 39
  Sunitinib: Cycle3/Day1 | 44.99 (23.031) | 38.56 (18.375)
  Sunitinib: Cycle5/Day1: number analyzed (Participants) | 43 | 35
  Sunitinib: Cycle5/Day1 | 42.49 (16.769) | 33.27 (16.733)
  SU012662: Cycle1/Day15: number analyzed (Participants) | 59 | 40
  SU012662: Cycle1/Day15 | 18.14 (11.059) | 14.79 (9.436)
  SU012662: Cycle2/Day1: number analyzed (Participants) | 55 | 36
  SU012662: Cycle2/Day1 | 16.01 (9.132) | 13.09 (7.684)
  SU012662: Cycle3/Day1: number analyzed (Participants) | 49 | 39
  SU012662: Cycle3/Day1 | 17.37 (10.233) | 14.22 (7.085)
  SU012662: Cycle5/Day1: number analyzed (Participants) | 43 | 35
  SU012662: Cycle5/Day1 | 15.35 (6.882) | 12.53 (6.914)

17. Secondary Outcome: Area Under the Curve (AUC24) of Sunitinib and Its Metabolite SU012662
Description: Area under the plasma concentration-time profile from time zero (pre-dose) to 24 hours post-dose. SU012662 is the metabolite of sunitinib.
Time Frame: Pre-dose (0 hour) and at multiple time points (up to 24 hours) post dose on Day 15 of Cycle 1, Day 1 of Cycle 2, 3 and 5 (each cycle 28 days)
Population: Due to insufficient data, there was substantial uncertainty associated with the parameter estimates; therefore, the population PK/PD analyses was not completed. Instead, the exposure response analyses with respect to different safety and efficacy endpoints were carried out and reported.
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Oral Clearance (CL/F) of Sunitinib and Its Metabolite SU012662
Description: Clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre dose on Day 15 of Cycle 1, Day 1 of Cycle 2, 3 and 5 (each cycle 28 days)
Population: as for outcome 17
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Half Maximal Effective Concentration (EC50) of Sunitinib
Description: Concentration of sunitinib in plasma at which 50 percent of the maximum effect was observed.
Time Frame: Pre dose on Day 15 of Cycle 1, Day 1 of Cycle 2, 3 and 5 (each cycle 28 days)
Population: as for outcome 17
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 1939 days that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants
  AEs | 59 | 45
  SAEs | 17 | 12

21. Secondary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 1939 days that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants
  AEs | 57 | 44
  SAEs | 9 | 3

22. Secondary Outcome: Number of Participants With Adverse Events (AEs) According to Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed according to severity grading based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. Grade 1 =mild; Grade 2 =moderate; within normal limits, Grade 3 =severe or medically significant but not immediately life-threatening; Grade 4 =life-threatening or disabling; urgent intervention indicated; Grade 5 =death.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants
  Grade 1 | 4 | 5
  Grade 2 | 9 | 9
  Grade 3 | 38 | 23
  Grade 4 | 6 | 6
  Grade 5 | 2 | 2

23. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, red blood cell count, platelet count, white blood cell count, total neutrophils, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine); electrolytes (sodium, potassium, chloride, calcium, magnesium, phosphate); urinalysis (urine protein), miscellaneous (pregnancy test, Chromogranin A). Clinically significant laboratory abnormalities were identified by the Investigator.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants | 30 | 22

24. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs Abnormalities
Description: Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, body temperature and heart rate.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants | 30 | 22

25. Secondary Outcome: Number of Participants With Increase From Baseline in Corrected QT Interval (QTc)
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants | 0 | 0

26. Secondary Outcome: Number of Participants With Change From Baseline in Physical Examinations Findings
Description: Physical examination included an examination of the general appearance, skin, heart, head, eyes, ears, nose, throat, breasts, abdomen, musculoskeletal, neck, extremities, thyroid and others.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants | 23 | 19

27. Secondary Outcome: Number of Participants With Change From Baseline in Body Weight
Description: Participants with increase of >=5 percent and decrease of >=5 percent from baseline in body weight were reported in this outcome measure.
Time Frame: Baseline up to 1939 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
Participants
  Increase of >=5 percent | 27 | 9
  Decrease of >=5 percent | 18 | 15

28. Secondary Outcome: Number of Participants With Eastern Co-operative Oncology Group Performance Status (ECOG-PS)
Description: ECOG-PS performance status is used to assess how the disease affects the daily living abilities of the participant. It was measured on 6-point scale ranging from 0-5, where 0= fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory/able to carry out light or sedentary work; 2= ambulatory for more than 50 percent of waking hours and capable of all self-care but unable to carry out any work activities; 3= capable of limited self-care, confined to bed or chair >50 percent of waking hours; 4= completely disabled, not capable of any self-care, totally confined to bed or chair; 5= dead. A higher score indicated greater functional impairment. Only those ECOG-PS categories, in which at least one participant had data at any indicated time point were reported in this outcome measure. Not reported (NR) category included participants with unavailable ECOG performance status.
Time Frame: as for outcome 12
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here, "0 participants" in the "number analyzed" field signifies none of the participants were evaluable in the given group at this time point, hence data was not reported.
Measure: Number; unit: participants
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Number analyzed (Participants) | 61 | 45
participants
  Cycle 1/Day 1: ECOG-PS =0 | 37 | 25
  Cycle 1/Day 1: ECOG-PS =1 | 15 | 14
  Cycle 1/Day 1: ECOG-PS =NR | 9 | 6
  Cycle 2/Day 1: ECOG-PS =0: number analyzed (Participants) | 59 | 44
  Cycle 2/Day 1: ECOG-PS =0 | 37 | 30
  Cycle 2/Day 1: ECOG-PS =1: number analyzed (Participants) | 59 | 44
  Cycle 2/Day 1: ECOG-PS =1 | 19 | 13
  Cycle 2/Day 1: ECOG-PS =NR: number analyzed (Participants) | 59 | 44
  Cycle 2/Day 1: ECOG-PS =NR | 3 | 1
  Cycle 3/Day 1: ECOG-PS =0: number analyzed (Participants) | 56 | 41
  Cycle 3/Day 1: ECOG-PS =0 | 37 | 29
  Cycle 3/Day 1: ECOG-PS =1: number analyzed (Participants) | 56 | 41
  Cycle 3/Day 1: ECOG-PS =1 | 17 | 10
  Cycle 3/Day 1: ECOG-PS =2: number analyzed (Participants) | 56 | 41
  Cycle 3/Day 1: ECOG-PS =2 | 0 | 1
  Cycle 3/Day 1: ECOG-PS =3: number analyzed (Participants) | 56 | 41
  Cycle 3/Day 1: ECOG-PS =3 | 0 | 1
  Cycle 3/Day 1: ECOG-PS =NR: number analyzed (Participants) | 56 | 41
  Cycle 3/Day 1: ECOG-PS =NR | 2 | 0
  Cycle 4/Day 1: ECOG-PS =0: number analyzed (Participants) | 51 | 39
  Cycle 4/Day 1: ECOG-PS =0 | 34 | 25
  Cycle 4/Day 1: ECOG-PS =1: number analyzed (Participants) | 51 | 39
  Cycle 4/Day 1: ECOG-PS =1 | 15 | 13
  Cycle 4/Day 1: ECOG-PS =NR: number analyzed (Participants) | 51 | 39
  Cycle 4/Day 1: ECOG-PS =NR | 2 | 1
  Cycle 5/Day 1: ECOG-PS =0: number analyzed (Participants) | 48 | 35
  Cycle 5/Day 1: ECOG-PS =0 | 34 | 23
  Cycle 5/Day 1: ECOG-PS =1: number analyzed (Participants) | 48 | 35
  Cycle 5/Day 1: ECOG-PS =1 | 13 | 11
  Cycle 5/Day 1: ECOG-PS =2: number analyzed (Participants) | 48 | 35
  Cycle 5/Day 1: ECOG-PS =2 | 1 | 1
  Cycle 6/Day 1: ECOG-PS =0: number analyzed (Participants) | 43 | 31
  Cycle 6/Day 1: ECOG-PS =0 | 30 | 21
  Cycle 6/Day 1: ECOG-PS =1: number analyzed (Participants) | 43 | 31
  Cycle 6/Day 1: ECOG-PS =1 | 13 | 9
  Cycle 6/Day 1: ECOG-PS =2: number analyzed (Participants) | 43 | 31
  Cycle 6/Day 1: ECOG-PS =2 | 0 | 1
  Cycle 7/Day 1: ECOG-PS =0: number analyzed (Participants) | 40 | 29
  Cycle 7/Day 1: ECOG-PS =0 | 27 | 21
  Cycle 7/Day 1: ECOG-PS =1: number analyzed (Participants) | 40 | 29
  Cycle 7/Day 1: ECOG-PS =1 | 13 | 7
  Cycle 7/Day 1: ECOG-PS =2: number analyzed (Participants) | 40 | 29
  Cycle 7/Day 1: ECOG-PS =2 | 0 | 1
  Cycle 8/Day 1: ECOG-PS =0: number analyzed (Participants) | 37 | 26
  Cycle 8/Day 1: ECOG-PS =0 | 24 | 20
  Cycle 8/Day 1: ECOG-PS =1: number analyzed (Participants) | 37 | 26
  Cycle 8/Day 1: ECOG-PS =1 | 13 | 6
  Cycle 9/Day 1: ECOG-PS =0: number analyzed (Participants) | 35 | 26
  Cycle 9/Day 1: ECOG-PS =0 | 24 | 20
  Cycle 9/Day 1: ECOG-PS =1: number analyzed (Participants) | 35 | 26
  Cycle 9/Day 1: ECOG-PS =1 | 11 | 6
  Cycle 10/Day 1: ECOG-PS =0: number analyzed (Participants) | 35 | 25
  Cycle 10/Day 1: ECOG-PS =0 | 22 | 18
  Cycle 10/Day 1: ECOG-PS =1: number analyzed (Participants) | 35 | 25
  Cycle 10/Day 1: ECOG-PS =1 | 13 | 6
  Cycle 10/Day 1: ECOG-PS =NR: number analyzed (Participants) | 35 | 25
  Cycle 10/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 11/Day 1: ECOG-PS =0: number analyzed (Participants) | 35 | 24
  Cycle 11/Day 1: ECOG-PS =0 | 22 | 18
  Cycle 11/Day 1: ECOG-PS =1: number analyzed (Participants) | 35 | 24
  Cycle 11/Day 1: ECOG-PS =1 | 13 | 6
  Cycle 12/Day 1: ECOG-PS =0: number analyzed (Participants) | 35 | 22
  Cycle 12/Day 1: ECOG-PS =0 | 22 | 16
  Cycle 12/Day 1: ECOG-PS =1: number analyzed (Participants) | 35 | 22
  Cycle 12/Day 1: ECOG-PS =1 | 13 | 6
  Cycle 13/Day 1: ECOG-PS =0: number analyzed (Participants) | 34 | 21
  Cycle 13/Day 1: ECOG-PS =0 | 21 | 15
  Cycle 13/Day 1: ECOG-PS =1: number analyzed (Participants) | 34 | 21
  Cycle 13/Day 1: ECOG-PS =1 | 13 | 6
  Cycle 14/Day 1: ECOG-PS =0: number analyzed (Participants) | 31 | 20
  Cycle 14/Day 1: ECOG-PS =0 | 19 | 12
  Cycle 14/Day 1: ECOG-PS =1: number analyzed (Participants) | 31 | 20
  Cycle 14/Day 1: ECOG-PS =1 | 11 | 6
  Cycle 14/Day 1: ECOG-PS =NR: number analyzed (Participants) | 31 | 20
  Cycle 14/Day 1: ECOG-PS =NR | 1 | 2
  Cycle 15/Day 1: ECOG-PS =0: number analyzed (Participants) | 30 | 17
  Cycle 15/Day 1: ECOG-PS =0 | 20 | 13
  Cycle 15/Day 1: ECOG-PS =1: number analyzed (Participants) | 30 | 17
  Cycle 15/Day 1: ECOG-PS =1 | 10 | 4
  Cycle 16/Day 1: ECOG-PS =0: number analyzed (Participants) | 27 | 16
  Cycle 16/Day 1: ECOG-PS =0 | 16 | 13
  Cycle 16/Day 1: ECOG-PS =1: number analyzed (Participants) | 27 | 16
  Cycle 16/Day 1: ECOG-PS =1 | 10 | 3
  Cycle 16/Day 1: ECOG-PS =NR: number analyzed (Participants) | 27 | 16
  Cycle 16/Day 1: ECOG-PS =NR | 1 | 0
  Cycle 17/Day 1: ECOG-PS =0: number analyzed (Participants) | 22 | 15
  Cycle 17/Day 1: ECOG-PS =0 | 15 | 13
  Cycle 17/Day 1: ECOG-PS =1: number analyzed (Participants) | 22 | 15
  Cycle 17/Day 1: ECOG-PS =1 | 6 | 2
  Cycle 17/Day 1: ECOG-PS =NR: number analyzed (Participants) | 22 | 15
  Cycle 17/Day 1: ECOG-PS =NR | 1 | 0
  Cycle 18/Day 1: ECOG-PS =0: number analyzed (Participants) | 17 | 14
  Cycle 18/Day 1: ECOG-PS =0 | 10 | 12
  Cycle 18/Day 1: ECOG-PS =1: number analyzed (Participants) | 17 | 14
  Cycle 18/Day 1: ECOG-PS =1 | 5 | 1
  Cycle 18/Day 1: ECOG-PS =NR: number analyzed (Participants) | 17 | 14
  Cycle 18/Day 1: ECOG-PS =NR | 2 | 1
  Cycle 19/Day 1: ECOG-PS =0: number analyzed (Participants) | 12 | 14
  Cycle 19/Day 1: ECOG-PS =0 | 8 | 12
  Cycle 19/Day 1: ECOG-PS =1: number analyzed (Participants) | 12 | 14
  Cycle 19/Day 1: ECOG-PS =1 | 3 | 1
  Cycle 19/Day 1: ECOG-PS =2: number analyzed (Participants) | 12 | 14
  Cycle 19/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 19/Day 1: ECOG-PS =NR: number analyzed (Participants) | 12 | 14
  Cycle 19/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 20/Day 1: ECOG-PS =0: number analyzed (Participants) | 12 | 13
  Cycle 20/Day 1: ECOG-PS =0 | 8 | 11
  Cycle 20/Day 1: ECOG-PS =1: number analyzed (Participants) | 12 | 13
  Cycle 20/Day 1: ECOG-PS =1 | 2 | 1
  Cycle 20/Day 1: ECOG-PS =2: number analyzed (Participants) | 12 | 13
  Cycle 20/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 20/Day 1: ECOG-PS =NR: number analyzed (Participants) | 12 | 13
  Cycle 20/Day 1: ECOG-PS =NR | 1 | 1
  Cycle 21/Day 1: ECOG-PS =0: number analyzed (Participants) | 11 | 12
  Cycle 21/Day 1: ECOG-PS =0 | 7 | 9
  Cycle 21/Day 1: ECOG-PS =1: number analyzed (Participants) | 11 | 12
  Cycle 21/Day 1: ECOG-PS =1 | 4 | 2
  Cycle 21/Day 1: ECOG-PS =NR: number analyzed (Participants) | 11 | 12
  Cycle 21/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 22/Day 1: ECOG-PS =0: number analyzed (Participants) | 11 | 11
  Cycle 22/Day 1: ECOG-PS =0 | 8 | 8
  Cycle 22/Day 1: ECOG-PS =1: number analyzed (Participants) | 11 | 11
  Cycle 22/Day 1: ECOG-PS =1 | 3 | 1
  Cycle 22/Day 1: ECOG-PS =3: number analyzed (Participants) | 11 | 11
  Cycle 22/Day 1: ECOG-PS =3 | 0 | 1
  Cycle 22/Day 1: ECOG-PS =NR: number analyzed (Participants) | 11 | 11
  Cycle 22/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 23/Day 1: ECOG-PS =0: number analyzed (Participants) | 11 | 10
  Cycle 23/Day 1: ECOG-PS =0 | 8 | 7
  Cycle 23/Day 1: ECOG-PS =1: number analyzed (Participants) | 11 | 10
  Cycle 23/Day 1: ECOG-PS =1 | 2 | 2
  Cycle 23/Day 1: ECOG-PS =NR: number analyzed (Participants) | 11 | 10
  Cycle 23/Day 1: ECOG-PS =NR | 1 | 1
  Cycle 24/Day 1: ECOG-PS =0: number analyzed (Participants) | 10 | 10
  Cycle 24/Day 1: ECOG-PS =0 | 9 | 7
  Cycle 24/Day 1: ECOG-PS =1: number analyzed (Participants) | 10 | 10
  Cycle 24/Day 1: ECOG-PS =1 | 0 | 2
  Cycle 24/Day 1: ECOG-PS =2: number analyzed (Participants) | 10 | 10
  Cycle 24/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 24/Day 1: ECOG-PS =NR: number analyzed (Participants) | 10 | 10
  Cycle 24/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 25/Day 1: ECOG-PS =0: number analyzed (Participants) | 10 | 8
  Cycle 25/Day 1: ECOG-PS =0 | 8 | 6
  Cycle 25/Day 1: ECOG-PS =1: number analyzed (Participants) | 10 | 8
  Cycle 25/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 25/Day 1: ECOG-PS =2: number analyzed (Participants) | 10 | 8
  Cycle 25/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 25/Day 1: ECOG-PS =NR: number analyzed (Participants) | 10 | 8
  Cycle 25/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 26/Day 1: ECOG-PS =0: number analyzed (Participants) | 7 | 8
  Cycle 26/Day 1: ECOG-PS =0 | 5 | 7
  Cycle 26/Day 1: ECOG-PS =1: number analyzed (Participants) | 7 | 8
  Cycle 26/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 26/Day 1: ECOG-PS =2: number analyzed (Participants) | 7 | 8
  Cycle 26/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 27/Day 1: ECOG-PS =0: number analyzed (Participants) | 7 | 8
  Cycle 27/Day 1: ECOG-PS =0 | 4 | 7
  Cycle 27/Day 1: ECOG-PS =1: number analyzed (Participants) | 7 | 8
  Cycle 27/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 27/Day 1: ECOG-PS =2: number analyzed (Participants) | 7 | 8
  Cycle 27/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 27/Day 1: ECOG-PS =NR: number analyzed (Participants) | 7 | 8
  Cycle 27/Day 1: ECOG-PS =NR | 1 | 0
  Cycle 28/Day 1: ECOG-PS =0: number analyzed (Participants) | 7 | 8
  Cycle 28/Day 1: ECOG-PS =0 | 5 | 6
  Cycle 28/Day 1: ECOG-PS =1: number analyzed (Participants) | 7 | 8
  Cycle 28/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 28/Day 1: ECOG-PS =2: number analyzed (Participants) | 7 | 8
  Cycle 28/Day 1: ECOG-PS =2 | 1 | 0
  Cycle 28/Day 1: ECOG-PS =NR: number analyzed (Participants) | 7 | 8
  Cycle 28/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 29/Day 1: ECOG-PS =0: number analyzed (Participants) | 6 | 7
  Cycle 29/Day 1: ECOG-PS =0 | 5 | 6
  Cycle 29/Day 1: ECOG-PS =1: number analyzed (Participants) | 6 | 7
  Cycle 29/Day 1: ECOG-PS =1 | 1 | 0
  Cycle 29/Day 1: ECOG-PS =NR: number analyzed (Participants) | 6 | 7
  Cycle 29/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 30/Day 1: ECOG-PS =0: number analyzed (Participants) | 5 | 7
  Cycle 30/Day 1: ECOG-PS =0 | 5 | 6
  Cycle 30/Day 1: ECOG-PS =NR: number analyzed (Participants) | 5 | 7
  Cycle 30/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 31/Day 1: ECOG-PS =0: number analyzed (Participants) | 3 | 7
  Cycle 31/Day 1: ECOG-PS =0 | 2 | 5
  Cycle 31/Day 1: ECOG-PS =1: number analyzed (Participants) | 3 | 7
  Cycle 31/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 31/Day 1: ECOG-PS =NR: number analyzed (Participants) | 3 | 7
  Cycle 31/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 32/Day 1: ECOG-PS =0: number analyzed (Participants) | 3 | 6
  Cycle 32/Day 1: ECOG-PS =0 | 3 | 5
  Cycle 32/Day 1: ECOG-PS =NR: number analyzed (Participants) | 3 | 6
  Cycle 32/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 33/Day 1: ECOG-PS =0: number analyzed (Participants) | 3 | 6
  Cycle 33/Day 1: ECOG-PS =0 | 2 | 4
  Cycle 33/Day 1: ECOG-PS =1: number analyzed (Participants) | 3 | 6
  Cycle 33/Day 1: ECOG-PS =1 | 1 | 1
  Cycle 33/Day 1: ECOG-PS =NR: number analyzed (Participants) | 3 | 6
  Cycle 33/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 34/Day 1: ECOG-PS =0: number analyzed (Participants) | 3 | 6
  Cycle 34/Day 1: ECOG-PS =0 | 3 | 4
  Cycle 34/Day 1: ECOG-PS =1: number analyzed (Participants) | 3 | 6
  Cycle 34/Day 1: ECOG-PS =1 | 0 | 1
  Cycle 34/Day 1: ECOG-PS =NR: number analyzed (Participants) | 3 | 6
  Cycle 34/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 35/Day 1: ECOG-PS =0: number analyzed (Participants) | 2 | 6
  Cycle 35/Day 1: ECOG-PS =0 | 2 | 4
  Cycle 35/Day 1: ECOG-PS =1: number analyzed (Participants) | 2 | 6
  Cycle 35/Day 1: ECOG-PS =1 | 0 | 1
  Cycle 35/Day 1: ECOG-PS =NR: number analyzed (Participants) | 2 | 6
  Cycle 35/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 36/Day 1: ECOG-PS =0: number analyzed (Participants) | 1 | 5
  Cycle 36/Day 1: ECOG-PS =0 | 1 | 3
  Cycle 36/Day 1: ECOG-PS =1: number analyzed (Participants) | 1 | 5
  Cycle 36/Day 1: ECOG-PS =1 | 0 | 1
  Cycle 36/Day 1: ECOG-PS =NR: number analyzed (Participants) | 1 | 5
  Cycle 36/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 37/Day 1: ECOG-PS =0: number analyzed (Participants) | 1 | 4
  Cycle 37/Day 1: ECOG-PS =0 | 1 | 2
  Cycle 37/Day 1: ECOG-PS =1: number analyzed (Participants) | 1 | 4
  Cycle 37/Day 1: ECOG-PS =1 | 0 | 1
  Cycle 37/Day 1: ECOG-PS =NR: number analyzed (Participants) | 1 | 4
  Cycle 37/Day 1: ECOG-PS =NR | 0 | 1
  Cycle 38/Day 1: ECOG-PS =0: number analyzed (Participants) | 1 | 4
  Cycle 38/Day 1: ECOG-PS =0 | 1 | 3
  Cycle 38/Day 1: ECOG-PS =1: number analyzed (Participants) | 1 | 4
  Cycle 38/Day 1: ECOG-PS =1 | 0 | 1
  Cycle 39/Day 1: ECOG-PS =0: number analyzed (Participants) | 1 | 3
  Cycle 39/Day 1: ECOG-PS =0 | 1 | 1
  Cycle 39/Day 1: ECOG-PS =1: number analyzed (Participants) | 1 | 3
  Cycle 39/Day 1: ECOG-PS =1 | 0 | 2
  Cycle 40/Day 1: ECOG-PS =0: number analyzed (Participants) | 1 | 3
  Cycle 40/Day 1: ECOG-PS =0 | 0 | 1
  Cycle 40/Day 1: ECOG-PS =1: number analyzed (Participants) | 1 | 3
  Cycle 40/Day 1: ECOG-PS =1 | 1 | 2
  Cycle 41/Day 1: ECOG-PS =0: number analyzed (Participants) | 0 | 3
  Cycle 41/Day 1: ECOG-PS =0 |  | 1
  Cycle 41/Day 1: ECOG-PS =1: number analyzed (Participants) | 0 | 3
  Cycle 41/Day 1: ECOG-PS =1 |  | 1
  Cycle 41/Day 1: ECOG-PS =NR: number analyzed (Participants) | 0 | 3
  Cycle 41/Day 1: ECOG-PS =NR |  | 1
  Cycle 42/Day 1: ECOG-PS =1: number analyzed (Participants) | 0 | 2
  Cycle 42/Day 1: ECOG-PS =1 |  | 2
  Cycle 43/Day 1: ECOG-PS =1: number analyzed (Participants) | 0 | 1
  Cycle 43/Day 1: ECOG-PS =1 |  | 1
  EOT: ECOG-PS =0: number analyzed (Participants) | 43 | 38
  EOT: ECOG-PS =0 | 20 | 14
  EOT: ECOG-PS =1: number analyzed (Participants) | 43 | 38
  EOT: ECOG-PS =1 | 13 | 12
  EOT: ECOG-PS =2: number analyzed (Participants) | 43 | 38
  EOT: ECOG-PS =2 | 0 | 4
  EOT: ECOG-PS =3: number analyzed (Participants) | 43 | 38
  EOT: ECOG-PS =3 | 1 | 1
  EOT: ECOG-PS =NR: number analyzed (Participants) | 43 | 38
  EOT: ECOG-PS =NR | 9 | 7

ADVERSE EVENTS:
Time Frame: Baseline up to 1939 days
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib: Treatment Naive Cohort | Sunitinib: Later-Line Cohort
Serious Adverse Events (participants affected / at risk) | 17/61 | 12/45
Other Adverse Events (participants affected / at risk) | 59/61 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Treatment Naive Cohort (N=61) | Sunitinib: Later-Line Cohort (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 2 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib: Treatment Naive Cohort (N=61) | Sunitinib: Later-Line Cohort (N=45)
Anaemia (Blood and lymphatic system disorders) | 11 | 9
Leukopenia (Blood and lymphatic system disorders) | 26 | 21
Lymphopenia (Blood and lymphatic system disorders) | 4 | 3
Neutropenia (Blood and lymphatic system disorders) | 37 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 15
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiovascular symptom (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Goitre (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 5 | 3
Thyroid disorder (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Eyelid bleeding (Eye disorders) | 0 | 1
Eyelid disorder (Eye disorders) | 0 | 1
Eyelid oedema (Eye disorders) | 2 | 1
Keratitis (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 3 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 1
Retinal vascular disorder (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 15 | 9
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 33 | 22
Dry mouth (Gastrointestinal disorders) | 2 | 1
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 14
Dysphagia (Gastrointestinal disorders) | 2 | 3
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4
Gingival bleeding (Gastrointestinal disorders) | 3 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 14 | 14
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 3 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 15 | 6
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 10
Asthenia (General disorders) | 11 | 7
Chest pain (General disorders) | 2 | 0
Discomfort (General disorders) | 1 | 0
Face oedema (General disorders) | 3 | 1
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 20 | 13
Feeling cold (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Hyperpyrexia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 6 | 5
Mucous membrane disorder (General disorders) | 1 | 0
Oedema (General disorders) | 5 | 2
Oedema peripheral (General disorders) | 5 | 3
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 6 | 8
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0
Liver injury (Hepatobiliary disorders) | 3 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 2
Cystitis (Infections and infestations) | 2 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Gingival abscess (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 3
Lung infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 2
Oral candidiasis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 6 | 2
Viral infection (Infections and infestations) | 1 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 8
Aspartate aminotransferase increased (Investigations) | 5 | 7
Blood alkaline phosphatase increased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 3
Blood chloride decreased (Investigations) | 1 | 0
Blood chromogranin A increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
Blood folate decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 2 | 0
Blood iron decreased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 3 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood thyroid stimulating hormone abnormal (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 5 | 2
Blood triglycerides increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 3 | 0
C-reactive protein increased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 2 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 4 | 2
Neutrophil count (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 5 | 3
Occult blood positive (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Protein urine (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 3
Red blood cell count decreased (Investigations) | 2 | 3
Red blood cells urine positive (Investigations) | 1 | 0
Thyroxine free decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Tri-iodothyronine decreased (Investigations) | 2 | 0
Tri-iodothyronine free decreased (Investigations) | 1 | 0
Urinary sediment present (Investigations) | 2 | 0
Urobilinogen urine increased (Investigations) | 1 | 0
Vitamin B12 decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 11 | 7
Weight increased (Investigations) | 5 | 2
White blood cell count (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 6 | 1
White blood cells urine positive (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 7
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 6
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 7
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 7
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 14 | 11
Headache (Nervous system disorders) | 12 | 9
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypogeusia (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Neurotoxicity (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 2
Depressed mood (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 5 | 7
Renal colic (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Genital erythema (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Penile erythema (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 | 14
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 8 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Flushing (Vascular disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 16 | 13
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0
Glucose urine present (Investigations) | 0 | 1
Glutathione s-transferase increased (Investigations) | 1 | 0
Procalcitonin increased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 1
Thyroid hormones decreased (Investigations) | 1 | 0
Total bile acids increased (Investigations) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Hypoalbuminaemia (Investigations) | 1 | 1
Bilirubin conjugated increased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.